

### **Clinical Trial Protocol**

| | Document Number: | c09049566-10 |
|---|---|---|
| EudraCT No.:<br>EU Trial No: | 2016-003142-85 | |
| BI Trial No.: | 1280.18 | |
| BI Investigational Product(s): | Xentuzumab (BI 836845) | |
| Title: | An open label, phase Ib, dose-escalation study evaluating the safety and tolerability of xentuzumab and abemaciclib in patients with locally advanced or metastatic solid tumours and in combination with endocrine therapy in patients with locally advanced or metastatic hormone receptor-positive, HER2-, breast cancer, followed by expansion cohorts. | |
| Lay Title: | This study in patients with different types of cancer (solid tumours) aims to find a safe dose of xentuzumab in combination with abemaciclib with or without hormonal therapies. The study also tests how effective these medicines are in patients with lung and breast cancer. | |
| Clinical Phase: | Phase Ib | |
| Trial Clinical<br>Monitor: | Phone: | |
| Coordinating<br>Investigator: | Phone: | |
| Status: | Final Protocol (Revised Protocol based on global amendment 8) | |
| Version and Date: | Version: 9.0 | Date: 04 Mar 2022 |

Proprietary confidential information.

© 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## **CLINICAL TRIAL PROTOCOL SYNOPSIS**

| Name of company: | | Boehringer Ingelheim | |
|---|---|---|---|
| Name of finished proc | luct: | Not applicable | |
| Name of active ingred | lient: | Xentuzumab (BI 836845) | |
| Protocol date: | Trial number: | | Revision date: |
| 30 Nov 2016 | 1280.18 | | 04 Mar 2022 |
| Title of trial: | and tolerability of<br>locally advanced of<br>endocrine therapy | ase Ib, dose-escalation sturb f xentuzumab and abem or metastatic solid tumours in patients with locally r-positive, HER2-, breas | aciclib in patients with<br>and in combination with<br>advanced or metastatic |
| Coordinating | | | |
| Investigator: Trial site(s): | Multi-centre trial, Asia including Jap | international in about 40 s | ites in US, Europe and |
| Clinical phase: | Ib | | |
| Trial Design | | SOLID TUMOURS Cohort A Abemaciclib + xentuzumab (N= approx. 12) RP2D=1 Doub | olet RP2D Part 1 |
| | Cohort B Abemaciclib* + xentuzumab + letrozole (N= approx. 12) RP2D=2 * Abemaciclib dose must b in these cohorts | Cohort C Abemaciclib* + xentuzumab + anastrozole (N= approx. 12) RP2D=3 RP2D=4 Cohort F Non-visceral disease Abemaciclib* + xentuzumab + fulvestrant (N= approx. 12) Cohort D1 Visceral disease Abemaciclib* + xentuzumab + fulvestrant (N= 30) | Cohort E Abemaciclib + xentuzumab (N= 20) Triplets RP2D Part 2 Cohort D2 Non-visceral disease Abemaciclib + xentuzumab + fulvestrant (N= 30) Part 3 |

c09049566-10 Trial Protocol 

| Name of company: | | Boehringer Ingelheim | |
|---|---|---|---|
| Name of finished product: | | Not applicable | |
| Name of active ingredient: | | Xentuzumab (BI 836845) | |
| Protocol date: | Trial number: | | Revision date: |
| 30 Nov 2016 | 1280.18 | | 04 Mar 2022 |
| | To determine the maximum tolerated dose (MTD) / recomment phase II dose (RP2D) of xentuzumab in combination value abemaciclib with or without hormonal therapy (letrozole, anastrozoful vestrant). Expansion cohorts E, F, D1 and D2: To assess the anti-tumour activity of xentuzumab in combination value abemaciclib in patients with non-small cell lung cancer (cohort E assess the anti-tumour activity of the triplet combination xentuzumabemaciclib and ful vestrant in patients with locally advancementastatic, HR+ breast cancer who have progressed following paromatase inhibitor therapy and prior CDK4/6 inhibitor treatmal (cohort F), and to assess anti-tumor activity of the triplet combination xentuzumab, abemaciclib and ful vestrant in patients with local advanced/metastatic HR+ breast cancer visceral disease (Cohort or non-visceral disease (Cohort D2) who have progressed followendocrine therapy. Exploratory Objective: To expand the understanding of the study drug and the disease explorative biomarkers will be measured and analysed. The standard combination of the study drug and the disease explorative biomarkers will be measured and analysed. | | ab in combination with g cancer (cohort E), to abination xentuzumab, the locally advanced/ressed following prior/6 inhibitor treatment the triplet combination patients with locally all disease (Cohort D1) progressed following drug and the disease |
| Methodology: | Prospective, open | analyses are hypothesis generating. Prospective, open-label, non-randomised, multiple dose finding, phase Ib study, followed by expansion cohorts | |

c09049566-10 Trial Protocol 

| Name of company: | | Boehringer Ingelheim | |
|---|---|---|---|
| Name of finished pro | duct: | Not applicable | |
| Name of active ingredient: | | Xentuzumab (BI 836845) | |
| Protocol date: | Trial number: | | Revision date: |
| 30 Nov 2016 | 1280.18 | | 04 Mar 2022 |
| | Cohort A: will ide xentuzumab/abentumours. Cohorts B, C & D the xentuzumab/a of letrozole OR arin postmenopausa hormone receptor Expansion cohort E: will fur preliminary effica a single-arm dose patients. Cohort F: will invocombination xentuarm expansion ground hormone receptor visceral disease w (aromatase inhibit Cohorts D1 and D | Dose finding cohorts: Cohort A: will identify the MTD/RP2D <sub>1</sub> of the xentuzumab/abemaciclib combination in patients with solid tumours. Cohorts B, C & D (dose finding): will identify the MTD/RP2D the xentuzumab/ abemaciclib combination on a background the of letrozole OR anastrozole OR fulvestrant (referred to as "trip in postmenopausal women with locally advanced/metastatic hormone receptor positive (HR+) breast cancer. Expansion cohorts: Cohort E: will further characterize safety, tolerability, PK, and preliminary efficacy of the xentuzumab/abemaciclib combination a single-arm dose expansion group of non-small cell lung cancer. | |
| No. of patients: | progressed following endocrine therapy (aromatase inhibitor or Selective Estrogen Receptor Modulator). N= approximately 148 Dose finding cohorts: Cohort A: approx. 12 evaluable patients Cohort B: approx. 12 evaluable patients | | |

| Name of company: Name of finished product: Name of active ingredient: | | Boehringer Ingelheim | |
|---|---|---|---|
| | | Not applicable | |
| | | Xentuzumab (BI 836845) | |
| Protocol date: Trial number: 1280.18 | | | Revision date:<br>04 Mar 2022 |
| total entered:<br>each treatment: | Cohort C: approx. 12 evaluable patients Cohort D (dose finding): approx. 12 evaluable patients Expansion cohorts: Cohort E: 20 evaluable patients with non-visceral disease Cohort D1: 30 evaluable patients with visceral disease Cohort D2: 30 evaluable patients with non-visceral disease Cohort D2: 30 evaluable patients with non-visceral disease Approximately 148 evaluable patients * Dose finding cohorts: Cohort A (xentuzumab + abemaciclib): ~12 evaluable patients Cohorts B, C, D (dose finding) (xentuzumab + abemaciclib + hormonal therapy): ~ 12 evaluable patients Cohort E (xentuzumab + abemaciclib): ~20 evaluable patients Cohort F (xentuzumab + abemaciclib + fulvestrant): evaluable patients with non-visceral disease Cohort D1: (xentuzumab + abemaciclib + fulvestrant 30 evaluable patients with visceral disease Cohort D2: (xentuzumab + abemaciclib + fulvestrant 30 evaluable patients with non-visceral disease | | ral disease di |
| Diagnosis : | Patients with advanced/metastatic solid tumours in Cohort A; non-small cell lung cancer in Cohort E; pre-/peri-/post- menopausal women with locally advanced/metastatic hormone receptor-positive HER2-negative breast cancer in Cohorts B, C, D (dose finding), an expansion cohorts F (with non-visceral disease), D1(with visceral disease) and D2 (with non-visceral disease). | | ost- menopausal<br>one receptor-positive<br>D (dose finding), and |
| Main criteria for inclusion: | (see section 3.3 fo | <u>r details)</u> | |

09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies c09049566-10

| Name of company: | | Boehringer Ingelheim | |
|---|---|---|---|
| Name of finished product: Name of active ingredient: | | Not applicable | |
| | | Xentuzumab (BI 836845) | |
| Protocol date: | Trial number: | | Revision date: |
| 30 Nov 2016 | 1280.18 | | 04 Mar 2022 |
| | <ul> <li>Male or fe only) at somethods or Patients will diagnosis of evaluable,</li> <li>Patients mintolerant for have no appropriate</li> <li>Life expect</li> <li>Cohort B, C, D (or Patient must be who have some part of the will be will</li></ul> | ative (local lab results at scre | O years for Japan ase highly effective cally confirmed c, measurable or so or have been after clinical benefit, e as deemed as deemed as deemed as deemed as deemed as deemed as a confirmed confirm |

09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies c09049566-10

| Name of company: Name of finished product: Name of active ingredient: | | Boehringer Ingelheim | |
|---|---|---|---|
| | | Not applicable | |
| | | Xentuzumab (BI 836845) | |
| Protocol date:<br>30 Nov 2016 | Trial number: 1280.18 | | Revision date:<br>04 Mar 2022 |
| | suitable for Cohort B, correspond previous the allowed. It steroidal as exemestant For Cohorts D1, • Have either disease. • No more the metastation of the progression of the section of | CT (CT portion of diagnostic quality) and which for accurate repeated measurement. B, C, D (dose finding): Must be eligible for the conding hormonal therapy. For Cohorts B and C is treatment with fulvestrant or exemestane is all. For Cohort D (dose finding) prior therapy with a aromatase inhibitors (anastrozole, letrozole) of tane are permitted. 1. D2 and F only: ther measurable disease or non-measurable bond is the endocrine therapy for the tic disease is allowed. Sign on or after endocrine therapy is required (see the condition of the condition of the endocrine therapy is required (see the condition of the c | |
| Male or fe<br>only) at so | | ust be able to swallow oral cases be able to swallow oral cases. See the patients \$\ge\$ 18 years (\$\ge\$) creening willing and able to a per total of birth control per ICH M3 | 0 years for Japan |

09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies c09049566-10

| Name of company: | | Boehringer Ingelheim | |
|---|---|---|---|
| Name of finished product | : | Not applicable | |
| Name of active ingredient: | | Xentuzumab (BI 836845) | |
| Protocol date: | Trial number: | | Revision date: |
| 30 Nov 2016 | 1280.18 | | 04 Mar 2022 |
| Protocol date: 30 Nov 2016 Histologic IV NSCLC The partice chemother inappropri physician) prior chem OR must be standard so epidermal (EGFR-TK inhibitors in either EGF Prior targe permitted. Have meast Exclusion Criterial All cohorts: Any docur of malignate years prior cell carcine cervix or do in opinion Prior anti-therapy, and any investing myelosupp immunoth. Prior anti-O | | ipant must have progressed at apy AND immunotherapy (unate candidates for immunother AND have received 1 or a material of a district and and a district and a district and an application of the judged by the physician as econd-line chemotherapy. Prigrowth factor receptor-tyrosis (II) and anaplastic lymphoma is mandatory in participants of AI ting agents and neoadjuvant/a sureable disease per RECIST | After platinum-based calculated by their treating aximum of 2 other aximum of 2 other and treating aximum of 2 other and treating aximum of 2 other are metastatic disease ineligible for further or treatment with the kinase inhibitor kinase (ALK) whose tumours have LK translocations. Endjuvant therapies are adjuvant therapies are alignancy or history ander study, within 3 intely treated basal sinoma of uterine and treation can anticancer agents, or (14 days for non-tikes for the trial drugs. |

09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies c09049566-10

| Name of company: Name of finished product: Name of active ingredient: | | Boehringer Ingelheim | |
|---|---|---|---|
| | | Not applicable | |
| | | Xentuzumab (BI 836845) | - |
| Protocol date: | Trial number: | | Revision date: |
| 30 Nov 2016 | 1280.18 | | 04 Mar 2022 |
| | when it was Unresolved CTCAE grages neuropathy Previous transition of the compression of | otherapy to ≥25% of bone may as received different related toxicity for ade 1 at study entry (except to grade 1 at study entry (except to grade 1 at study entry (except to grade 2 and along reatment with IGF-1R target to the uncontrolled or symptom to gradient symptoms, cerebrough entry clinical symptoms, cerebrough entry of CNS monare eligible if they have begung to gradiotherapy, stereotactic estable, off anticonvulsants and extincts with brain metastases to tomatic, completed radiotherare on a stable dose of steroide not eligible if they have sponorts D1, D2 and F). The bone marrow reserve or organg renal disease including globyndrome, Fanconi Syndrome of swallow the product, or present of the product, or present of the product | from prior therapy of > for stable sensory becia). ing compounds. matic CNS metastases, singeal disease, as al oedema, and/or etastases or cord een definitively surgery) and are ad steroids for at least s are eligible if they rapy for at least 4 ds for at least 4 weeks. inal cord compression gan function omerulonephritis, e or renal tubular ic GI diseases, evious significant dequate absorption of ade 2 or higher attrolled Type II |

| Name of company: Name of finished product: Name of active ingredient: | | Boehringer Ingelheim | |
|---|---|---|---|
| | | Not applicable | |
| | | Xentuzumab (BI 836845) | |
| Protocol date: | Trial number: | | Revision date: |
| 30 Nov 2016 | 1280.18 | | 04 Mar 2022 |
| and Nov 2016 effusions ( lymphanging metastases) Prior hema Have had initial dose surgery du Have a per syncope of (including ventricular with contretreatment at treatment at the Have active [IV] antibite treatment) Patients we with basel Patients no cannot be For Cohorts D1, Have recent neoadjuvate everolimus only: priore excluded. Patients we metastasis Have initiate | | atis, and over 50% of liver involutions. atopoietic stem cell or bone major surgery (excluding biogue of any of the study drugs or tring study participation. Is conal history of any of the fole of cardiovascular etiology, ventually but not limited to ventricular fibrillation), or sudden cardial colled atrial fibrillation for >30 are eligible. It is bacterial or fungal (that is, and/or known viral infection in the discount of the seline of the selline of the seline of the selline | parrow transplant psy) < 28 days of the planned major archythmia tachycardia and ac arrest. Subjects days prior to study requiring intravenous tiating study allowed are areast. Subjects and action of the planned major to study requiring intravenous tiating study and placemia or patients at inhibitors/inducers pendix 10.1) anotherapy (except for allowestrant, or cohorts D1 and D2 respectively in the property of the planned property of the planned property of the property of the planned property of the plan |

| Name of company: Name of finished product: Name of active ingredient: | | Boehringer Ingelheim | |
|---|---|---|---|
| | | Not applicable | |
| | | Xentuzumab (BI 836845) | |
| Protocol date: | Trial number: | | Revision date: |
| 30 Nov 2016 | 1280.18 | | 04 Mar 2022 |
| Test product(s): | Xentuzumab (Boe<br>Abemaciclib (LY) | hringer Ingelheim): IGF-1/-2<br>2835219; (CDK 4/6 inl | |
| dose: | * Cohort A: starting dose is 1000 mg iv once weekly for xentuzumab and 150 mg every 12 hours for abemaciclib * Cohorts B, C and D (dose finding): MTD <sub>1</sub> /RP2D <sub>1</sub> of xentuzumab in combination with abemaciclib as determined cohort A, plus letrozole (cohort B), anastrozole (Cohort C) or fulvestrant (cohort D). * Expansion cohorts: * Cohort E: MTD <sub>1</sub> /RP2D <sub>1</sub> of xentuzumab in combination with abemaciclib as determined in cohort A. * Cohorts F, D1 and D2: MTD <sub>4</sub> /RP2D <sub>4</sub> of the triplet combination xentuzumab, abemaciclib and fulvestrant as determined in | | r abemaciclib RP2D <sub>1</sub> of lib as determined in zole (Cohort C) or combination with |
| mode of<br>administration: | | avenously, weekly dosing | hours |
| Background endocrine therapy: | Abemaciclib: oral, continuous dosing every 12 hours Letrozole, anastrozole, fulvestrant | | |
| dose: | Letrozole/anastrozole/fulvestrant at standard doses | | |
| mode of administration: | Letrozole, anastrozole, fulvestrant standard mode of administration | | |
| Duration of treatment: | | be given until disease progre ion or consent withdrawal. | ssion, intolerability of |
| | Abemaciclib will be given until disease progression, intolerability of the study medication or consent withdrawal. | | |
| Endpoints | Primary endpoints: | | |

| Name of company: Name of finished product: | | Boehringer Ingelheim | |
|---|---|---|---|
| | | Not applicable | |
| Name of active ingred | dient: | Xentuzumab (BI 836845) | _ |
| Protocol date: | Trial number: | | Revision date: |
| 30 Nov 2016 | 1280.18 | | 04 Mar 2022 |
| | * Number of par (first 28-day c For expansion col* * Objective resp For cohorts D1 an * PFS rate at 18 For expansion col* * Disease control RECIST 1.1) Secondary endporation of each expansion * No secondary For each expansion * Disease control RECIST 1.1) (* Time to object * Duration of ob * Duration of di * Progression-fr* | Number of patients with DLT during the MTD evaluation por (first 28-day cycle) For expansion cohort E: * Objective response (CR, PR per RECIST 1.1) For cohorts D1 and D2: * PFS rate at 18 month For expansion cohort F: * Disease control (CR, PR, SD lasting at least 24 weeks per RECIST 1.1) Secondary endpoints: For each dose finding cohorts A, B, C and D: * No secondary endpoint For each expansion cohorts E, F, D1 and D2: * Disease control (CR, PR, SD lasting at least 24 weeks per RECIST 1.1) (only for Cohorts D1, D2 and E) * Time to objective response * Duration of disease control | |
| Safety criteria: | the National Canc | Objective response (only for Cohorts D1, D2 and F) Incidence and severity of reported AEs. AEs will be assessed using the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version 4.03 (R10-4848) | |

c09049566-10 Trial Protocol


| Name of company: | | Boehringer Ingelheim | |
|---|---|---|---|
| Name of finished produ | ect: | Not applicable | |
| Name of active ingredie | ent: | Xentuzumab (BI 836845) | |
| Protocol date: | Trial number: | | Revision date: |
| 30 Nov 2016 | 1280.18 | | 04 Mar 2022 |
| Statistical methods: | For dose finding of by a Bayesian Log | each dose finding cohorts and<br>alysed using descriptive statistic<br>cohorts, inter-patient dose (de<br>gistic Regression Model (BLI | stics)escalation is guided RM) with overdose |
| | of parameters will BLRM. At the end | e fitted to binary toxicity out<br>be updated as data are accurated of each dose finding, the toxill be calculated to determine | nulated using the xicity probability at |

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### FLOW CHART - COHORT A (SOLID TUMOURS)

| Study period | Screening (a) | | | | EOTV (c) | FU<br>(d) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | SCR | | Cou | se 1 | | Co | ourse 2 | onwa | rds | | |
| Visits (V) | Screening | 1 | 2 | 3 | 4 | 1 | 2 | 3 | 4 | | |
| Days | Within 28d<br>before<br>C1V1 | 1 | 8 ±1 | 15<br>±1 | 22±1 | 1<br>±2 | 8<br>±2 | 15<br>±2 | 22<br>±2 | Within 7d after last drug intake | 42 +7d<br>after<br>last<br>drug<br>intake |
| Informed consent (1) | X | | | | | | | | | | |
| Demographics | X | | | | | | | | | | |
| Medical history | X | | | | | | | | | | |
| Inclusion/exclusion criteria (2) | X (2) | X (2) | | | | | | | | | |
| Physical exam (3) | X | X | | | | X | | | | X | X |
| Height | X | | | | | | | | | | |
| Body weight | X | X | | | | X | | | | X | X |
| Vital signs (4) | X | X | X | X | X | X | | | | X | X |
| ECOG performance status | X | X | | | | X | | | | X | X |
| 12-lead ECG<br>(triplicate) (5) | X | X | | X | | X | | X | | X | X |
| Safety lab (6) | X | X | X | X | X | X | | X<br>(7) | | X | X |
| Archival tumour tissue collection (8) | X | | | | | | | | | | |
| Blood sample for biomarkers (9) | X | X | X | | | X | | | | X | X |
| Pharmacokinetics (10) | | X | X | | | X | | | | X | X |
| Pharmacogenomics<br>and cfDNA (11) | | X | | | | X<br>(12) | | | | X | |
| PGx Plasma -exosomal<br>RNA (13) | | X | | X | | X | | | | X | |
| DNA banking (14) | | X | | | | | | | | | |
| Immunogenicity (ADA) (15) | | X | X | | | X | | | | X | X |
| Tumour assessment<br>and bone scan by<br>RECIST 1.1 (16) | X | | | | | X<br>(16) | | | | X | |
| Adverse event | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant therapy | X | X | X | X | X | X | X | X | X | X | X |
| Abemaciclib dispensation (17) | | X | | | | X | | | | | |
| Xentuzumab i.v. (17) | | X | X | X | X | X | X | X | X | | |
| Compliance check abemaciclib (18) | | | | | | X | | | | X | |
| Termination of trial medication | | | | | | | | | | X | |
| Completion of the study participation | | | | | | | | | | | X |

a Screening: The screening visit should be performed within 28 days prior to first drug administration (C1V1). Safety lab at the screening assessment can serve as the C1V1 assessment if performed within 72 hours before the first treatment and does not need to be repeated

b Treatment courses: All courses are 4 weeks in duration (28 days). All subsequent visit dates should be calculated based on Course 1 Visit 1 date. One or more visits can be skipped in case of treatment interruption. Patients may continue on treatment until the criteria for stopping medication are met (see Section 3.3.4). A duration of approximately 6 cycles is expected.

c09049566-10

Trial Protocol


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- c EOTV: End of Treatment visit. If the decision to permanently discontinue all study treatments is taken during a scheduled visit, the End Of Treatment Visit (EOTV) should be performed instead of the scheduled visit (within 7 calendar days after last drug administration)
- d FU: All patients should have a follow-up visit 42 days (+7days) after the permanent discontinuation of the study drugs
- 1. Written informed consent must be obtained before any protocol specific screening assessment is performed
- 2. In/Exclusion criteria must be checked at screening and ensured before study medication has been firstly administered.
- 3. Physical exam: includes a thorough cardiopulmonary, abdominal and lymph node exam and an assessment of the mental and neurological status
- 4. Vital signs: includes respiratory rate, pulse, temperature and blood pressure
- 5. 12-lead ECG: 12-Lead resting electrocardiograms (ECG) are recorded locally and in triplicate. ECG will be performed at Screening, EOTV and FU visit. ECG will be repeated at Visit 1/Day 1, and Visit 3/Day 15 of Course 1, 2, 3; and at Visit 1/Day 1 of Courses 6,9,12, etc. ECG should be performed prior to xentuzumab infusion.
- 6. Safety labs: includes haematology (CBC), coagulation, negative serum pregnancy test for women with childbearing potential and biochemistry. Urinalysis only at screening and EOTV. Fasting blood test is required for metabolic panels. See <a href="Section 5.3.3">Section 5.3.3</a> for detail. Safety lab can be performed one day prior to the scheduled test. Unscheduled safety lab should be performed if clinically indicated and documented in the eCRF
- 7. For course 2 only
- 8. Archival tumour tissue collection: the most recent/appropriate archival tumour tissue must be collected prior to the start of trial treatment. Refer to <u>Appendix 10.3</u> for tissue requirements
- 9. Blood soluble biomarkers: for detailed sampling time schedule, refer to Section 5.5 and Appendix 10.2.1
- 10. Pharmacokinetics: Course 1, Course 2-12, 15, 18, EOTV and FU visits. For detailed PK sampling time schedule, refer to Section 5.4.1 and Appendix 10.2.1 for cohorts A, B, C and D
- 11. Pharmacogenomics and cfDNA. See Section 5.5 for more details on collection time points. Briefly, one blood sample to isolate genomic DNA will be obtained at C1V1 before treatment. 3 plasma samples will be collected to isolate circulating nucleic acids (e.g. cfDNA) from plasma: at C1V1 before treatment, at C3V1 and at the EOTV.
- 12. For course 3 only
- 13. PGx Plasma: blood samples will be collected before treatment on C1V1, C1V3 (Day 15), C2V1, C3V1 and beyond, and at the EOTV. Samples will be used to evaluate exosomal RNA.
- 14. DNA banking: For details please refer to Section 5.5.1.
- 15. Immunogenicity (ADA): On days when xentuzumab is dosed and EOTV and FU visit at time points specified in Flow Chart and Appendix 10.2.1, ADA samples are to be collected prior to xentuzumab infusion. ADA samples must be collected at Course 1, Course 2-12, 15, 18, at EOTV and at the FU visit. For detailed sampling schedule, refer to Appendix 10.2.1
- 16. Tumour assessments should include CT or MRI scans of the chest, abdomen and pelvis, and, if clinically indicated, any other known or suspected sites of disease (e.g. breast, neck, brain etc.) accordingly to RECIST 1.1. After study entry, all lesions identified as target and non-target lesions during the screening should be followed up at all pre-specified imaging time points. The same radiographic procedure must be used throughout the study. Bone scans must be performed at screening (see Section 5.2 for more detail).
  - Assessment will be performed at the following time points until progression/start of further treatment (tumour assessments after start of xentuzumab should be performed no more than 7 days prior to the scheduled tumour assessment date up to week 48 AND no more than 14 days prior to the scheduled tumour assessment date after week 48):
    - At screening (within 28 days prior to starting of treatment)
    - Every 8 weeks (±7days): during week 8 (49-63 days after start of xentuzumab), during week 16 (105-119 days after start of xentuzumab), during week 24 (161-175 days after start of xentuzumab), during week 32 (217-231 days after start of xentuzumab), during week 40 (273-287 days after start of xentuzumab), during week 48 (329-343 days after start of xentuzumab)
    - Every 12 weeks after week 48 (±7days) (e.g. during week 60 (406-434 days after start of xentuzumab), during week 72 (490-518 days after start of xentuzumab), etc.)
      - In the event of an interruption/delay to treatment, the tumour assessment schedule should not be changed.

Except in case of discontinuation from treatment due to progression, tumour assessment at EOTV is not necessary if the previous evaluation was done within 4 weeks of EOTV

- Unscheduled scan based on the investigator's judgement is allowed and should also be documented in eCRF
- 17. Abemaciclib and xentuzumab should be dispensed through IRT. Patient's screening, all drug dispensation visits and EOTV will be collected in the IRT system
- 18. Compliance check: on Day 1 of every course starting on course 2 and at EOTV

c09049566-10

#### **Trial Protocol**


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## FLOW CHART – COHORT B (BC TRIPLET WITH LETROZOLE)

| Study period | Screening (a) | | | | EOTV (c) | FU (d) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | SCR | | Cou | rse 1 | | С | ourse : | 2 onw | ards | | |
| Visits (V) | Screening | 1 | 2 | 3 | 4 | 1 | 2 | 3 | 4 | | |
| Days | Within<br>28d before<br>C1V1 | 1 | 8<br>±1 | 15<br>±1 | 22<br>±1 | 1<br>±2 | 8<br>±2 | 15<br>±2 | 22<br>±2 | Within 7d<br>after last<br>drug<br>intake | 42 +7d<br>after last<br>drug<br>intake |
| Informed consent(1) | X | | | | | | | | | | |
| Demographics | X | | | | | | | | | | |
| Medical history | X | | | | | | | | | | |
| Inclusion/exclusion criteria (2) | X (2) | X (2) | | | | | | | | | |
| Physical exam (3) | X | X | | | | X | | | | X | X |
| Height | X | | | | | | | | | | |
| Body weight | X | X | | | | X | | | | X | X |
| Vital signs (4) | X | X | X | X | X | X | | | | X | X |
| ECOG performance status | X | X | | | | X | | | | X | X |
| 12-lead ECG (triplicate) (5) | X | X | | X | | X | | X | | X | X |
| Safety lab (6) | X | X | X | X | X | X | | X<br>(7) | | X | X |
| Archival tumour tissue collection (8) | X | | | | | | | | | | |
| Blood sample for biomarkers (9) | X | X | X | | | X | | | | X | X |
| Pharmacokinetics (10) | | X | X | | | X | | | | X | X |
| Pharmacogenomics and cfDNA (11) | | X | | | | X<br>(12) | | | | X | |
| PGx Plasma -exosomal<br>RNA (13) | | X | | X | | X | | | | X | |
| DNA banking (14) | | X | | | | | | | | | |
| Immunogenicity (ADA) (15) | | X | X | | | X | | | | X | X |
| Tumour assessment and bone scan by RECIST 1.1 (16) | X | | | | | X<br>(16) | | | | X | |
| Adverse event | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant therapy | X | X | X | X | X | X | X | X | X | X | X |
| Abemaciclib and letrozole dispensation (17) | | X | | | | X | | | | | |
| Xentuzumab i.v. (17) | | X | X | X | X | X | X | X | X | | |
| Compliance check abemaciclib and | | Λ | Λ | Α | Λ | X | Λ | Α | Λ | X | |
| letrozole (18) Termination of trial medication | | | | | | | | | | X | |
| Completion of the study participation | | | | | | | | | | | X |

a Screening: The screening visit should be performed within 28 days prior to first drug administration (C1V1). Safety lab at the screening assessment can serve as the C1V1 assessment if performed within 72 hours before the first treatment and does not need to be repeated

# Boehringer Ingelheim BI Trial No.: 1280.18

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- b Treatment courses: All courses are 4 weeks in duration (28 days). All subsequent visit dates should be calculated based on Course 1 Visit 1 date. One or more visits can be skipped in case of treatment interruption. Patients may continue on treatment until the criteria for stopping medication are met (see Section 3.3.4). A duration of approximately 12 cycles is expected.
- c EOTV: End of Treatment visit. If the decision to permanently discontinue all study treatments is taken during a scheduled visit, the End Of Treatment Visit (EOTV) should be performed instead of the scheduled visit (within 7 calendar days after last drug administration)
- d FU: All patients should have a follow-up visit 42 days (+7days) after the permanent discontinuation of the study drugs
- 1. Written informed consent must be obtained before any protocol specific screening assessment is performed
- 2. In/Exclusion criteria must be checked at screening and ensured before study medication has been firstly administered.
- 3. Physical exam: includes a thorough cardiopulmonary, abdominal and lymph node exam and an assessment of the mental and neurological status
- 4. Vital signs: includes respiratory rate, pulse, temperature and blood pressure
- 5. 12-lead ECG: 12-Lead resting electrocardiograms (ECG) are recorded locally and in triplicate. ECG will be performed at Screening, EOTV and FU visit. ECG will be repeated at Visit 1/Day 1, and Visit 3/Day 15 of Course 1, 2, 3; and at Visit 1/Day 1 of Courses 6,9,12, etc. ECG should be performed prior to xentuzumab infusion.
- 6. Safety labs: includes haematology (CBC), coagulation, negative serum pregnancy test for women with childbearing potential and biochemistry. Urinalysis only at screening and EOTV. Fasting blood test is required for metabolic panels. See Section 5.3.3 for detail. Safety lab can be performed one day prior to the scheduled test. Unscheduled safety lab should be performed if clinically indicated and documented in the eCRF
- 7. For course 2 only
- 8. Archival tumour tissue collection: the most recent/appropriate archival tumour tissue must be collected prior to the start of trial treatment. Refer to <a href="Appendix 10.3">Appendix 10.3</a> for tissue requirements
- 9. Blood soluble biomarkers: for detailed sampling time schedule, refer to Section 5.5 and Appendix 10.2.1
- 10. Pharmacokinetics: Course 1, course 2-12, 15, 18, EOTV and FU visits. For detailed PK sampling time schedule, refer to Section 5.4.1 and Appendix 10.2.1 for cohorts A, B, C and D
- 11. Pharmacogenomics and cfDNA See Section 5.5 for more details about collection timepoints. Briefly, one blood sample to isolate genomic DNA will be obtained at C1V1 before treatment. 3 plasma samples will be collected to isolate circulating nucleic acids (e.g. cfDNA) from plasma: at C1V1 before treatment, at C3V1 and at the EOTV.
- 12. For course 3 only
- 13. PGx Plasma: blood samples will be collected before treatment on C1V1, C1V3 (Day 15), C2V1, C3V1 and beyond and at the EOTV. Samples will be used to evaluate exosomal RNA.
- 14. DNA banking: For details please refer to Section 5.5.1.
- 15. Immunogenicity (ADA): On days when xentuzumab is dosed and EOTV and FU visit at time point specified in the Flow Chart and Appendix 10.2.1, ADA samples are to be collected prior to xentuzumab infusion. ADA samples must be collected at Course 1, course 2-12, 15, 18, at EOTV and at the FU visit. For detailed sampling schedule, refer to Appendix 10.2.1
- 16. Tumour assessments should include CT or MRI scans of the chest, abdomen and pelvis, and, if clinically indicated, any other known or suspected sites of disease (e.g. breast, neck, brain etc.) accordingly to RECIST 1.1. After study entry, all lesions identified as target and non-target lesions during the screening should be followed up at all prespecified imaging time points. The same radiographic procedure must be used throughout the study. Bone scans must be performed at screening (see Section 5.2 for more detail).

Assessment will be performed at the following time points until progression/start of further treatment (tumour assessments after start of xentuzumab should be performed no more than 7 days prior to the scheduled tumour assessment date up to week 48 AND no more than 14 days prior to the scheduled tumour assessment date after week 48):

- At screening (within 28 days prior to starting of treatment)
- Every 8 weeks (±7days): during week 8 (49-63 days after start of xentuzumab), during week 16 (105-119 days after start of xentuzumab), during week 24 (161-175 days after start of xentuzumab), during week 32 (217-231 days after start of xentuzumab), during week 40 (273-287 days after start of xentuzumab), during week 48 (329-343 days after start of xentuzumab)
- Every 12 weeks after week 48 (±7days) (e.g. during week 60 (406-434 days after start of xentuzumab), during week 72 (490-518 days after start of xentuzumab), etc.)
  - In the event of an interruption/delay to treatment, the tumour assessment schedule should not be changed.

Except in case of discontinuation from treatment due to progression, tumour assessment at EOTV is not necessary if the previous evaluation was done within 4 weeks of EOTV

- Unscheduled scan based on the investigator's judgement is allowed and should also be documented in eCRF
- 17. Abemaciclib, letrozole (in certain countries) and xentuzumab should be dispensed through IRT. Patient's screening, all drug dispensation visits and EOTV will be collected in the IRT system
- 18. Compliance check: on Day 1 of every course starting at course 2 and at EOTV

c09049566-10

#### **Trial Protocol**


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## FLOW CHART – COHORT C (BC TRIPLET WITH ANASTROZOLE)

| Study period | Screening (a) | | | | EOTV (c) | FU<br>(d) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | SCR | | Cou | rse 1 | | Co | urse 2 | onwa | rds | | |
| Visits (V) | Screening | 1 | 2 | 3 | 4 | 1 | 2 | 3 | 4 | | |
| Days | Within<br>28d before<br>C1V1 | 1 | 8<br>±1 | 15<br>±1 | 22<br>±1 | 1<br>±2 | 8<br>±2 | 15<br>±2 | 22<br>±2 | Within 7d after last drug intake | 42 +7d<br>after last<br>drug<br>intake |
| Informed consent(1) | X | | | | | | | | | | |
| Demographics | X | | | | | | | | | | |
| Medical history | X | | | | | | | | | | |
| Inclusion/exclusion criteria (2) | X (2) | X<br>(2) | | | | | | | | | |
| Physical exam (3) | X | X | | | | X | | | | X | X |
| Height | X | | | | | | | | | | |
| Body weight | X | X | | | | X | | | | X | X |
| Vital signs (4) | X | X | X | X | X | X | | | | X | X |
| ECOG performance status | X | X | | | | X | | | | X | X |
| 12-lead ECG (triplicate) (5) | X | X | | X | | X | | X | | X | X |
| Safety lab (6) | X | X | X | X | X | X | | X<br>(7) | | X | X |
| Archival tumour tissue collection (8) | X | | | | | | | | | | |
| Blood sample for biomarkers (9) | X | X | X | | | X | | | | X | X |
| Pharmacokinetics (10) | | X | X | | | X | | | | X | X |
| Pharmacogenomics and cfDNA (11) | | X | | | | X<br>(12) | | | | X | |
| PGx Plasma -exosomal<br>RNA (13) | | X | | X | | X | | | | X | |
| DNA banking (14) | | X | | | | | | | | | |
| Immunogenicity (ADA) (15) | | X | X | | | X | | | | X | X |
| Tumour assessment and bone scan by RECIST 1.1 (16) | X | | | | | X<br>(16) | | | | X | |
| Adverse event | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant therapy | X | X | X | X | X | X | X | X | X | X | X |
| Abemaciclib and anastrozole dispensation (17) | | X | | | | X | | | | | |
| Xentuzumab i.v. (17) | | X | X | X | X | X | X | X | X | | |
| Compliance check abemaciclib and anastrozole (18) | | 21 | 71 | 71 | | X | 21 | 21 | 21 | X | |
| Termination of trial medication | | | | | | | | | | X | |
| Completion of the study participation | | | | | | | | | | | X |

a Screening: The screening visit should be performed within 28 days prior to first drug administration (C1V1). Safety lab at the screening assessment can serve as the C1V1 assessment if performed within 72 hours before the first treatment and does not need to be repeated

# Boehringer Ingelheim BI Trial No.: 1280.18

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- b Treatment courses: All courses are 4 weeks in duration (28 days). All subsequent visit dates should be calculated based on Course 1 Visit 1 date. One or more visits can be skipped in case of treatment interruption. Patients may continue on treatment until the criteria for stopping medication are met (see Section 3.3.4). A duration of approximately 12 cycles is expected.
- c EOTV: End of Treatment visit. If the decision to permanently discontinue all study treatments is taken during a scheduled visit, the End Of Treatment Visit (EOTV) should be performed instead of the scheduled visit (within 7 calendar days after last drug administration)
- d FU: All patients should have a follow-up visit 42 days (+7days) after the permanent discontinuation of the study drugs
- 1. Written informed consent must be obtained before any protocol specific screening assessment is performed
- 2. In/Exclusion criteria must be checked at screening and ensured before study medication has been firstly administered.
- 3. Physical exam: includes a thorough cardiopulmonary, abdominal and lymph node exam and an assessment of the mental and neurological status
- 4. Vital signs: includes respiratory rate, pulse, temperature and blood pressure
- 5. 12-lead ECG: 12-Lead resting electrocardiograms (ECG) are recorded locally and in triplicate. ECG will be performed at Screening, EOTV and FU visit. ECG will be repeated at Visit 1/Day 1, and Visit 3/Day 15 of Course 1, 2, 3; and at Visit 1/Day 1 of Courses 6,9,12, etc. ECG should be performed prior to xentuzumab infusion.
- 6. Safety labs: includes haematology (CBC), coagulation, and negative serum pregnancy test for women with childbearing potential and biochemistry. Urinalysis only at screening and EOTV. Fasting blood test is required for metabolic panels. See Section 5.3.3 for detail. Safety lab can be performed one day prior to the scheduled test. Unscheduled safety lab should be performed if clinically indicated and documented in the eCRF
- 7. For course 2 only
- 8. Archival tumour tissue collection: the most recent/appropriate archival tumour tissue must be collected prior to the start of trial treatment. Refer to <u>Appendix 10.3</u> for tissue requirements
- 9. Blood soluble biomarkers: for detailed sampling time schedule, refer to Section 5.5 and Appendix 10.2.1
- 10. Pharmacokinetics: Course 1, Course 2-12, 15 and 18, EOTV and FU visits. For detailed PK sampling time schedule, refer to Section 5.4.1 and Appendix 10.2.1 for cohorts A, B, C and D
- 11. Pharmacogenomics and cfDNA See Section 5.5 for more details about collection timepoints. Briefly, one blood sample to isolate genomic DNA will be obtained at C1V1 before treatment. 3 plasma samples will be collected to isolate circulating nucleic acids (e.g. cfDNA) from plasma: at C1V1 before treatment, at C3V1 and at the EOTV.
- 12. For course 3 only
- 13. PGx Plasma: blood samples will be collected before treatment on C1V1, C1V3 (Day 15), C2V1, C3V1 and beyond, and at the EOTV. Samples will be used to evaluate exosomal RNA.
- 14. DNA banking: For details please refer to Section 5.5.1.
- 15. Immunogenicity (ADA): On days when xentuzumab is dosed and EOTV and FU visit at time points specified in Flow Chart and Appendix 10.2.1, ADA samples are to be collected prior to xentuzumab infusion. ADA samples must be collected at Course 1, Course 2-12, 15 and 18, at EOTV and at the FU visit. For detailed sampling schedule, refer to Appendix 10.2.1
- 16. Tumour assessments should include CT or MRI scans of the chest, abdomen and pelvis, and, if clinically indicated, any other known or suspected sites of disease (e.g. breast, neck, brain etc.) accordingly to RECIST 1.1. After study entry, all lesions identified as target and non-target lesions during the screening should be followed up at all prespecified imaging time points. The same radiographic procedure must be used throughout the study. Bone scans must be performed at screening (see Section 5.2 for more detail).

Assessment will be performed at the following time points until progression/start of further treatment (tumour assessments after start of xentuzumab should be performed no more than 7 days prior to the scheduled tumour assessment date up to week 48 AND no more than 14 days prior to the scheduled tumour assessment date after week 48):

- At screening (within 28 days prior to starting of treatment)
- Every 8 weeks (±7days): during week 8 (49-63 days after start of xentuzumab), during week 16 (105-119 days after start of xentuzumab), during week 24 (161-175 days after start of xentuzumab), during week 32 (217-231 days after start of xentuzumab), during week 40 (273-287 days after start of xentuzumab), during week 48 (329-343 days after start of xentuzumab)
- Every 12 weeks after week 48 (±7days) (e.g. during week 60 (406-434days after start of xentuzumab), during week 72 (490-518 days after start of xentuzumab), etc.)
  - In the event of an interruption/delay to treatment, the tumour assessment schedule should not be changed.

Except in case of discontinuation from treatment due to progression, tumour assessment at EOTV is not necessary if the previous evaluation was done within 4 weeks of EOTV

- Unscheduled scan based on the investigator's judgement is allowed and should also be documented in eCRF
- 17. Abemaciclib, anastrozole (in certain countries) and xentuzumab should be dispensed through IRT. Patient's screening, all drug dispensation visits and EOTV will be collected in the IRT system
- 18. Compliance check: on Day 1 of every course starting at course 2 and at EOTV

c09049566-10

### **Trial Protocol**


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# FLOW CHART – COHORT D – DOSE FINDING (BC TRIPLET WITH **FULVESTRANT**)

| Study period | Screening (a) | Treatment Courses (b) | | | | | | | | | FU<br>(d) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | SCR | | Cou | rse 1 | (-) | Co | urse 2 | onwa | rds | (c) | () |
| Visits (V) | Screening | 1 | 2 | 3 | 4 | 1 | 2 | 3 | 4 | | |
| Days | Within 28d<br>before<br>C1V1 | 1 | 8 ±1 | 15<br>±1 | 22<br>±1 | 1 ±2 | 8<br>±2 | 15<br>±2 | 22<br>±2 | Within 7d after last drug intake | 42 +7d<br>after<br>last<br>drug<br>intake |
| Informed consent (1) | X | | | | | | | | | | |
| Demographics | X | | | | | | | | | | |
| Medical history | X | | | | | | | | | | |
| Inclusion/exclusion criteria (2) | X (2) | X (2) | | | | | | | | | |
| Physical exam (3) | X | X | | | | X | | | | X | X |
| Height | X | | | | | | | | | | |
| Body weight | X | X | | | | X | | | | X | X |
| Vital signs (4) | X | X | X | X | X | X | | | | X | X |
| ECOG performance status | X | X | | | | X | | | | X | X |
| 12-lead ECG (triplicate) (5) | X | X | | X | | X | | X | | X | X |
| Safety lab (6) | X | X | X | X | X | X | | X<br>(7) | | X | X |
| Archival tumour tissue collection (8) | X | | | | | | | | | | |
| Blood sample for biomarkers (9) | X | X | X | | | X | | | | X | X |
| Pharmacokinetics (10) | | X | X | | | X | | | | X | X |
| Pharmacogenomics and cfDNA (11) | | X | | | | X<br>(12) | | | | X | |
| PGx Plasma -exosomal<br>RNA (13) | | X | | X | | X | | | | X | |
| DNA banking (14) | | X | | | | | | | | | |
| Immunogenicity (ADA) (15) | | X | X | | | X | | | | X | X |
| Tumour assessment and bone scan by RECIST 1.1 (16) | X | | | | | X<br>(16) | | | | X | |
| Adverse event | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant therapy | X | X | X | X | X | X | X | X | X | X | X |
| Abemaciclib | | X | | | | X | | | | | |
| dispensation (17) | | | | | | | | | | | |
| Xentuzumab i.v. (17) | | X | X | X | X | X | X | X | X | | |
| Fulvestrant i.m. (17) | | X | | X | | X | | | | | |
| Compliance check abemaciclib (18) | | | | | | X | | | | X | |
| Termination of trial medication | | | | | | | | | | X | |
| Completion of the study participation | | | | | | | | | | | X |

Screening: The screening visit should be performed within 28 days prior to first drug administration (C1V1). Safety lab at the screening assessment can serve as the C1V1 assessment if performed within 72 hours before the first treatment and does not need to be repeated

# Boehringer Ingelheim BI Trial No.: 1280.18

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- b Treatment courses: All courses are 4 weeks in duration (28 days). All subsequent visit dates should be calculated based on Course 1 Visit 1 date. One or more visits can be skipped in case of treatment interruption. Patients may continue on treatment until the criteria for stopping medication are met (see Section 3.3.4). A duration of approximately 12 cycles is expected.
- c EOTV: End of Treatment visit. If the decision to permanently discontinue all study treatments is taken during a scheduled visit, the End Of Treatment Visit (EOTV) should be performed instead of the scheduled visit (within 7 calendar days after last drug administration)
- d FU: All patients should have a follow-up visit 42 days (+7days) after the permanent discontinuation of the study drugs
- 1. Written informed consent must be obtained before any protocol specific screening assessment is performed
- 2. In/Exclusion criteria must be checked at screening and ensured before study medication has been firstly administered
- 3. Physical exam: includes a thorough cardiopulmonary, abdominal and lymph node exam and an assessment of the mental and neurological status
- 4. Vital signs: includes respiratory rate, pulse, temperature and blood pressure
- 5. 12-lead ECG: 12-Lead resting electrocardiograms (ECG) are recorded locally and in triplicate. ECG will be performed at Screening, EOTV and FU visit. ECG will be repeated at Visit 1/Day 1, and Visit 3/Day 15 of Course 1, 2, 3; and at Visit 1/Day 1 of Courses 6,9,12, etc. ECG should be performed prior to xentuzumab infusion.
- 6. Safety labs: includes haematology (CBC), coagulation, negative serum pregnancy test for women with childbearing potential and biochemistry. Urinalysis only at screening and EOTV. Fasting blood test is required for metabolic panels. Baseline Local FSH and estradiol levels should be within 14 days of initial dose of study treatment. See Section 5.3.3 for detail. Safety lab can be performed one day prior to the scheduled test. Unscheduled safety lab should be performed if clinically indicated and documented in the eCRF
- 7. For course 2 only
- 8. Archival tumour tissue collection: the most recent/appropriate archival tumour tissue must be collected prior to the start of trial treatment. Refer to Appendix 10.3 for tissue requirements
- 9. Blood soluble biomarkers: for detailed sampling time schedule, refer to Section 5.5 and Appendix 10.2.1
- 10. Pharmacokinetics: Course 1, Course 2-12, 15, 18, EOTV and FU visits. For detailed PK sampling time schedule, refer to Section 5.4.1 and Appendix 10.2.1 for cohorts A, B, C and D
- 11. Pharmacogenomics and cfDNA See Section 5.5 for more details about collection timepoints. Briefly, one blood sample to isolate genomic DNA will be obtained at C1V1 before treatment. 3 additional blood samples will be collected to isolate circulating nucleic acids (e.g. cfDNA) from plasma: at C1V1 before treatment, at C3V1 and at the EOTV.
- 12. For course 3 only
- 13. PGx Plasma: blood samples will be collected before treatment on C1V1, C1V3 (Day 15), C2V1, C3V1 and beyond, and at the EOTV. Samples will be used to evaluate exosomal RNA.
- 14. DNA banking: For details please refer to Section 5.5.1.
- 15. Immunogenicity (ADA): On days when xentuzumab is dosed and EOTV and FU visit at time points specified in the Flow Chart and Appendix 10.2.1, ADA samples are to be collected prior to xentuzumab infusion. ADA samples must be collected at Course 1, Course 2-12, 15, 18, at EOTV and at the FU visit. For detailed sampling schedule, refer to Appendix 10.2.1
- 16. Tumour assessments should include CT or MRI scans of the chest, abdomen and pelvis, and, if clinically indicated, any other known or suspected sites of disease (e.g. breast, neck, brain etc.) accordingly to RECIST 1.1. After study entry, all lesions identified as target and non-target lesions during the screening should be followed up at all prespecified imaging time points. The same radiographic procedure must be used throughout the study. Bone scans must be performed at screening (see Section 5.2 for more detail).

Assessment will be performed at the following time points until progression/start of further treatment (tumour assessments after start of xentuzumab should be performed no more than 7 days prior to the scheduled tumour assessment date up to week 48 AND no more than 14 days prior to the scheduled tumour assessment date after week 48):

- At screening (within 28 days prior to starting of treatment)
- Every 8 weeks (±7days): during week 8 (49-63 days after start of xentuzumab), during week 16 (105-119 days after start of xentuzumab), during week 24 (161-175 days after start of xentuzumab), during week 32 (217-231 days after start of xentuzumab), during week 40 (273-287 days after start of xentuzumab), during week 48 (329-343 days after start of xentuzumab)
- Every 12 weeks after week 48 (±7days) (e.g. during week 60 (406-434 days after start of xentuzumab), during week 72 (490-518 days after start of xentuzumab), etc.)

In the event of an interruption/delay to treatment, the tumour assessment schedule should not be changed.

Except in case of discontinuation from treatment due to progression, tumour assessment at EOTV is not necessary if the previous evaluation was done within 4 weeks of EOTV

Unscheduled scan based on the investigator's judgement is allowed and should also be documented in eCRF

- 17. Abemaciclib, xentuzumab and fulvestrant (in certain countries) should be dispensed through IRT. Patient's screening, all drug dispensation visits and EOTV will be collected in the IRT system
- 18. Compliance check: on Day 1 of every course starting at course 2 and at EOTV

c09049566-10 Trial Protocol


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# FLOW CHART – COHORT E (NSCLC EXPANSION COHORT)

| Study period | Screening (a) | F | Run-i<br>(b) | n | | | | Treati | nent (c) | | | | | EOTV (d) | FU<br>(e) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | SCR | | R | | | C | ourse 1 | | | Cou | rse 2 on | ward | S | | |
| Visits (V) | Screenin<br>g | 1 | 2 | 3 | 1 | 2 | 3 | 4 | 1 | 1b | 2 | 3 | 4 | | |
| Days | Within<br>28d<br>before<br>Run-in<br>V1 | 9 | 2 | -<br>1 | 1 | 8<br>±<br>1 | 15±<br>1 | 22±<br>1 | 1<br>±2 | 4<br>±<br>1<br>(f) | 8<br>±2(g<br>) | 15<br>±<br>2 | 22±<br>2 | Withi<br>n 7d<br>after<br>last<br>drug<br>intake | 42<br>+7d<br>after<br>last<br>drug<br>intak<br>e |
| Informed consent (1) | X | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | |
| Medical history | X | 37 | | | | | | | | | | | | | |
| Inclusion/exclusio | | X | | | | | | | | | | | | | |
| n criteria (2) | X (2) | (2) | | | | | | | | | | | | | |
| Physical exam (3) | X | X | | | X | | | | X | | | | | X | X |
| Height | X | | | | | | | | | | | | | | |
| Body weight | X | X | | | X | | | | X | | | | | X | X |
| Vital signs (4) | X | X | X | X | X | X | X | X | X | | | | | X | X |
| Dispense Patient | | | | | | | | | | | | | | | |
| Diary (5) | | X | | | | | | X | | | | | | | |
| ECOG<br>performance<br>status | X | X | | | X | | | | X | | | | | X | X |
| 12-lead ECG | | | | | | | | | | | | | | | |
| (triplicate) (6) | X | | X | | X | | X | | X | | | X | | X | X |
| Safety lab (7) | X | X | | | X | X | X | X | X | | | X<br>(8 | | X | X |
| Archival tumour tissue collection (9) | X | | | | | | | | | | | | | | |
| Blood sample for biomarkers (10) | X | X | | | X | X | | | X | | | | | X | X |
| Pharmacokinetics (11) | | X | | X | X | X | | | X<br>* | X<br>(12) | X (12) | | | X | X |
| Pharmacogenomic s and cfDNA (13) | | X | | | X | | | | X<br>(14) | () | | | | X | |
| PGx Plasma -<br>exosomal RNA<br>(15) | | X | | | X | | X | | X | | | | | X | |
| DNA banking (16) | | X | | | | | | | | | | | | | |
| Immunogenicity (ADA) (17) | | X | | | X | X | | | X | | | | | X | X |
| Tumour assessment and bone scan by RECIST 1.1 (18) | X | | | | | | | | X<br>(18) | | | | | X | |
| Adverse event | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant therapy | X | X | | | X | X | X | X | X | | X | X | X | X | X |
| Abemaciclib | | | | | | | | | 1 | | | | | | |
| dispensation (19) | | X | | | X | | | | X | | | | | | |
| Xentuzumab i.v. (19) | | | | | X | X | X | X | X | | X | X | X | | |
| Compliance check abemaciclib (20) | | | | X | | | | | X | | | | | X | |

Boehringer Ingelheim BI Trial No.: 1280.18

c09049566-10

Trial Protocol


| Termination of trial medication | X | |
|---------------------------------|---|---|
| Completion of the | | v |
| study participation | | Λ |

- \* A 24 h sample is also required at C2V1D2 (see Appendix 10.2.2)
- Screening: The screening visit should be performed within 28 days prior to first drug administration (Run-in period). Safety lab at the screening assessment can serve as the Run-in Visit 1 assessment if performed within 72 hours before the first treatment and does not need to be repeated
- b Run in: Consists of 9 days. During the run-in period, patients should take daily abemaciclib treatment. At days with PK sampling, patients have to take their morning dose of abemaciclib in the hospital to allow proper PK sampling.
- c Treatment courses: All courses are 4 weeks in duration (28 days). All subsequent visit dates should be calculated based on Course 1 Visit 1 date. One or more visits can be skipped in case of treatment interruption. Patients may continue on treatment until the criteria for stopping medication are met (see Section 3.3.4). A duration of approximately 6 cycles is expected.
- d EOTV: End of Treatment visit. If the decision to permanently discontinue all study treatments is taken during a scheduled visit, the End Of Treatment Visit (EOTV) should be performed instead of the scheduled visit (within 7 calendar days after last drug administration)
- e FU: All patients should have a follow-up visit 42 days (+7days) after the permanent discontinuation of the study drugs
- f On course 2 only for PK purposes
- g No time window is applicable for course 2 when PK determinations are scheduled for the visit
- 1. Written informed consent must be obtained before any protocol specific screening assessment is performed
- 2. In/Exclusion criteria must be checked at screening and ensured before study medication has been firstly administered
- 3. Physical exam: includes a thorough cardiopulmonary, abdominal and lymph node exam and an assessment of the mental and neurological status
- 4. Vital signs: includes respiratory rate, pulse, temperature and blood pressure
- 5. A patient diary will be handed over to the patient at Run-In Visit 1 and at C1V4. Patients have to fill in this diary up to Run-In V3 and C2V1, respectively (see also Section 4.3 for a short description of the diary)
- 6. 12-lead ECG: 12-Lead resting electrocardiograms (ECG) are recorded locally and in triplicate. ECG will be performed at Screening, Run-in visit 2 Day -2, EOTV and FU visit. ECG will be repeated at Visit 1/Day 1, and Visit 3/Day 15 of Course 1, 2, 3; and at Visit 1/Day 1 of Courses 6,9,12, etc. ECG should be performed prior to xentuzumab infusion.
- 7. Safety labs: includes haematology (CBC), coagulation, negative serum pregnancy test for women with childbearing potential and biochemistry. Urinalysis only at screening and EOTV. Fasting blood test is required for metabolic panels. See <a href="Section 5.3.3">Section 5.3.3</a> for detail. Safety lab can be performed one day prior to the scheduled test. Unscheduled safety lab should be performed if clinically indicated and documented in the eCRF
- 8. For course 2 only
- 9. Archival tumour tissue collection: the most recent/appropriate archival tumour tissue must be collected prior to the start of trial treatment. Refer to <u>Appendix 10.3</u> for tissue requirements
- 10. Blood soluble biomarkers: for detailed sampling time schedule, refer to Section 5.5 and Appendix 10.2.2
- 11. Pharmacokinetics: to be collected at Run-In period as well as in treatment courses 1-12, 15, 18, EOTV and FU visit. For detailed PK sampling time schedule, refer to <a href="Section 5.4.1">Section 5.4.1</a> and <a href="Appendix 10.2.2">Appendix 10.2.2</a> for cohort E. Please note: At days of PK sampling of abemaciclib, patients have to take their morning dose in the hospital in order to allow for proper PK sampling
- 12. PK sampling at this visit only in course 2
- 13. Pharmacogenomics and cfDNA See Section 5.5 for more details on collection timepoints. Briefly, one blood sample to isolate genomic DNA will be obtained at Run-in V1 before treatment. 4 plasma samples will be collected to isolate circulating nucleic acids (e.g. cfDNA) from plasma: at Run-in V1, at C1V1 before treatment, at C3V1 and at the EOTV.
- 14. For course 3 only
- 15. PGx Plasma: Blood samples will be collected before treatment at run-in V1, on C1V1, C1V3 (Day 15), C2V1, C3V1 onwards and at the EOTV. Samples will be used to evaluate exosomal RNA.
- 16. DNA banking: For details please refer to Section 5.5.1.
- 17. Immunogenicity (ADA): On days when xentuzumab is dosed and EOTV and FU visit at time points specified in Flow Chart and Appendix 10.2.2, ADA samples are to be collected prior to xentuzumab infusion. ADA samples must be collected at Run In, in treatment courses 1-12, 15, 18, EOTV and at the FU visit. For detailed sampling schedule, refer to Appendix 10.2.2
- 18. Tumour assessments should include CT or MRI scans of the chest, abdomen and pelvis, and, if clinically indicated, any other known or suspected sites of disease (e.g. breast, neck, brain etc.) accordingly to RECIST 1.1. After study entry, all lesions identified as target and non-target lesions during the screening should be followed up at all prespecified imaging time points. The same radiographic procedure must be used throughout the study. Bone scans must be performed at screening (see Section 5.2 for more detail).

### Boehringer Ingelheim BI Trial No.: 1280.18

04 Mar 2022

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Assessment will be performed at the following time points until progression/start of further treatment (tumour assessments after start of xentuzumab should be performed no more than 7 days prior to the scheduled tumour assessment date up to week 48 AND no more than 14 days prior to the scheduled tumour assessment date after week 48):

- At screening (within 28 days prior to starting the run-in period)
- Every 8 weeks (±7days): during week 8 (49-63 days after start of xentuzumab), during week 16 (105-119 days after start of xentuzumab), during week 24 (161-175 days after start of xentuzumab), during week 32 (217-231 days after start of xentuzumab), during week 40 (273-287 days after start of xentuzumab), during week 48 (329-343 days after start of xentuzumab)
- Every 12 weeks after week 48 (±7days) (e.g. during week 60 (406-434 days after start of xentuzumab), during week 72 (490-518 days after start of xentuzumab), etc.)
  - In the event of an interruption/delay to treatment, the tumour assessment schedule should not be changed.

Except in case of discontinuation from treatment due to progression, tumour assessment at EOTV is not necessary if the previous evaluation was done within 4 weeks of EOTV

- Unscheduled scan based on the investigator's judgement is allowed and should also be documented in eCRF
- 19. Abemaciclib and xentuzumab should be dispensed through IRT. Patient's screening, all drug dispensation visits and EOTV will be collected in the IRT system
- 20. Compliance check: On Day -1, on Day 1 of every treatment course starting on course 2, and at EOTV

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### FLOW CHART – COHORT F (BC EXPANSION COHORT)

| Study period | Screening(a) | Treatment Courses (b) | | | | | | | | EOTV<br>(c) | FU (d) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | SCR | | C | ourse 1 | | Co | ourse | 2 onwa | ards | (0) | |
| Visits (V) | Screening | 1 | 2 | 3 | 4 | 1 | 2 | 3 | 4 | | |
| Days | Within 28d<br>before<br>C1V1 | 1 | 8<br>±1 | 15±1 | 22±1 | 1<br>±2 | 8*<br>±2 | 15*<br>±2 | 22*<br>±2 | Within 7d after last drug intake | 42 +7d after last drug<br>intake |
| Informed consent (1) | X | | | | | | | | | | |
| Demographics | X | | | | | | | | | | |
| Medical history | X | | | | | | | | | | |
| Inclusion/exclusion criteria (2) | X (2) | X (2) X (2) | | | | | | | | | |
| Physical exam (3) | X | X | | | | X | | | | X | X |
| Height | X | | | | | | | | | | |
| Body weight | X | X | | | | X | | | | X | X |
| Vital signs (4) | X | X | X | X | X | X | | | | X | X |
| ECOG performance status | X | X | | | | X | | | | X | X |
| 12-lead ECG<br>(triplicate) (5) | X | X | | X | | X | | X | | X | X |
| Safety lab (6) | X | X | X | X | X | X | | X<br>(7) | | X | X |
| Archival tumour tissue collection (8) | X | | | | | | | | | | |
| DNA banking (9) | | X | | | | | | | | | |
| Tumour assessment<br>and bone scan by<br>RECIST 1.1 (10) | | | | | Per i | nstitu | tional | praction | ce | | |
| Adverse event | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant therapy | X | X | X | X | X | X | X | X | X | X | X |
| Abemaciclib dispensation (11) | | X | | | | X | | | | | |
| Xentuzumab i.v. (11) | | X | X | X | X | X | X | X | X | | |
| Fulvestrant i.m. (11) | | X | | X | | X | | | | | |
| Compliance check abemaciclib (12) | | | | | | X | | | | X | |
| Termination of trial medication | | | | | | | | | | X | |
| Completion of the study participation | | | | | | | | | | | X |

- a Screening: The screening visit should be performed within 28 days prior to first drug administration (C1V1). Safety lab at the screening assessment can serve as the C1V1 assessment if performed within 72 hours before the first treatment and does not need to be repeated
- b Treatment courses: All courses are 4 weeks in duration (28 days). All subsequent visit dates should be calculated based on Course 1 Visit 1 date. One or more visits can be skipped in case of treatment interruption. Patients may continue on treatment until the criteria for stopping medication are met (see Section 3.3.4). A duration of approximately 24 cycles is expected.
- c EOTV: End of Treatment visit. If the decision to permanently discontinue all study treatments is taken during a scheduled visit, the End Of Treatment Visit (EOTV) should be performed instead of the scheduled visit (within 7 calendar days after last drug administration)
- d FU: All patients should have a follow-up visit 42 days (+7days) after the permanent discontinuation of the study drugs. Patients who have not progressed and not started further treatment at FU should have additional limited follow-up visits at scheduled tumor assessment until progression, start of further anticancer treatment, consent withdrawal, lost to follow-up or death. See <a href="Section 5.2">Section 5.2</a> and <a href="Section 6.2.3">Section 6.2.3</a>
- \* When xentuzumab is discontinued, the visit can be conducted by phone

### Boehringer Ingelheim BI Trial No.: 1280.18

c09049566-10

04 Mar 2022

Trial Protocol 

- 1. Written informed consent must be obtained before any protocol specific screening assessment is performed
- 2. In/Exclusion criteria must be checked at screening and ensured before study medication has been firstly administered
- 3. Physical exam: includes a thorough cardiopulmonary, abdominal and lymph node exam and an assessment of the mental and neurological status. When xentuzumab is discontinued, physical exam can be done as per institutional practice.
- 4. Vital signs: includes respiratory rate, pulse, temperature and blood pressure. When xentuzumab is discontinued, vital signs assessments can be done as per institutional practice.
- 5. 12-lead ECG: 12-Lead resting electrocardiograms (ECG) are recorded locally and in triplicate. ECG will be performed at Screening, EOTV and FU visit. ECG will be repeated at Visit 1/Day 1, and Visit 3/Day 15 of Course 1, 2, 3; and at Visit 1/Day 1 of Courses 6,9,12, etc. ECG should be performed prior to xentuzumab infusion. When xentuzumab is discontinued, ECGs can be omitted.
- 6. Safety labs: includes haematology (CBC), coagulation, and negative serum pregnancy test for women with childbearing potential and biochemistry. Urinalysis only at screening and EOTV. Fasting blood test is required for metabolic panels. Baseline Local FSH and estradiol levels should be within 14 days of initial dose of study treatment. See Section 5.3.3 for detail. Safety lab can be performed one day prior to the scheduled test. Unscheduled safety lab should be performed if clinically indicated and documented in the eCRF. When xentuzumab is discontinued, safety labs can be done as per institutional practice.
- 7. For course 2 only
- 8. Archival tumour tissue collection: the most recent/appropriate archival tumour tissue must be collected prior to the start of trial treatment. Refer to <u>Appendix 10.3</u> for tissue requirements
- 9. DNA banking: For details please refer to Section 5.5.1.
- 10. Tumour assessments will be performed according to institutional practice. Only the overall response will be collected in the eCRF.
- 11. Abemaciclib, xentuzumab and fulvestrant (in certain countries) should be dispensed through IRT. Patient's screening, all drug dispensation visits and EOTV will be collected in the IRT system
- 12. Compliance check: On Day -1, on Day 1 of every treatment course starting on course 2, and at EOTV

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### FLOW CHART – COHORTS D1 AND D2 (BC EXPANSION COHORTS)

| Study period | Screening (a) | Screening (a) Treatment Courses (b) | | | | | | | | | EOTV (c) | FU (d) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | SCR | | | ourse 1 | | | Coı | ırse 2 oı | ıwards | | | |
| Visits (V) | Screening | 1 | 2 | 3 | 4 | 1 | 1b | 2 | 3 | 4 | | |
| Days | Within 28d<br>before<br>C1V1 | 1 | 8<br>±1 | 15<br>±1 | 22<br>±1 | 1<br>±2 | 4<br>±1<br>(e) | 8*<br>±2<br>(f) | 15*<br>±2 | 22*<br>±2 | Within 7d after last drug intake | 42 +7d<br>after<br>last<br>drug<br>intake |
| Informed consent (1) | X | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | |
| Inclusion/exclusion<br>criteria (2) | X (2) | | | | | | | | | | | |
| Physical exam (3) | X | X | | | | X | | | | | X | X |
| Height | X | | | | | | | | | | | |
| Body weight | X | X | | | | X | | | | | X | X |
| Vital signs (4) | X | X | X | X | X | X | | | | | X | X |
| ECOG performance status | X | X | | | | X | | | | | X | X |
| 12-lead ECG (triplicate) (5) | X | X | | X | | X | | | X | | X | X |
| Safety lab (6) | X | X | X | X | X | X | | | X<br>(7) | | X | X |
| Archival tumour tissue collection (8) | X | | | | | | | | | | | |
| DNA banking (9) | | X | | | | | | | | | | |
| Tumour assessment and bone scan by RECIST 1.1 (10) | | | | | Per in | nstitut | ional p | practice | | | | |
| Adverse event | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant therapy | X | X | X | X | X | X | | X | X | X | X | X |
| Abemaciclib dispensation (11) | | X | | | | X | | | | | | |
| Xentuzumab i.v. (11) | | X | X | X | X | X | | X | X | X | | |
| Fulvestrant i.m. (11) | | X | Λ | X | / <b>\</b> | X | | Λ | Λ | Λ | | |
| Compliance check | | Λ | | Λ | | Λ | | | | | | |
| abemaciclib (12) | | | | | | X | | | | | X | |
| Termination of trial | | | | | | | | | | | | |
| medication | | | | | | | | | | | X | |
| Completion of the study participation | | | | | | | | | | | | X |

- \* A 24 h sample is also required at C2V1D2 (see Appendix 10.2.4)
- a Screening: The screening visit should be performed within 28 days prior to first drug administration (C1V1). Safety lab at the screening assessment can serve as the C1V1 assessment if performed within 72 hours before the first treatment and does not need to be repeated.
- b Treatment courses: All courses are 4 weeks in duration (28 days). All subsequent visit dates should be calculated based on Course 1 Visit 1 date. One or more visits can be skipped in case of treatment interruption. Patients may continue on treatment until the criteria for stopping medication are met (see Section 3.3.4). A duration of approximately 24 cycles is expected.
- c EOTV: End of Treatment visit. If the decision to permanently discontinue all study treatments is taken during a scheduled visit, the End Of Treatment Visit (EOTV) should be performed instead of the scheduled visit (within 7 calendar days after last drug administration)
- d FU: All patients should have a follow-up visit 42 days (+7days) after the permanent discontinuation of the study drugs. Patients who have not progressed and not started further treatment at FU should have additional limited follow-up visits at scheduled tumor assessment until progression, start of further anticancer treatment, consent withdrawal, lost to follow-up or death. See Sections 5.2 and 6.2.3
- e On course 2 only for PK purposes
- f No time window is applicable for course 2 when PK determinations are scheduled for the visit

### Boehringer Ingelheim BI Trial No.: 1280.18 c09049566-10

04 Mar 2022

0 Trial Protocol 

- When xentuzumab is discontinued, the visit can be conducted by phone
- 1. Written informed consent must be obtained before any protocol specific screening assessment is performed
- 2. In/Exclusion criteria must be checked at screening and ensured before study medication has been firstly administered
- 3. Physical exam: includes a thorough cardiopulmonary, abdominal and lymph node exam and an assessment of the mental and neurological status. When xentuzumab is discontinued, physical exam can be done as per institutional practice.
- 4. Vital signs: includes respiratory rate, pulse, temperature and blood pressure. When xentuzumab is discontinued, vital signs assessments can be done as per institutional practice.
- 5. 12-lead ECG: 12-Lead resting electrocardiograms (ECG) are recorded locally and in triplicate. ECG will be performed at Screening, EOTV and FU visit. ECG will be repeated at Visit 1/Day 1, and Visit 3/Day 15 of Course 1, 2, 3; and at Visit 1/Day 1 of Courses 6,9,12, etc. ECG should be performed prior to xentuzumab infusion. When xentuzumab is discontinued, ECGs can be omitted.
- 6. Safety labs: includes haematology (CBC), coagulation, and negative serum pregnancy test for women with childbearing potential (within 14 days of first study dose) and biochemistry. Urinalysis only at screening and EOTV. Fasting blood test is required for metabolic panels. Baseline Local FSH and estradiol levels should be within 14 days of initial dose of study treatment. See Section 5.3.3 for detail. Safety lab can be performed one day prior to the scheduled test. Unscheduled safety lab should be performed if clinically indicated and documented in the eCRF. When xentuzumab is discontinued, safety labs can be done as per institutional practice.
- 7. For course 2 only
- 8. Archival tumour tissue collection: the most recent/appropriate archival tumour tissue must be collected prior to the start of trial treatment. Refer to <a href="Appendix 10.3">Appendix 10.3</a> for tissue requirements
- 9. DNA banking: For details please refer to Section 5.5.1.
- Tumour assessments will be performed according to institutional practice. Only the overall response will be collected in the eCRF.
- 11. Abemaciclib, xentuzumab and fulvestrant (in certain countries) should be dispensed through IRT. Patient's screening, all drug dispensation visits and EOTV will be collected in the IRT system
- 12. Compliance check: on Day 1 of every treatment course starting on course 2, and at EOTV

c09049566-10 **Trial Protocol** 

 Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## **TABLE OF CONTENTS**

| TITLE P | PAGE | 1 |
|---|---|---|
| CLINIC | AL TRIAL PROTOCOL SYNOPSIS | 2 |
| FLOW ( | CHART – COHORT A (SOLID TUMOURS) | 14 |
| | CHART – COHORT B (BC TRIPLET WITH LETROZOLE) | |
| | CHART – COHORT C (BC TRIPLET WITH ANASTROZOLE) | |
| | CHART – COHORT D – DOSE FINDING (BC TRIPLET WITH | 10 |
| ILOW | FULVESTRANT) | 20 |
| FLOW ( | CHART – COHORT E (NSCLC EXPANSION COHORT) | 22 |
| | CHART – COHORT F (BC EXPANSION COHORT) | |
| | CHART – COHORTS D1 AND D2 (BC EXPANSION COHORTS) | |
| | OF CONTENTS | |
| | VIATIONS | |
| 1. | INTRODUCTION | |
| 1.1 | MEDICAL BACKGROUND. | |
| 1.1<br>1.2 | DRUG PROFILE | |
| 2. | RATIONALE, OBJECTIVES, AND BENEFIT - RISK ASSESSMENT | |
| 2.1 | RATIONALE FOR PERFORMING THE TRIAL | 41 |
| 2.2 | TRIAL OBJECTIVES | 42 |
| 2.3 | BENEFIT - RISK ASSESSMENT | |
| 3. | DESCRIPTION OF DESIGN AND TRIAL POPULATION | 46 |
| 3.1 | OVERALL TRIAL DESIGN AND PLAN | |
| 3.1.1 | Administrative structure of the trial | 48 |
| 3.2 | DISCUSSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF CONTROL GROUP(S) | 40 |
| 3.3 | SELECTION OF TRIAL POPULATION | |
| 3.3.1 | Main diagnosis for trial entry | |
| 3.3.2 | Inclusion criteria | |
| 3.3.3 | Exclusion criteria | 55 |
| 3.3.4 | Removal of patients from therapy or assessments | 58 |
| 3.3.4.1 | Removal of individual patients | |
| 3.3.4.2 | Discontinuation of the trial by the sponsor | |
| 3.3.5 | Replacement of patients | 60 |
| 4. | TREATMENTS | 61 |
| 4.1 | INVESTIGATIONAL TREATMENTS | |
| 4.1.1 | Identity of the Investigational Medicinal Products | 61 |
| 4.1.2 | Selection of doses in the trial | |
| 4.1.2.1 | Part 1 | 63 |

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | tary confidential information © 2024 Declininger ingenient international Onion of one of more of its arithmetic of | • |
|---|---|---|
| 4.1.2.2 | Part 2 | |
| 4.1.2.3 | Part 3 | |
| 4.1.3 | Method of assigning patients to treatment groups | 00 |
| <b>4.1.4</b> 4.1.4.1 | <b>Drug assignment and administration of doses for each patient</b> Initial study drug assignment and administration | |
| 4.1.4.1 | Temporary treatment interruption and dose reduction | |
| 4.1.4.2 | Blinding and procedures for unblinding | |
| 4.1.5.1 | Blinding | |
| 4.1.5.2 | Unblinding and breaking the code | |
| 4.1.6 | Packaging, labelling, and re-supply | |
| 4.1.7 | Storage conditions | |
| 4.1.8 | Drug accountability | |
| 4.2 | OTHER TREATMENTS, EMERGENCY PROCEDURES, | , _ |
| | RESTRICTIONS | 73 |
| 4.2.1 | Other treatments and emergency procedures | |
| 4.2.2 | Restrictions | |
| 4.2.2.1 | Restrictions regarding concomitant treatment | |
| 4.2.2.2 | Restrictions on diet and life style | |
| 4.2.2.3 | Restrictions regarding men and women of childbearing potential | |
| 4.2.2.4 | Supportive Care | |
| 4.2.2.5 | Growth Factor Therapy | 76 |
| 4.2.2.6 | Therapy for Diarrhoea | |
| 4.2.2.7 | Ovarian suppression with gonadotropin-releasing hormone agonists | |
| 4.3 | TREATMENT COMPLIANCE | 77 |
| 4.4 | MANAGEMENT OF EXPECTED ADVERSE EVENTS | |
| 4.4.1 | Increased Serum Creatinine | |
| 4.4.2 | Management and grading of infusion reactions | |
| 4.4.3 | Management of Neutropenia | |
| 4.4.4 | Management of Hepatotoxicity | |
| 4.4.5 | Venous Thromboembolism | |
| 4.4.6 | Guidance for Interstitial lung disease/Pneumonitis | 80 |
| 5. | VARIABLES AND THEIR ASSESSMENT | 81 |
| 5.1 | TRIAL ENDPOINTS | 81 |
| 5.1.1 | Primary Endpoint(s) | |
| 5.1.2 | Secondary Endpoint(s) | 82 |
| 5.2 | ASSESSMENT OF EFFICACY | 85 |
| 5.3 | ASSESSMENT OF SAFETY | |
| 5.3.1 | Physical examination | |
| 5.3.2 | Vital Signs | |
| 5.3.3 | Safety laboratory parameters | |
| 5.3.4 | Electrocardiogram | |
| 5.3.5 | Other safety parameters | |
| 5.3.6 | Assessment of adverse events | |
| 5.3.6.1 | Definitions of AEs | 87 |
| 5.3.6.2 | Adverse event collection and reporting | 91 |

| c09049566-10 Trial Protocol Page 31 | l O | f J | 17 | ľ | , | i |
|-------------------------------------|-----|-----|----|---|---|---|
|-------------------------------------|-----|-----|----|---|---|---|

| Proprie | tary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliate | d companies |
|---|---|---|
| 5.3.6.3 | Exemption to (S)AE Reporting | 92 |
| 5.3.7 | Dose Limiting Toxicities (DLTs) | |
| 5.4 | DRUG CONCENTRATION MEASUREMENTS AND | |
| | PHARMACOKINETICS | 94 |
| 5.4.1 | Assessment of Pharmacokinetics | |
| 5.4.2 | Methods of sample collection | |
| | The moust of sumple concertor with the manufacture of the manufacture | |
| 5.4.4 | Pharmacokinetic – Pharmacodynamic Relationship | 96 |
| 5.5 | ASSESSMENT OF BIOMARKER(S) | |
| 5.5.1 | Biobanking | |
| 5.5.1.1 | DNA Banking | |
| 5.6 | OTHER ASSESSMENTS | |
| 5.6.1 | Assessment of Immunogenicity | |
| 5.7 | APPROPRIATENESS OF MEASUREMENTS | 101 |
| 6. | INVESTIGATIONAL PLAN | 103 |
| 6.1 | VISIT SCHEDULE | 103 |
| 6.2 | DETAILS OF TRIAL PROCEDURES AT SELECTED VISITS | |
| 6.2.1 | Screening and run-in period(s) | |
| 6.2.2 | Treatment period(s) | |
| 6.2.2.1 | Cohort A, B, C, and D (dose finding) | |
| 6.2.2.2 | Cohort E | |
| 6.2.2.3 | Cohorts D1, D2 and F | |
| 6.2.3 | Follow Up Period and Trial Completion | |
| 6.2.3.1 | End of treatment visit. | |
| 6.2.3.2 | Follow-up period | |
| 6.2.3.3 | Trial Completion | |
| | • | |
| 7. | STATISTICAL METHODS AND DETERMINATION OF SAMP | |
| | | 108 |
| 7.1 | STATISTICAL DESIGN - MODEL | 108 |
| 7.2 | NULL AND ALTERNATIVE HYPOTHESES | |
| 7.3 | PLANNED ANALYSES | |
| 7.3.1 | Primary endpoint analyses | |
| 7.3.2 | Secondary endpoint analyses | |
| 7.3.4 | Safety analyses | 115 |
| 7.3.5 | Pharmacokinetic and pharmacodynamic analyses | 116 |
| 7.4 | INTERIM ANALYSES | |
| 7.5 | HANDLING OF MISSING DATA | |
| 7.6 | RANDOMISATION | |
| 7.7 | DETERMINATION OF SAMPLE SIZE | |
| 8. | INFORMED CONSENT, TRIAL RECORDS, DATA PROTECTI | |
| | PUBLICATION POLICY | 122 |
| 8.1 | TRIAL APPROVAL, PATIENT INFORMATION, INFORMED | |
| - | CONSENT | 122 |
| 8.2 | DATA QUALITY ASSURANCE | |
| | <u>~</u> | |

c09049566-10 Trial Protocol 

| Prop | orietary | confidential confidential | l informatioi | n © 2024 i | Boehringer In | gelheim | International | GmbH o | or one or more of its | affiliated com | panies |
|---|---|---|---|---|---|---|---|---|---|---|---|

| 8.3 | RECORDS | 23 |
|---|---|---|
| 8.3.1 | Source documents | 23 |
| 8.3.2 | Direct access to source data and documents12 | 4 |
| 8.3.3 | Storage period of records | 25 |
| 8.4 | EXPEDITED REPORTING OF ADVERSE EVENTS | 25 |
| 8.5 | STATEMENT OF CONFIDENTIALITY AND PATIENT PRIVACY 12 | 25 |
| 8.5.1 | Collection, storage and future use of biological samples and corresponding | |
| | data12 | |
| 8.6 | TRIAL MILESTONES | 26 |
| <b>8.7</b> | PROTOCOL VIOLATIONS | |
| 8.8 | COMPENSATION AVAILABLE TO THE PATIENT IN THE EVENT OF | i |
| | TRIAL RELATED INJURY12 | |
| 9. | REFERENCES | 28 |
| 9.1 | PUBLISHED REFERENCES | 28 |
| 9.2 | UNPUBLISHED REFERENCES 13 | |
| 10. | APPENDICES 13 | |
| 10.1 | INDUCERS AND STRONG INHIBITORS OF CYP3A4 13 | |
| 10.2 | PHARMACOKINETICS PLAN | |
| 10.2.1 | FLOW CHART for PK, immunogenicity, and biomarkers for cohorts A, B, | |
| | C, and D (dose finding) | 2 |
| 10.2.1.1 | Flowchart for PK, immunogenicity, and biomarkers for Cohorts A, B, C, and D | |
| | (dose finding) in treatment course 1 | 12 |
| 10.2.1.2 | FLOW CHART for PK, immunogenicity, and biomarkers for cohorts A, B, C, | |
| | and D (dose finding) in courses 2-12, 15, and 18, EOTV and FU13 | |
| 10.2.2 | FLOW CHART for PK, immunogenicity, and biomarkers for cohort E 13 | |
| 10.2.2.1 | FLOW CHART for PK, immunogenicity, and biomarkers for cohort E in Run-in | |
| | phase and treatment course 1 | 4 |
| 10.2.2.2 | FLOW CHART for PK, immunogenicity, and biomarkers for cohort E in | |
| | treatment course 2 | 5 |
| 10.2.2.3 | FLOW CHART for PK, immunogenicity, and biomarkers for cohort E in | |
| | treatment courses 3-12, 15, 18 and EOTV and FU visit | |
| 10.2.3 | FLOW CHART for PK, immunogenicity, and biomarkers for cohort F 13 | 7 |
| 10.2.3.1 | FLOW CHART for PK, immunogenicity, and biomarkers for cohort F in | |
| | screening and treatment course 1 | 57 |
| 10.2.3.2 | FLOW CHART for PK, Immunogenicity, biomarkers for cohort F in treatment | |
| | courses 2-12, 15, 18, EOTV and FU | 8 |
| 10.2.4 | FLOW CHART for PK, immunogenicity, and biomarkers for cohorts D1 | |
| | and D2 | |
| 10.2.4.1 | FLOW CHART for PK, immunogenicity, and biomarkers for cohorts D1 and D2 | 2 |
| | in treatment course 1 | |
| 10.2.4.2 | FLOW CHART for PK, immunogenicity, and biomarkers for cohorts D1 and D2 | |
| | in treatment course 2 | 0 |
| 10.2.4.3 | FLOW CHART for PK, Immunogenicity, biomarkers for cohorts D1 and D2 in | |
| | treatment courses 3, 4, 6, 12, 24, EOTV and FU14 | |
| 10.3 | TUMOUR TISSUE SAMPLE REQUIREMENTS14 | 12 |

c09049566-10

| Trial Protocol |
|----------------|
| 11141111000001 |

| 10.4 | TUMOUR RESPONSE ASSESSMENT ACCORDING TO RE | CIST 1.1143 |
|--------|--------------------------------------------|-------------|
| 10.5 | CLINICAL EVALUATION OF LIVER INJURY | 145 |
| 10.5.1 | Introduction | |
| 10.5.2 | Procedures | |
| 10.6 | STATISTICAL APPENDIX | 146 |
| 11. | DESCRIPTION OF GLOBAL AMENDMENT(S) | 151 |
| 11.1 | GLOBAL AMENDMENT 1 | 151 |
| 11.2 | GLOBAL AMENDMENT 2 | 154 |
| 11.3 | GLOBAL AMENDMENT 3 | |
| 11.4 | GLOBAL AMENDMENT 4 | 164 |
| 11.5 | GLOBAL AMENDMENT 5 | |
| 11.6 | GLOBAL AMENDMENT 6 | 168 |
| 11.7 | GLOBAL AMENDMENT 7 | 171 |
| 11.8 | GLOBAL AMENDMENT 8 | 175 |

04 Mar 2022

Boehringer Ingelheim BI Trial No.: 1280.18

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **ABBREVIATIONS**

AE Adverse Event

AESI Adverse Event of Special Interest

AUC Area under the Curve

BC Breast Cancer

b.i.d. bis in die (twice daily dosing)

BIRDS Boehringer Ingelheim Regulatory Documents for Submission

BLRM Bayesian Logistic Regression Model

CCDS Company Core Data Sheet
CDK Cyclin-dependent Kinase
CI Confidence Interval
CML Local Clinical Monitor
CRA Clinical Research Associate

CRF Case Report Form

CTCAE Common Terminology Criteria for Adverse Events

CTP Clinical Trial Protocol
CTR Clinical Trial Report
DILI Drug Induced Liver Injury
DLT Dose Limiting Toxicity
EDC Electronic Data Capture

ePRO Electronic Patient Reported Outcome

EOTV End of Trial Visit

EWOC Escalation With Overdose Control EudraCT European Clinical Trials Database

FAS Full Analysis Set
FC Flow Chart
FU Follow Up
FUV Follow Up Visit

GCP Good Clinical Practice

HR Hormone Receptor
IB Investigator's Brochure
ICF Informed Consent Form

ICH International Conference on Harmonization

IEC Independent Ethics Committee IGF Insulin-like Growth Factor

i.m. Intramuscular

IRB Institutional Review Board IRR Infusion Related Reaction

IRT Interactive Response Technology

ISF Investigator Site File

i.v. intravenous

LA Locally Advanced
LoEE List of Essential Element
mAB Monoclonal Antibody

MedDRA Medical Dictionary for Drug Regulatory Activities

Boehringer Ingelheim 04 Mar 2022

BI Trial No.: 1280.18

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

MST Medical Sub team

MTD Maximum Tolerated Dose NSCLC Non-Small Cell Lung Cancer

OPU Operative Unit
OS Overall Survival
PD Pharmacodynamics
PK Pharmacokinetics
p.o. per os (oral)

PCC Protocol Challenge Committee
PFS Progression-free survival
pRb Retinoblastoma protein
q.d. quaque die (once a day)

REP Residual effect period, after the last dose of medication with measureable

drug levels or pharmacodynamic effects still likely to be present

SAE Serious Adverse Event SC Steering Committee

s.c. subcutaneous

SmPC Summary of Product Characteristics

TCM Trial Clinical Monitor

TDMAP Trial Data Management and Analysis Plan

t.i.d. ter in die (3 times a day)

TMF Trial Master File
TMW Trial Medical Writer

TSAP Trial Statistical Analysis Plan

WHO/ECOG World Health Organization / Eastern Cooperative Oncology Group

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 1. INTRODUCTION

#### 1.1 MEDICAL BACKGROUND

#### Hormone receptor-positive (HR+) breast cancer (BC)

Breast cancer is one of the most common cancers in women. In 2012, there were approximately 226,870 new cases of breast cancer and 39,510 deaths from the disease among women in the United States (Siegel et al. 2012 R12-2864). While early stage disease is curable, patients with metastatic breast cancer (mBC) have a median overall survival (OS) of only 2 to 3 years (R16-3983). The treatment for women diagnosed with hormone receptor positive (HR+) mBC includes endocrine therapy (R16-3983). However, de novo or acquired resistance to endocrine therapy remains an important clinical problem. Many HR+ breast cancers demonstrate overexpression of cyclin D1 (R16-3978), which interacts with cyclin-dependent kinases 4 and 6 (hereafter CDK4/6) in an active protein complex that promotes cell proliferation. Consequently, CDK4/6 represents a potential therapeutic target for HR+ breast cancers, and CDK4/6 inhibitors need to be evaluated for their potential to improve clinical outcomes for women with HR+ mBC.

Despite recent advances, hormone-positive HR+ advanced or metastatic breast cancer still has a dismal prognosis with median progression-free survival (PFS) of less than a year; almost all patients will develop resistance to endocrine treatment and succumb to their disease eventually. Biochemical and genetic characterization of D-type cyclins, their cyclin D-dependent kinases (CDK4 and CDK6), and the polypeptide CDK4/6 inhibitor p16INK4A over two decades ago revealed how mammalian cells regulate entry into the DNA synthetic (S) phase of the celldivision cycle in a retinoblastoma protein (pRb)-dependent manner. These investigations provided proof-of-principle that CDK4/6 inhibitors, such as abemaciclib, particularly when combined with co-inhibition of allied mitogen-dependent signal transduction pathways, might prove valuable in cancer therapy. The recent FDA approval of the CDK4/6 inhibitor palbociclib (Ibrance<sup>TM</sup>), used with the aromatase inhibitor letrozole and fulvestrant for breast cancer treatment, highlights long-sought success by showing unprecedented efficacy in this setting. Moreover, the newest findings herald clinical trials targeting other cancers such as non-small cell lung cancer (NSCLC). Rapidly emerging data with selective inhibitors of CDK4/6 have validated these cell-cycle kinases as anticancer drug targets, corroborating longstanding preclinical predictions (R16-2249; R16-3979).

#### Non-small cell lung cancer (NSCLC)

Lung cancer is the most common cancer worldwide as well as the leading cause of cancer related deaths in both men and women. Non-small cell lung cancer (NSCLC) accounts for up to 85% of all lung cancers and of these, adenocarcinoma and squamous cell carcinoma (SCC) account for 50% and 30% respectively. Most of these patients present with locally advanced inoperable or metastatic disease, which makes their cancer incurable, and unfortunately almost all of these patients will die from their illness. Despite multiple advances in the staging, diagnostic procedures and therapeutic options, the overall outlook has not greatly changed for the majority of patients with the overall 5-year survival having only marginally increased over the last decade from 15.7% to 17.4% (P15-10237). Smoking remains the major cause of NSCLC, although the identification of driver oncogenes in non-smoking patients represents a critical novel finding during the last decades that fundamentally changed the management of
Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

this disease. The recognition that NSCLC is not a single disease entity today is a well-known reality that has led to divide NSCLC into different sub-types, each one with specific algorithms of treatment, based on histological and molecular features (reviewed in <u>P16-09577</u> and <u>P15-10237</u>).

Thus, the landscape of NSCLC therapies has rapidly been evolving beyond chemotherapy over the last few years. The discovery of oncogenic driver mutations has led to new ways in classifying NSCLC as well as offered novel therapeutic targets for anticancer therapy. Targets such as epidermal growth factor receptor (EGFR) mutations and anaplastic lymphoma kinase (ALK) gene rearrangements have successfully been targeted with appropriate tyrosine kinase inhibitors (TKIs). Other driver mutations such as ROS, MET, RET, BRAF have also been investigated with targeted agents with some success in the early phase clinical setting. Novel strategies in the field of immune-oncology have also led to the development of inhibitors of cytotoxic T lymphocyte antigen-4 (CTLA-4) and programmed death-1 receptor (PD-1), which are important pathways in allowing cancer cells to escape detection by the immune system (P15-10237).

Despite this impressive progress, however, there remain many patients that are refractory to immune checkpoint inhibitors (e.g. nivolumab and pembrolizumab) or chemotherapy and who do not benefit from targeted agents against activating -mutations in the EGFR gene or the ALK translocation, such as afatinib or crizotinib, respectively. Clearly, therefore, novel agents against additional molecular targets are desperately needed. In this regard, the insulin growth factor-1 receptor (IGF-1R) is a heterodimeric transmembrane tyrosine kinase receptor that is a mediator of cellular proliferation and frequently overexpressed in NSCLC.

# **CDK4/6 inhibitors (Abemaciclib)**

During the cell cycle, the G1 restriction point controls entry into S phase and is essential for maintaining control of cell division (R16-2249, R16-3704). The cyclin-dependent kinases (CDKs), CDK4 and CDK6 (hereafter designated CDK4/6), participate in a complex with D-type cyclins to initiate the transition through the G1 restriction point by phosphorylating and inactivating the retinoblastoma (Rb) tumour suppressor protein.

Alterations in this pathway occur frequently in human cancers, amongst others HR+ BC, NSCLC and Pancreatic Cancer, and involve 1) loss of CDK inhibitors by mutation or epigenetic silencing, 2) mutation/overexpression of either CDK4/6 or cyclin D, or 3) inactivation of Rb. These alterations render cells less dependent on mitogenic signalling for proliferation. With the possible exception of those tumours with complete inactivation of Rb, which functions downstream of the CDK4/6-cyclinD complex, most cancers are potentially sensitive to pharmacologic inhibition of CDK4/6. All of these cancers are potentially sensitive to pharmacologic inhibition of CDK4/6. From a therapeutic standpoint, the goal of inhibiting CDK4/6 with a small molecule inhibitor is to prevent cell cycle progression through the G1 restriction point, thus arresting tumour growth in the cancers investigated in the present trial.

#### **Targeting IGF in cancer (xentuzumab)**

The insulin-like growth factor (IGF) signalling system consists of ligands (insulin-like growth factors 1 and 2 (IGF-1, IGF-2), IGF-binding proteins (IGFBPs), and receptors (IGF-1R, IGF-2R and insulin receptor IR)). Evidence that targeting IGF may be useful in cancer treatment was first recognized decades ago. Research in IGF signalling has shown that it controls key cellular activities, including proliferation, growth, and survival and is often deregulated in


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

neoplasia (<u>R12-4524</u>, <u>P15-00363</u>, <u>P15-10395</u>). There is experimental and clinical evidence that cancer cells express insulin and IGF-1 receptors. Expression of IGF-1R or its ligand is increased in a variety of cancers, including lung, colon, prostate, breast, ovarian, liver cancer and sarcoma (<u>R12-4524</u>, <u>P15-00363</u>, <u>P15-10395</u>). Therefore, the IGF system is an attractive tempting target for anti-cancer drug development.

Pharmacologic targeting strategies include inhibition of receptor function with anti-receptor antibodies or small molecule receptor tyrosine kinase inhibitors (R12-4524, P15-00363, P15-10395). Xentuzumab offers an alternative approach by acting as a ligand specific antibody. Most cancers express IGF-1 receptors, but there is evidence that autocrine and/or paracrine expression of ligands, particularly IGF-2, is deranged in neoplasm (R10-5355). In addition, the IGF-2 gene is an imprinted gene; loss of imprinting is one of several mechanisms leading to IGF-2 overexpression (R10-5694). Further, IGF-2 activates insulin receptor which was not targeted by any of the IGF-1 receptor monoclonal antibodies. Thus, targeting IGF-1 and IGF-2 by neutralization may lead to a higher probability of response to a therapeutic strategy and may confer an advantage over previously attempted approaches. Xentuzumab is a humanized monoclonal antibody directed against insulin-like growth factors 1 and 2 (IGF-1/-2) with the potential of anti-neoplastic activity. Despite encouraging preliminary evidence of clinical activity of several anti-IGF-1R agents, the therapeutic value of targeting the IGF/IGF-1R signalling system remains incompletely tested, given that the development of certain promising agents (e.g., figitumumab, ganitumab, dalotuzumab, R1507) has been discontinued in some indications. Efficacy signals generated by these and other agents warrant further exploration of the potential therapeutic value of targeting the IGF pathway in patients with various cancers.

#### 1.2 DRUG PROFILE

For a more detailed description of the xentuzumab profile and abemaciclib profile please refer to the current Investigator's Brochure (IB) and for letrozole, anastrozole and fulvestrant to the SmPC or US PI.

#### Xentuzumab

Xentuzumab is a humanized IgG1 monoclonal antibody that binds with high affinity to IGF-1 and IGF-2, and potently neutralizes the proliferative and pro-survival cellular signalling triggered by both proteins. Mode of action differentiation to IGF-1 receptor (IGF-1R) targeted antibodies was demonstrated, in particular through inhibition of IGF-2 stimulated insulin receptor-A (IR-A) activation, an additional proliferative and pro-survival pathway not inhibited by IGF-1R targeted mAbs.

At the cut-off date of 18 January 2019, a total of about 494 patients were treated in the xentuzumab clinical program: Eighty-one (81) patients were treated in two xentuzumab Phase I dose-escalation trials, examining a weekly and a three-weekly dosing schedule. Dose escalation to 1800 mg weekly or 3600 mg q3w did not identify a maximum-tolerated dose. A relevant biological dose for xentuzumab monotherapy in solid tumours was determined at 1000 mg weekly, used as the recommended dose for further Phase II trials (RP2D).

Moreover, in a phase Ib / randomized phase II study of xentuzumab in combination with everolimus and exemestane in patients with advanced or metastatic hormone-receptor positive

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

(HR+) breast cancer (Study 1280.4), 24 patients were treated in the dose escalation part (Ib) of this trial.

The MTD of xentuzumab was 1000 mg/week in combination with exemestane 25 mg/day and everolimus 10 mg/day, which was also determined as the RP2D.

Lastly, a completed phase Ib trial evaluates the safety and anti-tumour activity of xentuzumab in combination with afatinib in patients with non-small cell lung cancer with resistant to epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors. At the time of the data cut-off (18 January 2019), the safety profile was as expected for monotherapy of afatinib. The RP2D has been determined at 40 mg/day afatinib and 1000 mg/week xentuzumab.

No relevant hyperglycaemia has been observed so far. Xentuzumab was well tolerated, with no relevant side effects reported. The type and pattern of adverse events (AEs) observed to date have generally been of mild to moderate intensity (CTCAE Grades 1 or 2) or consistent with the safety profile of combination backbone treatment or consistent with the underlying neoplastic conditions of patients enrolled on the study. The most frequently reported AEs for xentuzumab monotherapy were fatigue, decreased appetite, nausea, diarrhoea, and vomiting. Infusion-related reaction (IRR) is a listed side effect of xentuzumab treatment.

Promising early efficacy signals in the dose escalation part of the 2 phase I studies have been observed with two confirmed antitumour responses (Partial Responses) according to RECIST criteria in a patient with nasopharyngeal cancer and a patient with a peripheral primitive neuroectodermal tumour (PPNET) or Ewing sarcoma. Moreover, twelve confirmed disease stabilizations (SD) have been observed in heavily pre-treated patients suffering from advanced or metastatic solid tumours. In the expansion cohorts at R2PD, no further objective responses have been observed.

At a planned interim analysis of the randomized phase II part, based on the recommendation of data monitoring committee, recruitment of phase II part was stopped and xentuzumab treatment was discontinued. According to latest analysis, in the overall population, PFS did not improve with the addition of xentuzumab to everolimus plus exemestane. Nevertheless, a favorable signal was observed in the pre-specified subgroup of patients without visceral metastasis (report c22665932-01).

In the aforementioned ongoing trial in HR+ metastatic breast cancer, the safety profile of xentuzumab in combination with everolimus and exemestane is considered favourable and as expected, since the observed safety profile of this triple combination is consistent with previously reported data for the combination doublet everolimus and exemestane (Bolero-2 trial) (Baselga et al. 2011: R12-5635). The same applies for the combination with enzalutamide in CRPC, where the safety profile of this doublet is consistent with previously reported data for enzalutamide (Affirm and Prevail trials) (R13-1229, R15-1307).

### **Abemaciclib**

Abemaciclib (LY2835219) is a small-molecule inhibitor of CDK4 and CDK6 that is structurally distinct from other dual inhibitors (such as palbociclib and ribociclib) and notably exhibits greater selectivity for CDK4 compared with CDK6. Consistent with its activity against CDK4 and CDK6, abemaciclib inhibits Rb phosphorylation and leads to G 1 arrest in RB-proficient cell lines. In a colorectal cancer xenograft model used to develop an integrated pharmacokinetic/pharmacodynamic model, abemaciclib can be dosed orally on a continuous schedule to achieve sustained target inhibition and demonstrates not only durable cell cycle

Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

inhibition but also single-agent antitumour activity. Abemaciclib demonstrates suitable physical and pharmacokinetic (PK) properties, an acceptable toxicity profile in nonclinical species, and antitumour activity in multiple mouse models of human cancer.

Tumour growth inhibition is observed in multiple other human cancer xenograft models, including those derived from non–small cell lung cancer (NSCLC), melanoma, glioblastoma, and mantle cell lymphoma. Abemaciclib distributes across the blood–brain barrier and prolongs survival in an intracranial glioblastoma xenograft model, suggesting potential efficacy against primary and metastatic tumours involving the central nervous system (R16-3982). Importantly, abemaciclib has demonstrated early evidence of activity against HR+ mBC with a confirmed objective response rate (ORR) of 19.7% in the recent Monarch 1 study (R16-5327).

Abemaciclib has been approved by US FDA for the treatment of metastatic breast cancer in three different settings. The approval include combination with an aromatase inhibitor as initial endocrine-based therapy for the treatment of postmenopausal women with HR+, HER2- advanced or metastatic breast cancer (Monarch 3), in combination with fulvestrant for the treatment of women with HR+, HER2- advanced or metastatic breast cancer with disease progression following endocrine therapy. (Monarch 2), and as monotherapy for the treatment of HR+, HER2- advanced or metastatic breast cancer with disease progression following endocrine therapy and prior chemotherapy in the metastatic setting (Monarch 1).

The approval of abemaciclib plus fulvestrant was based on Monarch 2 study, which is a randomized, placebo-controlled study in women with HR-positive and HER2-negative metastatic breast cancer. A total of 669 patients who had disease progression following endocrine therapy and had not received chemotherapy for metastatic disease were randomized 2:1 to either oral abemaciclib or placebo plus intramuscular fulvestrant injection. Treatment was continued in the absence of disease progression or unmanageable toxicity. The study was positive for primary endpoint investigator-assessed PFS. Abemaciclib plus fulvestrant significantly improved PFS versus placebo plus fulvestrant (median 16.4 v 9.3 months, hazard ratio 0.553) (R17-2796).

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 2. RATIONALE, OBJECTIVES, AND BENEFIT - RISK ASSESSMENT

#### 2.1 RATIONALE FOR PERFORMING THE TRIAL

In early-phase clinical studies, abemaciclib has shown encouraging clinical activity in HRpositive breast cancer and NSCLC as well as other solid tumours with a favourable safety profile (Study JPBA and Monarch 1 trial; R16-3982, R16-5327). In September 2017, abemaciclib in combination with fulvestrant was approved by US FDA for the treatment of women with HR-positive, HER2-negative advanced or metastatic breast cancer with disease progression following endocrine therapy (R18-2693). Oncogenic activation of the PI3KmTOR pathway, which is governed by IGF1/IGF-1R, is also capable of stimulating cyclin D1– CDK4/6 activity, due in part to the increased translation of the cyclin D1 mRNA transcript, and to the stabilization of the cyclin D1 protein (see R16-3979). This scenario prompts the implementation of triple combination studies involving the addition of a IGF/IGF-1R signalling inhibitor such as xentuzumab, to the established antihormonal plus CDK4/6 inhibitor regimens in the present trial. It seems likely that CDK4/6 inhibitors will generally prove most effective when used in combination with other agents that either reinforce the cytostatic activity of CDK4/6 inhibitors or convert reversible cytostasis into irreversible growth arrest or cell death (R16-3979). In this regard, preclinical and clinical data indicate that aberrant regulation of the IGF system is attributed to the pathogenesis of breast cancer and also contributes to the resistance to endocrine therapy (R16-3981).

Despite recent progress in the treatment of metastatic NSCLC, these neoplasms basically remain intractable in the metastatic setting, with a median overall survival of less than 12 months in patients with stage IV disease. Hence, new therapeutic approaches are urgently warranted in these areas of high unmet medical need. The IGF/IGF-1R signalling network has also been implicated in the pathogenesis of NSCLC. Specifically, a large body of literature has highlighted the ability of IGF/IGF-1R to mediate resistance to other treatment modalities in NSCLC, and conversely has identified proteins capable of compensating for IGF-1R blockade (P15-00363).

Early evaluations of ongoing clinical trials of anti-IGF/IGF-1R agents including xentuzumab as a single agent, as well as in combination with everolimus and exemestane in HR+ BC (P16-09570), have shown clinical benefit (objective tumour responses or disease stabilizations) in patients with advanced and otherwise incurable cancers.

The insulin-like growth factor receptor (IGF-1R) signalling pathway has been an active area of oncology research for the last decade. IGF-1R is present on most cancer cells, and inhibition of this receptor slowed tumour growth and increased the antitumour activity of chemotherapy, radiation, and biologic agents in xenograft models. In addition, activation of the IGF-1R pathway has been postulated as a mechanism of signalling escape from other anticancer treatments including hormones and targeted agents, including CDK4/6 inhibitors.

In this regard, a drug synergy screen and network modelling in dedifferentiated liposarcoma recently identified CDK4 and IGF-1R as synergistic drug targets (R16-0845). Further experiments confirmed that combined inhibition of CDK4 and IGF-1R cooperatively suppresses the activation of proteins within the AKT pathway. These data suggest that dual

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

blockade of CDK4 and IGF1R signalling results in cooperativity such that two prosurvival pathways are inhibited.

More recently, Heilman and co-workers found that concurrent targeting of CDK4/6 and IGF-1R resulted in synergistic effects on proliferation of CDKN2A-mutant PaC cell lines in vitro and potent suppression of tumour growth in vivo, suggesting that alterations in these pathways converge to promote the growth of CDKN2A-deleted PaC cells (R16-0844).

This study therefore aims to determine the safety, toxicity and recommended phase II dose (RP2D) as well as potential early efficacy signals for the further development of the combination therapy of xentuzumab and abemaciclib in a variety of cancers with a high unmet medical need, especially NSCLC. In an attempt to further improve outcomes for patients with HR+ BC, the combination of abemaciclib, xentuzumab and hormonal therapy (fulvestrant) is also investigated in this trial in expansion cohorts to determine the RP2D and efficacy for that triple combination. After the US FDA's approval of abemaciclib in combination with fulvestrant and based on the above mentioned potential synergy with supports the triple combination (xentuzumab, abemaciclib, and endocrine therapy), expansion cohorts in patients HR-positive, HER2-negative advanced or metastatic breast cancer will be added to this trial to evaluate the efficacy and safety of triple combination of xentuzumab, abemaciclib, and fulvestrant. Early efficacy signal of addition of xentuzumab to new standard-of-care could be obtained in the expansion cohorts.

#### 2.2 TRIAL OBJECTIVES

## For each dose finding cohorts (A, B, C and D):

The primary objective of each dose finding cohort is to determine the maximum tolerated dose (MTD) / recommended phase II dose (RP2D) of xentuzumab in combination with abemaciclib with or without hormonal therapy (letrozole, anastrozole, fulvestrant). Dose limiting toxicities (DLT) will be assessed during the first treatment cycle to assess the MTD/RP2D.

In case that no MTD is reached a RP2D dose will be determined taking into account safety data and other available information. This will be agreed with the Steering Committee.

# For each expansion cohorts (E, F, D1 and D2):

The objective of the cohort E is to assess the anti-tumour activity of xentuzumab in combination with abemaciclib in patients with non-small cell lung cancer.

Cohort F will assess the anti-tumour activity of the triplet combination xentuzumab / abemaciclib and fulvestrant in a single-arm expansion group of patients with locally advanced / metastatic hormone receptor positive (HR+) HER2- breast cancer who have progressed following prior therapy with an aromatase inhibitor and a different CDK4/6 inhibitor (excluding abemaciclib).

The primary objective of cohorts D1 and D2 is to assess the anti-tumour activity of the triplet combination xentuzumab, abemaciclib and fulvestrant in patients with locally advanced / metastatic HR+ breast cancer who have progressed on prior endocrine therapy. Cohort D1

566-10 Trial Protocol


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

will assess the anti-tumos activity for subjects with visceral metastasis and Cohort D2 for subjects with non-visceral metastasis.

## 2.3 BENEFIT - RISK ASSESSMENT

There is a high unmet medical need for patients with advanced or metastatic HR+ BC and NSCLC, as described in <u>Sections 1.1</u> and <u>2.1</u>. Both abemaciclib and xentuzumab have shown encouraging preliminary anti-cancer activity in early-phase clinical trials.

Therefore, and because this trial will enrol patients without curative therapeutic options, it is believed that patients with solid tumours, NSCLCor HR+ BC treated with xentuzumab plus abemaciclib with or without hormonal background therapy at standard doses will have better efficacy (clinical benefit) compared to abemaciclib with or without hormonal background therapy alone.

#### **Abemaciclib**

Hematologic toxicities including neutropenia, leukopenia, anaemia, and thrombocytopenia have been observed in patients treated with abemaciclib, and causality has been established. Patients will therefore be monitored closely for signs of infection, anaemia, and bleeding. Gastrointestinal toxicities including diarrhoea, nausea, and vomiting have been observed in patients treated with abemaciclib, and causality has been established. Patients will therefore be monitored closely for gastrointestinal side effects. Patients with these symptoms will be evaluated promptly, treated supportively, and monitored closely for sequelae such as dehydration. Because diarrhoea possibly related to abemaciclib has been manageable with standard antidiarrheal agents such as loperamide, early treatment of diarrhoea is recommended in this trial.

#### Xentuzumab

As of 18 January 2019, xentuzumab was well tolerated in clinical trials, with no relevant specific side effects reported. The type and pattern of adverse events (AEs) observed to date have generally been of mild to moderate intensity (CTCAE Grades 1 or 2) or consistent with the safety profile of combination backbone treatment or consistent with the underlying neoplastic conditions of patients enrolled on the study. The most frequently reported AEs for xentuzumab monotherapy were fatigue, decreased appetite, nausea, diarrhoea, and vomiting.

Infusion-related reaction (IRR) is a listed side effect of xentuzumab treatment. There have been 3 serious IRRs reported. One event was Grade 3 or higher. All events recovered with management per protocol. Only 1 patient discontinued the study due to an infusion-related reaction. Infusions of xentuzumab should be administered under close supervision of a medically qualified staff member with availability of resuscitation facilities. As mannitol is


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

used in the formulation of xentuzumab, infusion durations of less than one hour should be avoided. Following each infusion, a one hour observation period is recommended.

Infusion reactions will be graded and treated following standard of care or local guidance in this trial.

Although rare, a potential for drug-induced liver injury (DILI) is under constant surveillance by sponsors and regulators. Therefore, this trial requires timely detection, evaluation, and follow-up of laboratory alterations in selected liver laboratory parameters to ensure patients' safety, see also Section 5.3.6.1.

More information about the known and expected benefits, risks, and reasonably anticipated adverse events (AEs) of abemaciclib and xentuzumab may be found in the Investigators' Brochures (IBs) (see current versions). Information on AEs expected to be related to the investigational product may be found in Section 7 of the IBs. Information on serious adverse events (SAEs) expected in the study population independent of drug exposure and that will be assessed by the sponsor in aggregate, periodically during the course of the study, may be found in Sections 6 (Effects in Humans) of the IBs.

The sponsor, monitor, and investigators will perform this study in compliance with the protocol, good clinical practice (GCP) and International Conference on Harmonisation (ICH) guidelines, and applicable regulatory requirements.

During the trial, investigators are advised to manage treatment-related side-effects proactively. Suggested supportive care measures for the management of treatment related AEs and instructions for dose reductions for individual patients are provided in Section 4.4 Regular and frequent assessment of clinical benefit throughout the trial will ensure that any patient not deriving clinical benefit will be withdrawn from the trial treatment. The safety of all patients, dose selection and benefit/risk assessment are under frequent surveillance by a Steering Committee (SC) (refer to Section 3.1.1). The SC will carefully assess the observed benefits and adverse events and give advice on potential treatment discontinuation.

Based on the good safety profiles of xentuzumab and abemaciclib, as well as standard hormonal therapy with letrozole, anastrozole or fulvestrant, as single agents, it is expected that the combination treatment can be safely initiated at the doses specified in Section 4.1.2.

As part of the trial, patients are required to provide blood samples and archival tumour tissue to analyse candidate predictive biomarkers, pharmacokinetics and immunogenicity. For blood samples, in some instances this is already becoming standard clinical practice at specialised oncology centres, but for some patients this will be an additional procedure compared to routine clinical practice. Apart from that, there are no invasive procedures in addition to standard oncology practice.

Based on the disease under study, the inclusion of women of childbearing potential, using contraception as described in <u>Section 4.2.2.3</u>, in this study is justified. To minimize the risk of unintentional exposure of an embryo or foetus to the investigational drug, men and women of childbearing potential must agree to the requirements for pregnancy testing and contraceptive methods described in this protocol.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Based on previous experiences with these drugs, the side effect profile is predictable and manageable for each compound. Safe doses will be established for each set of combination partners during the dose finding parts of the trial. It is expected that those combinations will improve the efficacy of abemaciclib in NSCLC as well as abemaciclib in combination with hormonal therapy in HR+ BC (i.e. letrozole, anastrozole, fulvestrant) by delaying or reversing the resistance mechanisms to these drugs. Additionally, abemaciclib and xentuzumab have exhibited preliminary activity signal in cancers with a high unmet medical need for a new treatment armamentarium.

Based on the pharmacological mechanism and existing non-clinical and clinical data, there is currently no definitive evidence that xentuzumab, either as monotherapy or in combination with abemaciclib/endocrine therapy, will increase the occurrence or worsen the outcomes of a COVID-19 infection. In the target population of patients with advanced or metastatic breast cancer and progression on at least one prior endocrine based regimen, the benefit-risk assessment for xentuzumab remains positive also in the presence of a COVID-19 outbreak. The decision on whether to continue study drugs if a patient develops COVID-19 will be left to the investigator's benefit/risk assessment on a case-by-case basis. Based on laboratory data and any adverse event that may occur, the clinical trial protocol include guidance for continuation, interruption, dose reduction, and discontinuation of study drugs.

In conclusion, given the good tolerability profile, non-overlapping and manageable toxicities as well as preliminary activity of abemaciclib and xentuzumab as well as the established hormonal therapy (letrozole, anastrozole, fulvestrant) in the aforementioned life-threatening cancers with high unmet medical need, the potential benefits expected from xentuzumab in combination with abemaciclib with or without hormonal background therapy are anticipated to outweigh its risks.

The 1280-0022 phase II trial recently completed primary endpoint analysis and showed no added benefit of xentuzumab compared to placebo, in patients with everolimus and exemestane backbone therapy, when treating trial participants with metastatic breast cancer, HR+, HER2-and non-visceral disease. No new safety signals were observed with the addition of xentuzumab to the everolimus and exemestane combination.

In consideration of these top line results of 1280-0022, as of 19 October 2021, Boehringer Ingelheim recommended to immediately discontinue xentuzumab treatment. Sites were also recommended to discontinue associated assessments, including central laboratory sampling.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 3. DESCRIPTION OF DESIGN AND TRIAL POPULATION

#### 3.1 OVERALL TRIAL DESIGN AND PLAN

This trial is an open-label, non-randomised, phase Ib international, multicentre study of the combination of xentuzumab and abemaciclib (doublet) with or without a background of hormonal therapy, such as 2.5 mg letrozole or 1 mg anastrozole or 500 mg fulvestrant (referred to as triplets).

The study consists of

- 4 dose finding cohorts (A, B, C, D (dose finding)) and
- 4 expansion cohorts (E, F, D1 and D2)

The different dose levels to be used at each cohort are described under <u>Section 4.1.2.</u> The study will be conducted, chronologically, in 3 parts:

#### Part 1

Cohort A is a dose finding cohort in approximately 12 evaluable patients to determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D<sub>1</sub>) of the doublet xentuzumab and abemaciclib in solid tumours. Once the RP2D<sub>1</sub> has been established Part 2 of this trial will commence.

# Part 2 (all cohorts in part 2 can be conducted in parallel)

Cohort B is a dose finding cohort in approximately 12 evaluable patients to determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D<sub>2</sub>) of the triplet xentuzumab and abemaciclib and letrozole in breast cancer.

Cohort C is a dose finding cohort in approximately 12 evaluable patients to determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D<sub>3</sub>) of the triplet xentuzumab and abemaciclib and anastrozole in breast cancer.

Cohort D (dose finding) is a triplet-dose finding investigation in approximately 12 evaluable patients to determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D<sub>4</sub>) of the triplet xentuzumab and abemaciclib and fulvestrant in breast cancer. Once the RP2D<sub>4</sub> has been established Part 3 of this trial will commence.

Cohort E is a single arm expansion in 20 NSCLC patients evaluable for response based on the abemaciclib and xentuzumab doublet RP2D<sub>1</sub> as defined in Cohort A.

# Part 3

Cohort F will investigate the efficacy of the triplet combination with fulvestrant at the RP2D<sub>4</sub> of the abemaciclib and xentuzumab and fulvestrant triplet, as defined by cohort D data, in a single arm expansion cohort in 20 breast cancer patients evaluable for response. Based on the subgroup findings from the previous study 1280.4 (see Section 1.2), cohort F will recruit patients without visceral disease.

Cohort D1 and Cohort D2 will be opened once the RP2D4 of Cohort D (dose finding) has been determined. At least 30 patients will be treated to evaluate anti-tumour activity, safety, and pharmacokinetics of the triplet combination in Cohorts D1 and D2. Cohort D1 will recruit patients with visceral metastasis (at least one visceral metastasis) and Cohort D2 will recruit patients with non-visceral metastasis (absence of visceral metastasis). Visceral metastasis is


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

defined as lung, liver, pleural, peritoneal, malignant pleural effusion and malignant peritoneal effusion involvement (i.e. an internal organ in the great cavity of the trunk proper) at the time of study entry.



Figure 3.1:1 Trial Design

#### For dose finding cohorts A, B, C and D:

There are 4 dose-finding cohorts in this trial (i.e. cohorts A, B, C, and D). Each of them may end-up to a different RP2D (i.e. RP2D<sub>1</sub>, RP2D<sub>2</sub>, RP2D<sub>3</sub> and RP2D<sub>4</sub>, respectively). For each dose finding cohort, dose (de-)escalation is guided by a Bayesian logistic regression model (BLRM) with overdose control (R13-4803) that will be fitted to binary toxicity outcomes. For further details, please refer to Section 4.1.2 and Section 7.1.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



Figure 3.1:2 Trial plan for patients in Cohorts A, B, C, D (dose finding), D1, D2 and F



Figure 3.1:3 Trial plan for patients in Cohort E

#### 3.1.1 Administrative structure of the trial

The trial is sponsored by Boehringer Ingelheim (BI).

A Coordinating Investigator is responsible to coordinate Investigators at different centres participating in this multicentre trial. Tasks and responsibilities are defined in a contract.

Boehringer Ingelheim has appointed a Trial Clinical Monitor, responsible for coordinating all required activities, in order to

- manage the trial in accordance with applicable regulations and internal SOPs,

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- direct the clinical trial team in the preparation, conduct, and reporting of the trial,
- ensure appropriate training and information of local clinical monitors (CML), Clinical Research Associates (CRAs), and Investigators of participating countries.

The organisation of the trial in the participating countries will be performed by the respective local or regional BI-organisation (Operating Unit, OPU) in accordance with applicable regulations and internal SOPs, or by a Contract Research Organisation (CRO) with which the responsibilities and tasks will have been agreed and a written contract filed before initiation of the clinical trial.

Data Management and Statistical Evaluation will be done by BI according to BI SOPs.

Tasks and functions assigned in order to organise, manage, and evaluate the trial are defined according to BI SOPs. A list of responsible persons and relevant local information can be found in the ISF.

A Steering Committee (SC) consisting of independent experts and sponsor representatives will be established to support the Coordinating Investigator who will be the chair of the Steering Committee. The composition and the frequency of the meetings of the SC will be documented in the Trial Master File (TMF). The tasks and responsibilities will be agreed in contracts between the SC members and the sponsor and also summarised in an SC-charter filed in the TMF. The Steering Committee will monitor the trial on a regular basis (all operational aspects, recruitment issues, data quality, etc.) and will be responsible for advising on the escalation/deescalation in the dose finding cohorts and the different RP2D's. The SC can also advice to stop a cohort or the trial based on the emerging clinical trial data.

BI will appoint CROs and independent service providers for special services such as central laboratory services for biomarker testing and part of bioanalytical testing, biosample collection and logistics, and Interactive Response Technologies (IRT) for trial medication logistics. The analysis of biomarker and PK will be performed by BI or a CRO appointed by BI.

On-site monitoring will be performed by BI or Contract Research Organisations (CRO) appointed by BI.

All trial relevant documentation will be stored in the (e-) trial master file (e-TMF) at BI. In addition each site will have an Investigator Site File (ISF) containing all trial documents relevant for the site.

Relevant documentation on the participating (Principal) Investigators and other important participants, including their curricula vitae, will be filed in ISF.

# 3.2 DISCUSSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF CONTROL GROUP(S)

This is an open-label, phase Ib study consisting of 4 dose finding cohorts and 4 expansion cohorts. An open-label design is standard for a dose finding study. Inclusion of a control group is not required for this investigation.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

As no data on the optimal dose for the xentuzumab/abemaciclib combination therapy exist so far, the study will first determine the MTD<sub>1</sub>/RP2D<sub>1</sub> of the double drug regimen (in Part 1 cohort A) prior to further exploring its anti-tumour activity in Part 2.

The dose escalation/de-escalation steps and the dose-level cohort sizes (in each dose finding cohort) will be determined based on the recommendation of the SC, guided by a Bayesian model with overdose control. A potential escalation with overdose control design will increase the flexibility in terms of intermediate dose levels and number of patients in each dose-level cohort. This will increase the chance of treating patients at efficacious doses, while reducing the risk of overdosing. This design is not only an efficient method for dose finding studies, but also for dose confirmation studies due to its flexibility to react to unforeseen toxicity rates (R13-4802). This design is based on practical experience and is an efficient method due to its ability to identify the dose with a desired toxicity rate and its allocation of a greater proportion of patients to doses at, or close to, that desired dose (R13-4802, R13-4804, R13-4805). The use of Bayesian models for Phase I studies has also been advocated by the EMA guideline on small populations (R07-4856) and by the FDA (R16-2270).

In expansion cohorts, a single arm design is justified as the trial is exploratory in its design to generate safety and efficacy data. If a positive efficacy signal is observed in this trial, a comparative trial may be considered if deemed justified.

The primary endpoint of the expansion cohorts is Objective Response (OR) or PFS rate, which is a well-accepted endpoint for such studies. OR rate defined as the proportion of patients with tumor size reduction of a predefined amount and for a minimum time period is used as primary endpoint for cohort E and F. PFS18 defined as the proportion of patients who were absence of disease progression or death at 18<sup>th</sup> month is use as primary endpoint for cohorts D1 and D2. A good response of sufficient duration is reasonably likely surrogate for clinical benefit in refractory solid tumour indications or where there is no effective therapy.

PK assessments in the dose escalation cohorts (A, B, C, D (dose finding)) will be limited to the assessment of immunogenicity (anti-drug antibodies ADA) together with a concomitant PK sample for xentuzumab. The basic PK properties of each of the components have been described already.

The potential development of ADAs (immunogenicity against xentuzumab) will be monitored in all patients throughout the trial duration and beyond this (at EOTV and FUV). Regulatory guidelines recommend the monitoring of immunogenicity before, during and beyond treatment. A concomitant PK sample is necessary in order to assess whether an ADA sample result is conclusive or not and to monitor whether any effects of potential ADAs affect the drug concentration.

According to guidelines, combination therapies in oncology should be assessed for their potential effects on the exposure of each other. Therefore, PK investigations of the combination therapies in the trial will be conducted in the expansion cohort E for abemaciclib with xentuzumab and in the expansion cohorts D1 and D2 for fulvestrant with xentuzumab in an exploratory fashion. This approach ensures that a certain number of patients, treated at the same dose, can be evaluated. An intraindividual assessment of the PK of abemaciclib with and without xentuzumab treatment is planned for cohort E. These investigations are performed when the drug to be investigated is at steady state. In order to reach steady state levels with the


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

mono-treatment abemaciclib, a Run-in phase of 9 days is necessary. The assessment of the PK of the combination is planned to be performed at steady state as well. Xentuzumab reaches steady state after around 30d, therefore, the assessment of the combination treatment will be conducted in the second treatment cycle (that is >28 days after the first xentuzumab infusion). The exposure of xentuzumab will be evaluated descriptively and only a historical comparison to mono-treatment with xentuzumab will be done.

In cohorts D1 and D2 no intraindividual comparison of abemaciclib is planned. Exposure to abemaciclib, fulvestrant and xentuzumab is to be evaluated descriptively and only compared across cohorts or to historical or literature data for fulvestrant.

# 3.3 SELECTION OF TRIAL POPULATION

A log of all patients enrolled into the trial (i.e. who have signed informed consent) will be maintained in the ISF at the investigational site irrespective of whether they have been treated with investigational drug or not.

It is estimated that a total of about 148 evaluable patients will be necessary to determine the MTD or the Recommended Phase II Dose, pharmacokinetics and efficacy of xentuzumab and abemaciclib with or without background hormone treatment.

Part 1 of the trial will be conducted in about 3-6 sites in US, Europe and Japan. Parts 2 and 3 of the trial will be conducted in about 40 sites in US, Europe and Japan. If needed, sites from other regions may also participate. Each site is expected to enrol about one to five patients. If site(s) are unable to recruit patients, additional sites may be opened and underperforming sites may be closed.

## 3.3.1 Main diagnosis for trial entry

Patients to be included in this trial must have diagnosed and histologically, or cytologically, confirmed advanced and/or metastatic, measurable or evaluable, non-resectable solid tumours (Cohort A), or diagnosed and histologically, or cytologically, confirmed locally advanced and/or metastatic HR+ HER2- breast cancer (Cohorts B, C, D (dose finding), F, D1 and D2), or diagnosis of stage IV NSCLC (Cohort E).

Patients must not have received prior anti CDK agents (except cohort F) or previous treatment with IGF-1R targeting compounds in any setting.

Please refer to <u>Section 8.3.1</u> (Source Documents) for the documentation requirements pertaining to the in- and exclusion criteria.

## 3.3.2 Inclusion criteria

## **Cohort A (Solid Tumours)**

1. Age  $\geq$  18 years ( $\geq$ 20 years for Japan only) at screening


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 2. Signed and dated written informed consent in accordance with GCP and local legislation prior to admission to the trial
- 3. WHO/ECOG performance status 0-1 assessed at screening
- 4. Patient must be able to swallow oral capsules or tablets.
- 5. Male or female patients ready and able to use highly effective methods of birth control during the study and for 3 weeks following the last dose of abemaciclib per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information. Women of childbearing potential must have a negative serum pregnancy test at screening.
- 6. Patients with histologically or cytologically confirmed diagnosis of advanced and/or metastatic, measurable or evaluable, non-resectable solid tumours
- 7. Patients must have received and failed, or have been intolerant to, all treatment known to confer clinical benefit or have no therapeutic options available as deemed appropriate by their treating physician
- 8. Life expectancy  $\geq$  3 months in the opinion of the investigator assessed at screening;

# **Cohorts B, C, D (dose finding) (Breast Cancer):**

- 1. Age  $\geq$  18 years ( $\geq$ 20 years for Japan only) at screening
- 2. Signed and dated written informed consent in accordance with GCP and local legislation prior to admission to the trial
- 3. WHO/ECOG performance status 0-1 assessed at screening
- 4. Patient must be able to swallow oral capsules or tablets.
- 5. Women who have postmenopausal status due to either surgical/natural menopause or chemical ovarian suppression (initiated at least 28 days prior to Day 1 of Cycle 1) with a gonadotropin-releasing hormone (GnRH) agonist such as goserelin or radiation-induced ovarian suppression.
  - postmenopausal status due to surgical/natural menopause requires at least one of the following conditions:
    - prior bilateral oophorectomy
    - age  $\geq 60$  years
    - age < 60 years and amenorrheic (in the absence of tamoxifen, toremifene, ovarian suppression, or chemotherapy) for at least 12 months; and follicle-stimulating hormone (FSH) and estradiol within the postmenopausal range as per institutional reference ranges.</p>
  - Postmenopausal status due to radiation-induced ovarian suppression must be confirmed by FSH and estradiol level in the postmenopausal range.
- 6. Histologically or cytologically proven diagnosis of breast cancer with evidence of locally advanced disease not amenable to curative resection or metastatic disease
- 7. HR+ (local lab results at screening or, if not available, at the time of diagnosis)

- having experienced menarche and

<sup>&</sup>lt;sup>1</sup> Women of childbearing potential are defined as:

<sup>-</sup> not postmenopausal (12 months with no menses without an alternative medical cause) and

not permanently sterilized (e.g. hysterectomy, bilateral oophorectomy or bilateral salpingectomy).

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

To fulfil the requirement of HR+ disease, the primary tumour or metastatic lesion of the breast cancer must express at least one of the hormone receptors (estrogen receptor [ER] or progesterone receptor [PgR]) by immunohistochemistry (IHC). Estrogen receptor and PgR assays are considered positive if there are at least 1% positive tumour nuclei in the sample as defined in the relevant American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) Guidelines (Hammond et al. 2010).

- 8. HER2 negative (local lab results at screening or, if not available, at the time of diagnosis) as defined by the most recent American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) Guidelines (Hammond et al. 2010).
- 9. Previous adjuvant and neoadjuvant chemotherapy is permitted. 0-2 prior lines of chemotherapy for the metastatic setting are allowed.
- 10. At least 1 lesion (measurable or non-measurable) that can be accurately assessed at baseline with CT or MRI or PET-CT (CT portion of diagnostic quality) and which is suitable for accurate repeated measurement.
- 11. Cohort B, C, D: Must be eligible for the corresponding hormonal therapy (letrozole, anastrozole or fulvestrant). For Cohorts B and C previous treatment with fulvestrant or exemestane is allowed. For Cohort D prior therapy with non steroidal aromatase inhibitors (anastrozole, letrozole) or exemestane are permitted.

## **Cohort E (NSCLC):**

- 1. Age  $\geq$  18 years ( $\geq$ 20 years for Japan only) at screening
- 2. Signed and dated written informed consent in accordance with GCP and local legislation prior to admission to the trial
- 3. WHO/ECOG performance status 0-1 assessed at screening
- 4. Patient must be able to swallow oral capsules or tablets.
- 5. Male or female patients ready and able to use highly effective methods of birth control during the study and for 3 weeks following the last dose of abemaciclib per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information. Women of childbearing potential<sup>2</sup> must have a negative serum pregnancy test at screening.
- 6. Histologically or cytologically confirmed diagnosis of stage IV NSCLC.
- 7. The participant must have progressed after platinum-based chemotherapy AND immunotherapy (unless deemed inappropriate candidates for immunotherapy by their treating physician) AND have received 1 or a maximum of 2 other prior chemotherapy for advanced and/or metastatic disease OR must be judged by the physician as ineligible for further standard second-line chemotherapy. Prior treatment with epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI) and anaplastic lymphoma kinase (ALK) inhibitors is mandatory in participants whose tumour has EGFR-activating mutations or ALK translocations. Prior targeting agents and neoadjuvant/adjuvant therapies are permitted.
- 8. Have adequate organ function including haematology, renal, and liver.
- 9. Have measureable disease per RECIST 1.1.

<sup>&</sup>lt;sup>2</sup> Women of childbearing potential are defined as:

<sup>-</sup> having experienced menarche and

<sup>-</sup> not postmenopausal (12 months with no menses without an alternative medical cause) and

<sup>-</sup> not permanently sterilized (e.g. hysterectomy, bilateral oophorectomy or bilateral salpingectomy).

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# **Cohort D1, Cohort D2 and Cohort F (Breast Cancer):**

- 1. Age ≥ 18 years (≥20 years for Japan only) at screening
- 2. Signed and dated written informed consent in accordance with GCP and local legislation prior to admission to the trial
- 3. WHO/ECOG performance status 0-1 assessed at screening
- 4. Patient must be able to swallow oral capsules or tablets.
- 5. Women who have postmenopausal status due to either surgical/natural menopause or chemical ovarian suppression (initiated at least 28 days prior to Day 1 of Cycle 1) with a gonadotropin-releasing hormone (GnRH) agonist such as goserelin or radiation-induced ovarian suppression.
  - postmenopausal status due to surgical/natural menopause requires at least one of the following conditions:
    - prior bilateral oophorectomy
    - age  $\geq$  60 years
    - age < 60 years and amenorrheic (in the absence of tamoxifen, toremifene, ovarian suppression, or chemotherapy) for at least 12 months; and follicle-stimulating hormone (FSH) and estradiol within the postmenopausal range as per institutional reference ranges.</p>
  - Postmenopausal status due to radiation-induced ovarian suppression must be confirmed by FSH and estradiol level in the postmenopausal range.
- 6. Histologically or cytologically proven diagnosis of breast cancer with evidence of locally advanced disease not amenable to curative resection or metastatic disease
- 7. HR+ (local lab results at screening or, if not available, at the time of diagnosis)

  To fulfil the requirement of HR+ disease, the primary tumour or metastatic lesion of the breast cancer must express at least one of the hormone receptors (estrogen receptor [ER] or progesterone receptor [PgR]) by immunohistochemistry (IHC). Estrogen receptor and PgR assays are considered positive if there are at least 1% positive tumour nuclei in the sample as defined in the relevant American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) Guidelines (Hammond et al. 2010).
- 8. HER2 negative (local lab results at screening or, if not available, at the time of diagnosis) as defined by the most recent American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) Guidelines (Hammond et al. 2010).
- 9. Have a negative serum pregnancy test at baseline (within 14 days prior to randomization) and agree to use medically approved precautions to prevent pregnancy during the study and for 3 weeks following the last dose of abemaciclib and for at least 6 months after last dose of xentuzumab if postmenopausal status is due to ovarian suppression with a GnRH agonist.
- 10. Have either measurable disease or non-measurable bone only disease. Measurable and nonmeasurable diseases are defined according to the Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1 [v1.1]. Nonmeasurable bone only disease may include any of the following: blastic bone lesions, lytic bone lesions without a measurable soft tissue component, or mixed lytic-blastic bone lesions without a measurable soft tissue component.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## Cohort D1 and D2 only:

11. Patients must fulfil 1 of the following criteria:

- a. Relapsed with radiologic evidence of progression while receiving neoadjuvant or adjuvant endocrine therapy, with no subsequent endocrine therapy received following progression.
- b. Relapsed with radiologic evidence of progression within 1 year from completion of adjuvant endocrine therapy, with no subsequent endocrine therapy received following progression.
- c. Relapsed with radiologic evidence of progression more than 1 year from completion of adjuvant endocrine therapy and then subsequently relapsed with radiologic evidence of progression after receiving treatment with either an antiestrogen or an aromatase inhibitor as first-line endocrine therapy for metastatic disease. Patients may not have received more than 1 line of endocrine therapy or any prior chemotherapy for metastatic disease.
- d. Presented de novo with metastatic disease and then relapsed with radiologic evidence of progression after receiving treatment with either an antiestrogen or an aromatase inhibitor as first-line endocrine therapy for metastatic disease. Patients may not have received more than 1 line of endocrine therapy or any prior chemotherapy for metastatic disease.
- 12. For cohort D1 (visceral disease) patient must have at least one documented visceral metastasis; for cohort D2 (non-visceral disease), patient must not have any visceral metastasis.

## **Cohort F only:**

- 13. Patients with resistance to prior therapy with an aromatase inhibitor (AI) and CDK4/6 inhibitor (excluding abemaciclib) for locally advanced or metastatic breast cancer, defined as radiologic evidence of disease progression while on, or within 30 days after last dose of AI and/or CDK4/6 inhibitor (excl. abemaciclib) administered as first-line therapy for locally advanced or metastatic disease. Patients may not have received more than 1 line of prior endocrine based therapy or any prior chemotherapy for advanced/metastatic disease.
- 14. Patient must not have any visceral metastasis (example of allowed lesions are in breast, lymph nodes, soft tissue, bone).

#### 3.3.3 Exclusion criteria

# Cohorts A, B, C, D (dose finding), and E:

- 1. Any documented active or suspected malignancy or history of malignancy, other than the disease under study, within 3 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix or ductal carcinoma in situ (DCIS) if properly treated in opinion of the investigator.
- 2. Patients who must or wish to continue the intake of restricted medications (see <u>Section 4.2.2.1</u>) or any drug considered likely to interfere with the safe conduct of the trial
- 3. Previous treatment in this trial

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 4. Currently enrolled in another investigational device or drug study, or less than 21 days since ending another investigational device or drug study(s), or receiving other investigational treatment(s).
- 5. Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes them an unreliable study subject or unlikely to complete the trial
- 6. Women who are pregnant, nursing, or who plan to become pregnant while in the trial. Men who plan to father a child while in the trial.
- 7. Prior anti-cancer chemotherapy, biological or radiation therapy, androgens, thalidomide, other anticancer agents, or any investigational drug within 21 days (14 days for non-myelosuppressive agents); and/or 4 weeks for immunotherapy, before starting any of the trial drugs.
- 8. Prior anti CDK agents
- 9. Prior radiotherapy to  $\geq 25\%$  of bone marrow regardless of when it was received
- 10. Unresolved treatment related toxicity from previous therapy of > CTCAE grade 1 at study entry (except for stable sensory neuropathy ≤ CTCAE grade 2 and alopecia)
- 11. Previous treatment with IGF-1R targeting compounds
- 12. Known active uncontrolled or symptomatic CNS metastases, carcinomatous meningitis, or leptomeningeal disease, as indicated by clinical symptoms, cerebral oedema, and/or progressive growth. History of CNS metastases or cord compression are eligible if they have been definitively treated (e.g. radiotherapy, stereotactic surgery) and are clinically stable, off anticonvulsants and steroids for at least 4 weeks. Patients with brain metastases are eligible if they are asymptomatic, completed radiotherapy for at least 4 weeks or are on a stable dose of steroids for at least 4 weeks. Patients are not eligible if they have spinal cord compression.
- 13. The patient has serious and/or uncontrolled pre-existing medical condition(s) that, in the judgement of the Investigator, would preclude participation in this study, including interstitial lung disease, severe dyspnoea at rest or requiring oxygen therapy.
- 14. Inadequate bone marrow reserve or organ function as demonstrated by any of the following: ANC < 1.5 x 10<sup>9</sup>/L, platelets < 100 x 10<sup>9</sup>/L, haemoglobin <90g/L, ALT > 2.5 x ULN or > 5 x ULN in the presence of liver metastases, total bilirubin >1.5 x ULN or >3 x ULN in patients with Gilbert's Syndrome, serum creatinine > 1.5 x ULN concurrent with creatinine clearance ≤ 50 mL/min.
- 15. Pre-existing renal disease including glomerulonephritis, nephritic syndrome, Fanconi Syndrome or renal tubular acidosis
- 16. Refractory nausea and vomiting, chronic GI diseases, inability to swallow the product, or previous significant bowel resection that would preclude adequate absorption of abemaciclib or resulting in baseline Grade 2 or higher diarrhoea.
- 17. History of hypersensitivity to active or inactive excipients of xentuzumab, abemaciclib or letrozole/anastrozole/fulvestrant, or loperamide hydrochloride, or drugs with similar chemical structures
- 18. Patients with Diabetes Type I or uncontrolled Type II (defined by HgBA1C > 8%).
- 19. Patients with advanced/metastatic, symptomatic, visceral spread, that are at risk of life-threatening complications in the short term including patients with massive uncontrolled effusions (pleural, pericardial, peritoneal), pulmonary lymphangitis, and over 50% of liver involvement in metastases.
- 20. Prior hematopoietic stem cell or bone marrow transplant

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 21. Have a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia (including but not limited to ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest. Subjects with controlled atrial fibrillation for >30 days prior to study treatment are eligible.
- 22. Erythropoietin, G-CSF, and GM-CSF are not allowed within 2 weeks prior to study. The primary prophylactic use of G-CSF is not permitted but it may be used to treat treatment-emergent neutropenia.
- 23. Have had major surgery (excluding biopsy) < 28 days of the initial dose of any of the study drugs or planned major surgery during study participation.
- 24. Have active bacterial or fungal infection (that is, requiring IV antibiotics or therapy at time of initiating study treatment), and/or known viral infection (for example, human immunodeficiency virus [HIV] antibodies, hepatitis B surface antigen, or hepatitis C antibodies). Screening is not required for enrolment.
- 25. Patients with baseline Grade ≥2 hyperglycaemia or patients with baseline Grade ≥ 2 diarrhoea
- 26. Patients needing treatment with CYP3A4 inhibitors/inducers cannot be included in the trial. (See <u>Appendix 10.1</u>)

## Cohort D1, Cohort D2 and Cohort F (Breast Cancer):

- 1. Any documented active or suspected malignancy or history of malignancy (including inflammatory breast cancer), other than the disease under study, within 3 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix or ductal carcinoma in situ (DCIS) if properly treated in opinion of the investigator.
- 2. Patients who must or wish to continue the intake of restricted medications (see <u>Section 4.2.2.1</u>) or any drug considered likely to interfere with the safe conduct of the trial
- 3. Previous treatment in this trial
- 4. Currently enrolled in another investigational device or drug study, or less than 21 days since ending another investigational device or drug study(s), or receiving other investigational treatment(s).
- 5. Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes them an unreliable study subject or unlikely to complete the trial
- 6. Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
- 7. Prior anti-cancer chemotherapy, biological or radiation therapy, androgens, thalidomide, other anticancer agents, or any investigational drug within 21 days (14 days for non-myelosuppressive agents); and/or 4 weeks for immunotherapy, before starting any of the trial drugs. For cohort F only: prior palbociclib or ribociclib treatment within 14 days before starting any of the trial drugs.
- 8. Have received prior treatment with chemotherapy (except for neoadjuvant/adjuvant chemotherapy), fulvestrant, everolimus, alpelisib or abemaciclib. For cohorts D1 and D2 only: prior treatment with palbociclib or ribociclib is also excluded
- 9. Prior radiotherapy to  $\geq 25\%$  of bone marrow regardless of when it was received
- 10. Unresolved treatment related toxicity from previous therapy of > CTCAE grade 1 at study entry (except for stable sensory neuropathy ≤ CTCAE grade 2 and alopecia)
- 11. Previous treatment with IGF-1R targeting compounds
- 12. Have clinical evidence or history of central nervous system metastasis. Screening is not required for enrolment.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 13. The patient has serious and/or uncontrolled pre-existing medical condition(s) that, in the judgement of the Investigator, would preclude participation in this study, including interstitial lung disease, severe dyspnoea at rest or requiring oxygen therapy.
- 14. Inadequate bone marrow reserve or organ function as demonstrated by any of the following: ANC < 1.5 x 10<sup>9</sup>/L, platelets < 100 x 10<sup>9</sup>/L, haemoglobin <90g/L, ALT > 2.5 x ULN or > 5 x ULN in the presence of liver metastases, total bilirubin >1.5 x ULN or >3 x ULN in patients with Gilbert's Syndrome, serum creatinine > 1.5 x ULN concurrent with creatinine clearance < 50 mL/min.
- 15. Pre-existing renal disease including glomerulonephritis, nephritic syndrome, Fanconi Syndrome or renal tubular acidosis
- 16. Refractory nausea and vomiting, chronic GI diseases, inability to swallow the product, or previous significant bowel resection that would preclude adequate absorption of abemaciclib or resulting in baseline Grade 2 or higher diarrhoea.
- 17. History of hypersensitivity to active or inactive excipients of xentuzumab, abemaciclib or fulvestrant, or loperamide hydrochloride, or drugs with similar chemical structures
- 18. Patients with Diabetes Type I or uncontrolled Type II (defined by HgBA1C > 8%).
- 19. Patients with advanced/metastatic, symptomatic, visceral spread, that are at risk of life-threatening complications in the short term including patients with massive uncontrolled effusions (pleural, pericardial, peritoneal), pulmonary lymphangitis, and over 50% of liver involvement in metastases.
- 20. Prior hematopoietic stem cell or bone marrow transplant
- 21. Have a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia (including but not limited to ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest. Subjects with controlled atrial fibrillation for >30 days prior to study treatment are eligible.
- 22. Erythropoietin, G-CSF, and GM-CSF are not allowed within 2 weeks prior to study. The primary prophylactic use of G-CSF is not permitted but it may be used to treat treatment-emergent neutropenia.
- 23. Have had major surgery (excluding biopsy) < 28 days of the initial dose of any of the study drugs or planned major surgery during study participation.
- 24. Have active bacterial or fungal infection (that is, requiring IV antibiotics or therapy at time of initiating study treatment), and/or known viral infection (for example, human immunodeficiency virus [HIV] antibodies, hepatitis B surface antigen, or hepatitis C antibodies). Screening is not required for enrolment.
- 25. Patients with baseline Grade ≥2 hyperglycaemia or patients with baseline Grade ≥ 2 diarrhoea
- 26. Patients needing treatment with CYP3A4 inhibitors/inducers cannot be included in the trial. (See Appendix 10.1)
- 27. Have initiated bisphosphonates or approved RANK ligand (RANK-L) targeted agents (for example, denosumab) <7 days prior to initiation of any study drug.

## 3.3.4 Removal of patients from therapy or assessments

# 3.3.4.1 Removal of individual patients

An excessive withdrawal rate can have a severe negative impact on the scientific value of the trial. Every effort should be made to keep patients in the trial as scheduled. This includes

66-10 Trial Protocol


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

careful patient selection and appropriate explanation of the trial requirements and procedures prior to enrolment as well as an explanation of the consequences of premature withdrawal.

An individual patient is to be withdrawn from trial treatment if:

- \* The patient withdraws consent for trial treatment or trial participation, without the need to justify the decision.
- \* The patient develops unequivocal disease progression, supported by radiological evidence where possible.
- \* The patient needs to take concomitant drugs that interfere with the investigational product or other trial medication in the opinion of both the investigator and sponsor representative.
- \* The patient can no longer be treated with trial medication for other medical reasons (such as surgery, adverse events, other diseases, or pregnancy)
- The patient has repeatedly shown to be non-compliant with important trial procedures and, in the opinion of both, the investigator and sponsor representative, is not willing or able to stick to the trial requirements in the future. (See Section 4.3)
- \* The trial is terminated for any of the reasons listed in <u>Section 3.3.4.2</u> "Discontinuation of the trial by the sponsor".

Given the patient's agreement, the patient will undergo the procedures for early treatment discontinuation and follow up as outlined in the <u>Flow Chart (FC)</u> and <u>Section 6.2.3</u>. For all patients the reason for withdrawal (e.g. adverse events) must be recorded in the eCRF. These data will be included in the trial database and reported.

# 3.3.4.2 Discontinuation of the trial by the sponsor

Boehringer Ingelheim reserves the right to discontinue the trial overall or at a particular trial site at any time for the following reasons:

- 1. Failure to meet expected enrolment goals overall or at a particular trial site
- 2. Emergence of any efficacy/safety information invalidating the earlier positive benefit-risk-assessment that could significantly affect the continuation of the trial

As described in <u>Section 2.3</u> Benefit-risk assessment, topline results of 1280-0022 showed no added benefit of xentuzumab compared to placebo when treating participants with metastatic breast cancer. Although xentuzumab treatment was recommended to be discontinued in 1280.18, continuation of treatment of patients with xentuzumab was based on an individual assessment by the investigator. Due to the worsening in benefit-risk, the trial will proceed towards termination based on the following 3 steps:

a. For xentuzumab-treated patients, the xentuzumab treatment will not extend past the drug expiration date (May 2023) of the last planned GMP manufacturing batch of IMP xentuzumab (provided that all patients are on xentuzumab for at least 2 years when they are tolerating the drug without tumor progression). Patients that will discontinue xentuzumab can still be eligible for continued treatment with abemaciclib and

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

fulvestrant (standard of care in this setting) provided they are tolerating the drugs without tumor progression.

- b. When all patients have discontinued xentuzumab treatment, if any patient on abemaciclib and fulvestrant is able to continue taking these approved medications off study, then, at the request of the Sponsor, the patient may end such treatment as part of the trial and discontinue study participation (if both the Investigator and patient agree).
- c. After all patients end treatment with all study drugs, the trial will be terminated.
- 3. Violation of GCP, the CTP, or the contract disturbing the appropriate conduct of the trial

The Investigator / the trial site will be reimbursed for reasonable expenses incurred in case of trial termination (except in case of the third reason).

# 3.3.5 Replacement of patients

Patients may be replaced for determination of the primary endpoint (MTD) in cases of:

- Patient's withdrawal during the first cycle of treatment for reasons other than DLT, e.g. patient no longer wishes to participate, or lost to follow up during first cycle.
- Patients who do not experience DLT, but miss more than one dose of xentuzumab during the first cycle of treatment, except for dose interruption caused by AE
- Patients who do not experience DLT, but miss 3 or more consecutive doses of abemaciclib during the first cycle of treatment, except for dose interruption caused by AE.
- Patients who miss one complete cycle at any time beyond the first cycle of treatment may be replaced after discussion between the sponsor and the investigator.
- Patients who are non-evaluable with respect to DLT.
- Patients with CTCAE grade ≥3 allergic reaction/hypersensitivity to the study drug(s) within the first cycle may be replaced.
- For cohorts E and F, where objective response or DC is the primary endpoint: if patient doesn't have post-treatment radiological tumor assessment for reason other than worsening of underlying disease

Patients that have been replaced might continue treatment in the trial should criteria in <u>Section 4.1.4.2</u> apply; however these patients will not be considered for analysis of the primary endpoint.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 4. TREATMENTS

#### 4.1 INVESTIGATIONAL TREATMENTS

Patients will receive xentuzumab plus abemaciclib.

Additionally in cohorts B, C, D (dose finding), F, D1 and D2, patients will receive in addition background hormonal therapy with letrozole, anastrozole or fulvestrant.

The sources for each of the products are listed in Section 4.1.1.

As of 19 Oct 2021, based on the primary analysis of top line results of 1280-0022, Boehringer Ingelheim recommended to immediately discontinue xentuzumab in 1280.18 trial. (see Section 2.3)

# 4.1.1 Identity of the Investigational Medicinal Products

Table 4.1.1: 1 Xentuzumab (Investigational product, IMP)

| Substance: | Xentuzumab humanized monoclonal antibody |
|---|---|
| Pharmaceutical formulation: | Concentrate for solution for infusion |
| Source: | Boehringer Ingelheim Pharma GmbH & Co. KG |
| Unit strength: | 10 mg/ml of xentuzumab supplied in 20 ml vials (200 mg/vial) |
| Posology | Once weekly administrated through one hour intravenous infusion. |
| | Infusion duration may be extended to over one hour and up to a maximum of three hours in cases of grade $\geq 2$ infusion reactions |
| Route of administration: | Intravenous infusion. Appropriate dose of xentuzumab will be diluted in isotonic sodium chloride solution (0.9%) |
| Duration of use: | Continuous weekly dosing (days 1, 8, 15 and 22 in a 28-day course) in the absence of disease progression, intolerable AEs or other reason necessitating withdrawal |

Detailed preparation and handling of xentuzumab, including information on infusion equipment and infusion procedure, will be described in ISF.


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 4.1.1: 2 Abemaciclib (Investigational product, IMP)

| Substance: | Abemaciclib. Small molecule CDK4 and CDK6 inhibitor |
|---|---|
| Pharmaceutical formulation: | Capsules |
| Source: | |
| Unit strength: | A white hypromellose capsule containing <b>50 mg</b> of abemaciclib and the inactive ingredients pregelatinized starch, dimethicone, and colloidal silicon dioxide. |
| Posology | Treatment/28-day cycle 150 mg p.o. Q12H on Days 1-28 (Starting dose Cohort A) Abbreviations: PO = orally; Q12H = every 12 (± 2) hours |
| Route of administration: | p.o. |
| Pharmaceutical formulation: | Tablets |
| Source: | |
| Unit strength: | Film-coated 50 mg tablets |
| Posology | Treatment/28-day cycle 150 mg p.o. Q12H on Days 1-28 (Starting dose Cohort A) Abbreviations: PO = orally; Q12H = every 12 (± 2) hours |
| Route of administration: | p.o. |

Table 4.1.1: 3 Fulvestrant. Background endocrine therapy. (Auxiliary Medicinal Product, AMP)

| Substance: | Fulvestrant (Faslodex®) |
|---|---|
| Pharmaceutical formulation: | Solution for injection |
| Source: | |
| Unit strength: | Prefilled syringes (250 mg fulvestrant in 5mL solution). |
| Route of administration: | Intramuscular injection |

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 4.1.1: 3 (cont.) Fulvestrant. Background endocrine therapy. (Auxiliary Medicinal Product, AMP):

| Substance: | Fulvestrant (Faslodex®) |
|---|---|
| Posology | 500 mg given once a month, with an additional 500-mg dose given two weeks after the first dose. Each dose is given as two slow 250 mg injections lasting one to two minutes, with one injection being given into the muscle of each buttock |
| Route of administration: | Intramuscular injection |

Table 4.1.1: 4 Anastrozole. Background endocrine therapy. (Auxiliary Medicinal Product, AMP)

| Substance: | Anastrozole |
|---|---|
| Pharmaceutical formulation: | Film Coated Tablet |
| Source: | EU, US or Japan commercial product as applicable |
| Unit strength: | 1 mg |
| Posology | 1 mg tablet once a day |
| Route of administration: | p.o. |

Table 4.1.1: 5 Letrozole. Background endocrine therapy. (Auxiliary Medicinal Product, AMP)

| Substance: | Letrozole |
|---|---|
| Pharmaceutical formulation: | Film coated tablet. |
| Source: | EU, US or Japan commercial product as applicable |
| Unit strength: | 2.5 mg |
| Posology | 2.5 mg once daily |
| Route of administration: | p.o. |

# 4.1.2 Selection of doses in the trial

#### 4.1.2.1 Part 1

A semi-mechanistic PK/PD model was developed describing the kinetics of the interaction between xentuzumab and the different PD biomarkers (i.e. IGF-1, IGF-2, and IGFBP3). Simulations using this model indicate that a weekly dosing of 1000 mg xentuzumab reduces free IGF-1 concentration by more than 90% and in addition free IGF-2 by 64 % at trough steady-state relative to pre-treatment; this is considered a relevant biological effect. Therefore, a weekly dose of 1000 mg xentuzumab is considered a suitable dose.


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

In dose finding cohort A, the starting dose of abemaciclib is 150 mg every 12 ( $\pm 2$ ) hours. Based on the recommended phase II dose in one dose finding study using combination of a targeted therapy agent with xentuzumab (please refer to the current version of the Investigator's Brochure,  $\underline{c01690707-08}$ ), a dose level of 1000 mg with weekly dose schedule is selected as the starting dose for this study. This dose combination has a prior probability of overdosing below 25% (see Section 7.1). Planned dose levels for patients in cohort A are displayed in Table 4.1.2.1: 1 below.

Table 4.1.2.1: 1 Concomitant dosing schedule schemes of Cohort A

| Dose level | Xentuzumab (mg weekly) | Abemaciclib (mg/12h) |
|---------------------|------------------------|----------------------|
| DL0 (starting dose) | 1000 | 150 |
| DL-1a | 750 | 150 |
| DL-1b | 1000 | 100 |

Dose escalation beyond the highest dose levels planned as shown above will not be considered. Above dose levels may be modified and/or additional dose levels/administration regimens may be added based on safety profile and other emerging data upon discussion and agreement between the sponsor and the SC.

Intra-patient dose escalation is not permitted. Successive dose-level cohorts of patients will receive doses of xentuzumab in combination with abemaciclib until the  $MTD_1/RP2D_1$  is established or until the trial is terminated for other reasons (see Section 3.3.4.2). The trial may be terminated at any time based on emerging safety concerns without establishing the  $MTD_1/RP2D_1$ .

For any dose-level cohort, at least 3 evaluable patients will be required. However, in the case that only 2 patients are evaluable and neither has experienced a DLT within the MTD evaluation period, then dose-escalation can occur based on these 2 patients.

If DLTs are observed in the first two consecutive patients of a previously untested dose level, subsequent enrolment to that dose-level cohort will be stopped. The BLRM will then be re-run to confirm that the dose level still fulfils the EWOC principle. Based on this information, the SC will evaluate whether the next patients will be enrolled at the same dose level, or if they will be enrolled at a lower dose level.

After all patients in the initial dose-level cohort have either experienced a DLT or have been observed for at least one course (28 days) without experiencing a DLT, the Bayesian model will be updated with the newly accumulated data. The SC will then determine the dose regimen for the next dose-level cohort, based on the available toxicity information (including DLTs, AEs that are not DLTs, and AE information post-cycle 1), recommendations from the BLRM, and other data (e.g. anti-tumour activity, pharmacokinetics) if applicable. Details on the Bayesian design are provided in Sections 7.1 and Appendix 10.6.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The overdose risk will be calculated for each further dose combination, and patient enrolment into dose levels will be permitted to all dose combinations which fulfil the escalation with overdose control (EWOC) criterion. Based on the Bayesian model and the additional information as defined above, the SC will decide on the next dose level to be investigated. In the SC meeting, data for each patient in the current dose-level cohort will be described in detail, updated safety data on other ongoing patients, including data in later courses, will be discussed as well.

The SC must reach a consensus on whether to de-escalate, re-escalate and/or expand recruitment into particular cohorts, or to declare the MTD<sub>1</sub>/RP2D<sub>1</sub>. BI will prepare minutes from the SC meetings and circulate them to each Investigator.

To further assess the safety (e.g. specific suspected treatment-related adverse events) of xentuzumab in combination with abemaciclib, one or several doses that are considered acceptably safe, i.e. shown to be lower than or equal to any potential MTD, may be explored to determine the RP2D<sub>1</sub>. Nevertheless, a minimum of 6 evaluable patients need to be treated at the MTD<sub>1</sub>/RP2D<sub>1</sub> in the dose finding cohort A prior to starting part 2 (cohorts B, C, D and E) and any dose declared as MTD<sub>1</sub>/RP2D<sub>1</sub> by the SC needs to fulfil the escalation with overdose control (EWOC) criteria.

The SC may recommend stopping the dose finding cohort A after the criterion for MTD (Section 7.1) is fulfilled. Further patients may be included to confirm the  $MTD_1/RP2D_1$  estimate, i.e. to confirm that the EWOC criterion is still fulfilled prior to the start of part 2 (cohorts B, C, D and E).

#### 4.1.2.2 Part 2

The decision on dose escalation/de-escalation, MTD (or Biological Relevant Dose) and RP2D will be determined in discussion with at least BI Trial Clinical Monitor, BI project physician (TMM) and Coordinating Investigator and taking into account patients' safety. This decision will be documented.

#### Dose finding cohorts B, C and D (dose finding):

For each cohort, starting dose of xentuzumab and abemaciclib will be the RP2D<sub>1</sub> determined in cohort A, even if RP2D<sub>1</sub> equals the highest dose levels planned (see <u>Table 4.1.2.1: 1</u>). This is because the maximum dose of abemaciclib to be explored in triple combination cohorts is 150mg b.i.d. In that case, the starting dose would then be 1000 mg weekly xentuzumab plus 150 mg / 12h abemaciclib.

In the three cohorts, patients will receive the dose of background hormonal therapy as defined in <u>Tables 4.1.1: 3</u> to <u>4.1.1: 5</u> (i.e. letrozole in cohort B, anastrozole in Cohort C and fulvestrant in cohort D).

Dose escalation/de-escalation of xentuzumab and abemaciclib will be conducted as described in <u>Section 4.1.2.1</u> for cohort A using a BLRM with a fixed dose of the background hormonal therapy.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### **Expansion cohort E:**

Patients will be treated at the RP2D<sub>1</sub> determined in Cohort A.

#### 4.1.2.3 Part 3

## Cohorts F, D1 and D2

For Cohort F and Cohorts D1 and D2 patients will be treated at the RP2D<sub>4</sub> of abemaciclib and xentuzumab and fulvestrant triplet as determined in Cohort D (dose finding).

## 4.1.3 Method of assigning patients to treatment groups

For the dose finding cohorts, the treatment slots are assigned by the BI Clinical Monitor (CM) in close communication (email/phone/fax) with the recruiting sites and IRT system and will be assigned on a competitive basis. After the BI Clinical Monitor has been notified by a site about a potential patient, the slot will be reserved to this site for a period of time (approximately a week) until patient signs ICF, otherwise the slot will be opened up again for all recruiting sites. If more than one site notifies potential patients and there are no slots for all proposed candidates, BI Clinical Monitor will allocate the slot prioritizing by planned visits calendar, balanced number of patients per site and other parameters as applicable.

Patients that meet the eligibility criteria and who have given their written informed consent may not be entered into the study depending on the cohort which is being explored at that particular time (for example, but not restricted to, the dose finding cohort A). This needs to be discussed and agreed with BI Trial Team.

Prior to inclusion of a new patient, once the slot has been confirmed, the investigator should also confirm the respective dose with the BI clinical monitor.

# 4.1.4 Drug assignment and administration of doses for each patient

The treatment medication assignment for xentuzumab and abemaciclib will be managed through IRT system. The treatment medication assignment for anastrozole, letrozole and fulvestrant will be managed through IRT system in certain countries only.

In addition, patient's screening, run-in, all drug dispensation visits and EOTV will be collected in the IRT system.

## 4.1.4.1 Initial study drug assignment and administration

General information that applies in this study regardless of IRT is described in below sections of individual study drug. The medication kit as well as the treatment will be assigned with the support from IRT.

Before entering patients at the next dose level of the dose finding cohorts, it will be ensured that all patients at the current ongoing dose level have completed at least one course of treatment.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### **Xentuzumab**

Patients will start treatment with their assigned dose tier (see Section 4.1.2) or RP2D of xentuzumab from course 1 day 1. Xentuzumab will be administered at the investigator site intravenously over one hour with a constant infusion rate on the treatment day as specified in the Flow Chart. If scheduled infusion of xentuzumab is not performed within the time window, this treatment will be skipped and will not be made up. Subsequent visits should follow the original visit date schedule. Mannitol is used in the formulation of xentuzumab, so infusion duration of less than one hour must be avoided. The infusion time may be extended to over one hour and up to a maximum of three hours in cases of CTCAE grade ≥ 2 infusion reactions. In case of a delay or an interruption of infusion, the reason and the exact time of deviation must be recorded in the specific eCRF. The accuracy of this information is crucial for the proper evaluation and appraisal of the pharmacokinetics – in the relevant cohorts – and other data.

Detailed information of dispensation, preparation, and handling of xentuzumab will be described in ISF.

## **Abemaciclib**

Abemaciclib will be taken orally every  $12 (\pm 2)$  hours on days 1 through 28 of a 28-day cycle for a total of 56 doses per cycle. During all cycles, abemaciclib should be taken at approximately the same times each day. If a patient misses or vomits a dose, that dose should be omitted.

No more than 56 doses of abemaciclib should be dispensed for each 28-day cycle. Abemaciclib dose omissions will be evaluated on a case by case basis and patients may be replaced if dose omissions occur within MTD period of a dose finding cohort or if the number of dose omissions makes the patient non evaluable regardless of the cohort.

# 4.1.4.2 Temporary treatment interruption and dose reduction

DLT, or those AEs requiring dose adjustment as indicated on the label, should be managed by treatment interruptions and subsequent dose reductions of the presumed causal study drug(s) according to the schedule described in <u>Table 4.1.4.2: 1</u>. Please also refer to <u>Section 4.4</u> for additional recommendations.

In case of an intolerable adverse event which is suspected to be related to either xentuzumab or abemaciclib in the opinion of investigator, the treatment can be interrupted with subsequent dose reduction for the suspected agent(s) according to <u>Tables 4.1.4.2: 1</u> (xentuzumab) and <u>4.1.4.2: 2</u> (abemaciclib).

In the case of DLT with suspected overlapping toxicities where assigning relatedness to one study drug or the other is difficult, or considered related to both xentuzumab and abemaciclib the dosing with both study drugs should be held until the adequate resolution of AE (CTCAE grade  $\leq 1$ ). Treatment should then be resumed and/or dose reduced as shown in <u>Table 4.1.4.2: 1</u> for xentuzumab and in <u>Table 4.1.4.2: 2</u> for abemaciclib.

Recurrent in the context of dose interruptions and delays refers to the same event and severity occurring within 8 weeks (as measured from the stop date of the first event). This does not


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

include events in the same class (for example, neutropenia followed by anemia 1 month later).

Further to these recommendations, in Part 1, Cohort A, both xentuzumab and abemaciclib must be paused when a DLT occurs during the first treatment course.

The treatment should be paused until patient has recovered from the DLT to grade  $\leq 1$  or baseline. Baseline is defined as the CTCAE grade at the start of treatment. For patients who develop DLT, treatment may be resumed at reduced dose according to dose reduction scheme of the patient's starting dosage. If a patient has not recovered to Grade  $\leq 1$  or baseline within 28 days, study treatment must be permanently discontinued. In the event that the patient is deriving obvious clinical benefit according to the investigator's judgement, further treatment with study drug(s) will be decided in agreement between the sponsor and the investigator.

If one or more of the study drugs is permanently discontinued, the patient can remain on either abemaciclib or xentuzumab or endocrine therapy only.

Dose reductions will apply to individual patients only. Doses of xentuzumab and/or abemaciclib can be reduced independent of each other. Once the treatment dose of xentuzumab is reduced for a particular patient, it should not be increased back to the previous dose.

Abemaciclib dose adjustments are allowed within a cycle and between cycles. Abemaciclib must be reduced sequentially by one dose level. For further instructions as regards dose adjustments of abemaciclib, please refer to Section 4.2.2.

For patients requiring dose reduction(s) of abemaciclib, any re-escalation to a prior dose level is permitted only after discussion and agreement with the sponsor. After re-escalation, subsequent dose adjustments should be based on the dose of abemaciclib that the patient is currently receiving.

Table 4.1.4.2: 1 Individual dose reductions schedule

| Xentuzumab mg/weekly | | Abemaciclib mg/12 h | |
|---|---|---|---|
| Current dose is 1000 | Dose reduce to 750 | Current dose is 150 | Dose reduce to 100 |
| Current dose is 750 | Dose reduce to 500 | Current dose is 100 | Dose reduce to 50 |
| Current dose is 500 | No further dose reductions allowed. | Current dose is 50 | No further dose reductions allowed. |

No dose reduction is allowed below 500 mg/weekly for xentuzumab or 50 mg b.i.d. for abemaciclib.

Alternative dose modification scheme can only be considered after discussion and agreement between the investigator and the BI clinical monitor.

c09049566-10

04 Mar 2022

**Trial Protocol** 


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

In the event of any unrelated AEs, the study drug(s) may be interrupted for up to 28 days, but no dose reduction should occur. Otherwise, the decision to continue with the study treatment will be made by the BI Clinical Monitor in agreement with the investigator.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 4.1.4.2: 2 Dose Adjustments and Delays for Toxicity Possibly Related to Abemaciclib\*

| Toxicity Type | <b>Toxicity Profile and Severity</b> | <b>Dose Suspension</b> | Dose Reduction |
|---|---|---|---|
| Hematologic Toxicity | Grade 3 | Dose MUST be<br>suspended until toxicity<br>resolves to at least<br>Grade 2. | Dose MAY be reduced by 1 dose level - investigator's discretion. |
| Hematologic Toxicity | Recurrent Grade 3 <sup>1</sup> | Dose MUST be<br>suspended until toxicity<br>resolves to at least<br>Grade 2. | Dose MUST be reduced by 1 dose level. |
| Hematologic Toxicity | Grade 4 | Dose MUST be<br>suspended until toxicity<br>resolves to at least<br>Grade 2. | Dose MUST be reduced by 1 dose level. |
| Hematologic toxicity: If patient requires administration of blood cell growth factors. | Regardless of severity. (Use of growth factors according to ASCO Guidelines) | Dose MUST be<br>suspended for at least<br>48 hours after the last<br>dose of blood cell<br>growth factors was<br>administered and until<br>toxicity resolves to at<br>least Grade 2. | Dose MUST be reduced by 1 dose level unless already performed for incidence of toxicity that led to the use of growth factor. |
| Nonhematologic Toxicity <sup>2</sup> (except diarrhoea, ALT increase and ILD/pneumonitis) | Persistent or recurrent <sup>3</sup> Grade<br>2 that does not resolve with<br>maximal supportive measures<br>within 7 days to baseline or<br>Grade 1 | Dose MUST be<br>suspended until toxicity<br>resolves to either<br>baseline or Grade 1. | Dose MUST be reduced by 1 dose level. |
| ILD/pneumonitis <sup>5</sup> | Grade 2 that persists or recurs despite maximal supportive measures and does not return to baseline or Grade 1 within 7 days | Suspend dose until toxicity resolves to baseline or ≤Grade 1. | Dose MUST be reduced by 1 dose level. |
| ILD/pneumonitis | Grade 3 and 4 | Dose MUST be discontinued | NA |
| Nonhematologic Toxicity | Grade 3 or 4 | Dose MUST be<br>suspended until toxicity<br>resolves to either<br>baseline or Grade 1. | Dose MUST be reduced by 1 dose level. |
| Diarrhoea | Grade 2 that does not resolve within 24 hours to at least Grade 1 | Dose MUST be<br>suspended until toxicity<br>resolves to at least<br>Grade 1. | Dose MAY be reduced by 1 dose level - investigator's discretion. |

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 4.1.4.2: 2 (cont.) Dose Adjustments and Delays for Toxicity Possibly Related to Abemaciclib\*

| <b>Toxicity Type</b> | <b>Toxicity Profile and Severity</b> | <b>Dose Suspension</b> | Dose Reduction |
|---|---|---|---|
| Diarrhoea | Requires hospitalization or Grade 3 or 4 | Dose MUST be<br>suspended until toxicity<br>resolves to at least<br>Grade 1. | Dose <b>MUST</b> be reduced by 1 dose level. |
| Diarrhoea | Grade 2 that persists or recurs<br>after resuming the same dose<br>despite maximal supportive<br>measures | Dose MUST be<br>suspended until toxicity<br>resolves to at least<br>Grade 1. | Dose MUST be reduced by 1 dose level. |
| Increased ALT | Persistent or Recurrent <sup>3</sup> Grade 2 (>3.0-5.0xULN), or Grade 3 (>5.0-20.0xULN) <sup>4</sup> | Dose MUST be<br>suspended until toxicity<br>resolves to either<br>baseline or Grade 1. | Dose MUST be reduced by 1 dose level. |
| Increased ALT with increased total bilirubin, in the absence of cholestasis | Grade 3 (>5.0xULN) with total bilirubin>2xULN | Abemaciclib MUST be discontinued | NA |
| Increased ALT | Grade 4 (>20.0xULN) | Abemaciclib MUST be discontinued | NA |

<sup>\*</sup>In case that the Toxicity Profile and Severity qualifies for DLT according to Section 5.3.7, dose suspension and dose reduction will be followed according to the DLT management instructions

- shows stable hematological counts (Grade ≤2) during that timeframe
- has absence of any signs or risk of infection
- is benefiting from study treatment

Abbreviation: ASCO = American Society of Clinical Oncology.

Note: MAY = per the investigator's clinical judgment; MUST = mandatory.

#### 4.1.5 Blinding and procedures for unblinding

## 4.1.5.1 Blinding

In this open-label trial, treatment allocation will not be concealed throughout the trial. The trial will be handled in an open fashion by the Sponsor during the conduct, data cleaning and preparation for analysis.

<sup>&</sup>lt;sup>1</sup> Recurrent toxicity refers to the same event occurring within the next 8 weeks (as measured from the stop date of the preceding event). As a general guidance, based on the risk/benefit balance assessment per the investigator, for a patient who experiences a new episode of Grade 3 hematological toxicity after more than 8 weeks following the last episode of same Grade 3 hematological toxicity, the investigator may consider resuming the patient on the same drug dose should the patient satisfy the following conditions:

<sup>&</sup>lt;sup>2</sup> Additional guidance for renal monitoring is in <u>Section 4.4.1</u>

<sup>&</sup>lt;sup>3</sup> Determination of persistent events will be at the discretion of the investigator. Recurrent toxicity refers to the same event occurring within the next 8 weeks (as measured from the stop date of the preceding event).

<sup>&</sup>lt;sup>4</sup> Grade 3 ALT increased is a trigger for additional assessments and possibly hepatic monitoring. See Section 4.4.4 for additional guidance for hepatic monitoring

<sup>&</sup>lt;sup>5</sup> For Japan only: refer to local amendment in Japan for ILD guidance

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 4.1.5.2 Unblinding and breaking the code

Not applicable.

# 4.1.6 Packaging, labelling, and re-supply

The investigational products will be provided by BI or a designated CRO. They will be packaged and labelled in accordance with the principles of Good Manufacturing Practice (GMP). Re-supply to the sites will be managed via an IRT system, which will also monitor expiry dates of supplies available at the sites.

For details of packaging and the description of the label, refer to the ISF.

# 4.1.7 Storage conditions

Drug supplies will be kept in their original packaging and in a secure limited access storage area according to the recommended storage conditions on the medication label for anastrozole, letrozole and fulvestrant. For recommended storage conditions regarding abemaciclib and xentuzumab, please refer to the medication label. A temperature log must be maintained for documentation.

**Abemaciclib** will be supplied as capsules or tablets for oral administration. The capsules and tablets should be stored at room temperature according to the range provided on the product label and not opened, crushed, or dissolved. Investigators should instruct patients to store the capsules and tablets in the original package and in a location inaccessible to children. Clinical study materials will be labelled according to country regulatory requirements.

**Xentuzumab** is supplied as a liquid formulation at a concentration of 10 mg/mL in 20 mL single use vials, which contain 200 mg of xentuzumab per vial. All vials containing xentuzumab must be kept refrigerated according to the temperature range provided on the product label prior to dosage preparation.

The vials should not be frozen or shaken and should be kept in the outer carton in order to protect from light. They should not be used beyond the expiration date.

If the storage conditions are found to be outside the specified range, the local clinical monitor (as provided in the list of contacts) must be contacted immediately and product quarantined.

# 4.1.8 Drug accountability

The Investigator and/or Pharmacist and/or investigational drug storage manager will receive the investigational drugs delivered by the sponsor when the following requirements are fulfilled:

- \* Approval of the trial protocol by the IRB / ethics committee and HA approval,
- \* Availability of a signed and dated clinical trial contract between the sponsor and the head of the investigational site,
c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Approval/notification of the regulatory authority, e.g. competent authority,
- \* Availability of the curriculum vitae of the principal Investigator,
- Availability of a signed and dated clinical trial protocol,
- Availability of the proof of a medical license for the principal Investigator,
- \* Availability of Form 1572 (USA specific requirement)

The Investigator and/or Pharmacist and/or investigational drug storage manager must maintain records of the product's delivery to the trial site, the inventory at the site, the use by each patient, and the return to the sponsor or warehouse / drug distribution centre or alternative disposal of unused products. If applicable, the sponsor or warehouse / drug distribution centre will maintain records of the disposal.

These records will include dates, quantities, batch / serial numbers, expiry ('use- by') dates, and the unique code numbers assigned to the investigational product and trial patients. The Investigator / Pharmacist / investigational drug storage manager will maintain records that document adequately that the patients were provided the doses specified by the CTP and reconcile all investigational products received from the sponsor. At the time of return to the sponsor and/or appointed CRO, the Investigator / Pharmacist / investigational drug storage manager must verify that all unused or partially used drug supplies have been returned by the clinical trial patient and that no remaining supplies are in the Investigator's possession.

## 4.2 OTHER TREATMENTS, EMERGENCY PROCEDURES, RESTRICTIONS

## 4.2.1 Other treatments and emergency procedures

There are no special emergency procedures to be followed.

Symptomatic treatments of tumour-associated symptoms are allowed. Concomitant medications or therapy to provide adequate supportive care may be given as clinically necessary.

After study enrolment, palliative radiotherapy may be given for analgesic purposes, lytic lesions at risk of fracture or for other reasons (e.g. bronchial obstruction, skin lesions), provided that the total dose delivered is in a palliative range to non-target lesion according to institutional standards. Information on palliative radiotherapy will be captured in eCRF. It is at the investigator's discretion to withhold the study treatment during palliative radiotherapy. The investigators should assess the signs/symptoms carefully to exclude the progressive disease prior to the administration of the palliative radiotherapy.

The acute use of bisphosphonates and denosumab for symptomatic treatment of bone metastases is permitted during the study, but chronic use for the prevention of bone metastases is prohibited. Bisphosphonate therapy for the treatment of osteoporosis, at the doses indicated under prescribing information, is permitted during the study. If bisphosphonate therapy is initiated after enrolment, the reason for its use must be clearly documented in the eCRF.


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

All medications (other than study drug), including anaesthetic agents, vitamins, homeopathic/herbal remedies, nutritional supplements, and significant non-drug therapies (including physical therapy and blood transfusions) starting or changing after the patient signed informed consent must be listed on the concomitant medication page of eCRF including trade name, start and end dates, indication for use etc. as specified in the Flow Chart.

If patients receive parenteral nutrition during the trial, the components need not be specified in detail. It should just be indicated as "parenteral nutrition". If a patient requires anaesthesia, it will be sufficient to indicate "anaesthesia" without specifying details.

In case of major surgery (as judged by the investigator), it is recommended to stop treatment with xentuzumab and/or abemaciclib around one week prior to the surgery, and to restart treatment after complete wound healing. If the patient can't recover within 28 days since stopping study medication, patient should be removed from the study. Exception to this in patients who derive obvious clinical benefit according to the investigator's judgement could be agreed upon discussion with the Sponsor's Clinical Monitor.

#### 4.2.2 Restrictions

## 4.2.2.1 Restrictions regarding concomitant treatment

With the exceptions listed in the sections below, no other chemotherapy, experimental medications, other anticancer therapy, including but not limited to immunotherapy, hormonal cancer therapy, radiation, experimental medications, or surgery for cancer will be permitted while patients are on study treatment. Use of megestrol acetate as an appetite stimulant is not permitted.

Abemaciclib is extensively metabolized through oxidation by CYP3A. In clinical drug interaction studies, coadministration of clarithromycin, a strong CYP3A inhibitor, increased exposure (AUC) to abemaciclib by 3.4 fold (Study JPBE) and coadministration of rifampin, a strong CYP3A inducer, decreased exposure to abemaciclib by 95% (Study JPBF). Therefore, grapefruit juice should be avoided and inducers and strong inhibitors of CYP3A should be substituted or avoided whenever possible (See Appendix 10.1).

During PK assessments of abemaciclib, the concomitant use of inhibitors or inducers of CYP3A4 should be avoided whenever possible, i.e. during Run-In, course 1 and course 2 of cohort E and during course 1 and 2 of expansion cohorts D1, D2 and F.

Apart from those assessments, patients are recommended to avoid concomitant use of strong CYP3A inhibitors and use caution with coadministered moderate or weak CYP3A inhibitors. Patients who continue to take strong CYP3A inhibitors should reduce the abemaciclib dose. In patients who are taking the starting dose of 150 mg twice daily, reduce the abemaciclib dose to 100 mg twice daily or, specifically in the case of ketoconazole, the abemaciclib dose should be reduced to 50 mg twice daily. In patients who have had a dose reduction to 100 mg twice daily due to adverse reactions, further reduce the abemaciclib dose to 50 mg twice daily. If a patient taking abemaciclib discontinues a strong CYP3A inhibitor, increase the abemaciclib


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

dose (after 3-5 half-lives of the inhibitor) to the dose that was used before starting the strong inhibitor. Please refer to current SmPC of Verzenio (abemaciclib).

In case it is unavoidable to treat a patient with a comedication that is a moderate to potent inducer or inhibitor of CYP3A4 dose adaptation of abemaciclib should be done as described above and according to the SmPC of Verzenio (abemaciclib). Furthermore, the patient should be closely monitored and precautions should be taken as described in the SmPC of Verzenio (abemaciclib).

Abemaciclib can be coadministered with drugs which are substrates of CYP enzymes.

Abemaciclib and/or its major metabolites inhibit the efflux transporters P-glycoprotein and breast cancer resistance protein and renal transporters organic cation transporter 2, multidrug and toxin extrusion protein 1 (MATE1), and MATE2-K at clinically relevant concentrations. Therefore, substrates of these transporters such as metformin and those with a narrow therapeutic index such as digoxin, dofetilide, or dabigatran should be substituted or avoided if possible.

Restrictions regarding concomitant treatment with fulvestrant, letrozole or anastrozole: please refer to the most up to date labelling information of each product, as appropriate (i.e. depending on the treatment cohort).

## 4.2.2.2 Restrictions on diet and life style

Patients have to show up in fasting condition at the site when blood draw for safety lab is required.

Grapefruit and/or Seville orange juices must be avoided during treatment with abemaciclib.

## 4.2.2.3 Restrictions regarding men and women of childbearing potential

Women of childbearing potential must use the contraception methods described in the patient information per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information, and must be used from the screening period until 3 weeks following the last dose of abemaciclib and at least 6 months after the last dose of xentuzumab.

Men should not father a child during treatment with xentuzumab and for at least 70 days after the last dose of xentuzumab.

## 4.2.2.4 Supportive Care

Patients should receive full supportive care to maximize quality of life. Patients will receive supportive care based on the judgment of the treating physician. If it is unclear whether a therapy should be regarded as supportive care, the investigator should consult the BI clinical monitor.


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Use of any supportive care therapy should be reported on the electronic case report form (eCRF).

## 4.2.2.5 Growth Factor Therapy

Growth factors may be administered in accordance with American Society of Clinical Oncology guidelines (Smith et al. 2006; Rizzo et al. 2008).

## 4.2.2.6 Therapy for Diarrhoea

At enrolment, patients should receive instructions on the management of diarrhoea. In the event of diarrhoea, supportive measures should be initiated <u>as early as possible</u>. These include the following:

- \* At the first sign of loose stools, the patient should initiate anti-diarrheal therapy, if not already receiving such therapy (for example, loperamide), and notify the investigator/site for further instructions and appropriate follow-up.
- \* Patients should also be encouraged to drink fluids (for example, 8 to 10 glasses of clear liquids per day).
- \* Site personnel should assess response within 24 hours.
- \* If diarrhoea does not resolve with anti-diarrheal therapy within 24 hours to either baseline or Grade 1, study drug should be suspended until diarrhoea is resolved to baseline or Grade 1.
- \* When study drug recommences, dosing should be adjusted, refer to the dose adjustment guidelines in <u>Section 4.1.4.2</u>.

In cases of significant diarrhoea, Grade 2 through 4 which has not responded to interventions as outlined above, if the investigators are considering the addition of steroids to treat potential colitis, the sponsor strongly recommends an endoscopic procedure to document colitis prior to initiating steroids.

In severe cases of diarrhoea, the measuring of neutrophil counts and body temperature and proactive management of diarrhoea with antidiarrheal agents should be considered.

If diarrhoea is severe (requiring IV rehydration) and/or associated with fever or severe neutropenia, broad-spectrum antibiotics such as fluoroquinolones must be prescribed.

Patients with severe diarrhoea or any grade of diarrhoea associated with severe nausea or vomiting should be carefully monitored and given intravenous fluid (IV hydration) and electrolyte replacement.

## 4.2.2.7 Ovarian suppression with gonadotropin-releasing hormone agonists

Patients who are postmenopausal due to ovarian suppression should continue GnRH agonist therapy during study treatment.


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4.3 TREATMENT COMPLIANCE

The study medications will be given in accordance with the protocol and the instructions of a site investigator. The investigator should instruct the patient to take the study drugs exactly as prescribed to promote compliance.

A patient will be considered noncompliant if he or she is judged by the investigator to have intentionally or repeatedly taken more than 125% the prescribed amount of abemaciclib or less than 75%. Abemaciclib dose suspensions or delays related to toxicity may occur and will not result in a patient being considered as noncompliant. Same rules apply to background hormonal therapy.

Patients are requested to bring all remaining trial medication including empty package material with them when attending visits.

Based on counts, treatment compliance will be calculated as the number of doses taken, divided by the number of doses which should have been taken according to the scheduled period, multiplied by 100. Compliance will be verified by the on-site monitor authorised by the sponsor.

Treatment compliance (%) =  $\frac{\text{Number of doses actually taken} \times 100}{\text{Number of doses which should have been taken}}$ 

If the number of doses taken is not between 75-125%, site staff will explain the patient the importance of treatment compliance.

The investigator and/or the sponsor can withdraw a patient from the study in the event of serious and persistent non-compliance which jeopardizes the patient's safety or render study results.

Xentuzumab will be administered as a single infusion under supervision of the investigator or dedicated study personnel. In the event that the full dose of xentuzumab is not administered to the patient, it must be documented and explained.

A maximum of three consecutive xentuzumab infusions may be skipped for the recovery from AEs. Missing xentuzumab treatment for any other reasons is considered non-compliant.

#### Patient diary for cohort E

For the purpose of PK characterisation of abemaciclib, patients of cohort E will be dispensed a patient diary two times during the conduct of the study: at run-in visit 1 and again at Cycle 1 visit 4. These patient diaries will collect information about daily intake of abemaciclib and potential vomiting events. The first patient diary will collect information during the 3 days prior to Run-In Visit 3. The second patient diary will collect information of the 3 days before Cycle 2 Visit 1. Site staff will be required to transfer the data from the patient diary into the corresponding eCRF fields.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 4.4 MANAGEMENT OF EXPECTED ADVERSE EVENTS.

#### 4.4.1 Increased Serum Creatinine

Abemaciclib has been shown to increase serum creatinine due to inhibition of renal tubular secretion of creatinine without affecting glomerular filtration rate (GFR [as measured by ioxhexol clearance]). In clinical studies, increases in serum creatinine occurred within the first month of abemaciclib dosing (remainder elevated but stable through the treatment period), were reversible upon treatment discontinuation, and were not accompanied by changes in markers of renal function such as blood urea nitrogen, cystatin C, or calculated GFR based on cystatin C.

Dose adjustment (omission, reduction, or discontinuation) should not solely be based on interpretation of serum creatinine values because these may not reflect renal function. If deterioration of renal function is suspected per the investigator's clinical assessment, dose alteration should follow the protocol guidance for non-hematological toxicities (Section 4.1.4.2).

## 4.4.2 Management and grading of infusion reactions

The xentuzumab infusion should always be administered under close supervision of a medically qualified staff member with immediate availability of appropriate resuscitation facilities.

Infusion reactions may occur during infusion with xentuzumab and include pyrexia, chills, rigors, dyspnoea, urticaria, bronchospasm, hypotension and hypertension. **A one hour observation period is recommended following each infusion.** If there is no infusion reaction during the first treatment course, the observation period following xentuzumab infusion may be adjusted at the discretion of the investigators. Mild to moderate infusion reactions may be managed with a slower infusion rate and prophylactic antihistamines for subsequent dosing. Severe reactions require immediate and permanent discontinuation of infusion. The hypersensitivity reactions will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 (R10-4848).

The infusion duration may be extended to over one hour and up to a maximum of three hours.

The infusion reactions should be treated symptomatically as judged clinically relevant by the investigator. For symptomatic treatment of infusion reactions: hydrocortisone, antihistamines such as chlorphenamine accompanied by an antipyretic/analgesic and/or a bronchodilator is recommended.

Infusion reactions will not be reported on the standard AE page but will be reported on a separate page specifically for infusion reactions in the CRF.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 4.4.2: 1 Infusion reaction management

| <b>Infusion Reaction Grade</b> | Management |
|---|---|
| CTCAE Grade 1 or 2 | In the event of a CTCAE grade 1 infusion reaction, the infusion |
| | rate should be reduced by 50%. |
| | A Grade 2 infusion reaction may require symptomatic |
| | treatment, as described above (with infusion interruption). |
| | Once the event has resolved, the infusion may be restarted at |
| | the reduced rate. |
| CTCAE Grade 3 | For patients experiencing a CTCAE grade 3 infusion reaction, |
| | infusion should be interrupted immediately and patients should |
| | receive aggressive symptomatic treatment, as described above. |
| | Only after all the symptoms have disappeared, the infusion may |
| | be re-started if it is within 3 hours since the infusion start. The |
| | infusion rate should be reduced by half after re-start |
| CTCAE Grade 4 | Patients experiencing CTCAE grade 4 such as anaphylaxis |
| | during an infusion should have infusion immediately stopped |
| | and receive appropriate treatment, as described above, |
| | including use of resuscitation medications If needed. Such |
| | patients should NOT receive any further xentuzumab treatment. |

## 4.4.3 Management of Neutropenia

Adverse events of neutropenia have been observed in studies with xentuzumab and causality has been established with abemaciclib. Patients should be monitored closely for signs of infection. Dose adjustment for severe neutropenia (≥ Grade 3) should follow as per <u>Table 4.1.4.2: 1</u> (xentuzumab) and <u>Table 4.1.4.2: 2</u> (abemaciclib) in the protocol. Fever or infection in the presence of severe neutropenia should be managed promptly with broad-spectrum antibacterial therapy.

#### 4.4.4 Management of Hepatotoxicity

Grade  $\geq 3$  increased ALT was reported in patients receiving abemaciclib in breast cancer studies. Monitor ALT, prior to the start of abemaciclib therapy, every 2 weeks for the first 2 months, monthly for the next 2 months, and as clinically indicated. Please refer to Flow Chart for time points. Based on the level of ALT elevations, abemaciclib may require dose modification. (see Table 4.1.4.2:2).

In addition, for hepatic toxicity, additional monitoring should be considered. Details for hepatic monitoring depend upon the severity and persistence of observed laboratory test abnormalities. If the abnormality persists or worsens, clinical and laboratory monitoring should be initiated by the investigator, based on the hepatic monitoring tests (see Section 10.5) and in consultation with the Sponsor. Monitoring of ALT, AST, and total bilirubin should continue until levels normalize or return to approximate baseline levels. Additional diagnostic testing should be considered to rule out cause of increased liver enzymes per the investigator's discretion.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4.4.5 Venous Thromboembolism

Venous thromboembolic events were reported in patients receiving abemaciclib plus fulvestrant or aromatase inhibitors in breast cancer studies. The majority of the events were non-serious and were treated with low-molecular-weight heparin. Generally, these events did not result in discontinuation of the study treatment. At this time, the mechanism underlying the association between abemaciclib and the occurrence of VTEs is not known. Monitor patients for signs and symptoms of deep vein thrombosis and pulmonary embolism and treat as medically appropriate.

## 4.4.6 Guidance for Interstitial lung disease/Pneumonitis

ILD/pneumonitis has been identified as an adverse drug reaction for abemaciclib. Additional information is available in the IB of abemaciclib.

Ask your patients to report any new or worsening respiratory symptoms such as cough, dyspnea, fever, and investigate and treat as per your local clinical practice (including corticosteroids as appropriate). If ILD/pneumonitis is suspected, investigations may include imaging such as high resolution computed tomography (HRCT), broncheoalveolar lavage, and biopsy as clinically indicated. Refer to <u>Table 4.1.4.2:2</u> for guidance on dose adjustments of abemaciclib for patients with ILD/pneumonitis. Discontinue abemaciclib in cases of severe ILD/pneumonitis.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 5. VARIABLES AND THEIR ASSESSMENT

#### 5.1 TRIAL ENDPOINTS

## 5.1.1 Primary Endpoint(s)

### For dose finding cohorts A, B, C, and D (dose finding):

The primary endpoints for each dose finding cohort are the MTD and the number of patients with dose limiting toxicities (DLT) in the MTD evaluation period.

The MTD evaluation period is defined as the first treatment cycle (28 days). The MTD is defined as the highest dose with less than 25% risk of the true DLT rate being above 33%. For definition of DLTs, refer to Section 5.3.7

A Bayesian Logistic Regression Model (BLRM) employing the escalation with overdose control (EWOC) principle will be used during each dose finding cohort for a selection of doses to investigate and for estimation of the MTD. Cohorts of patients will receive xentuzumab and abemaciclib (with or without endocrine therapy) until the MTD is reached or until the Steering Committee (SC) decides on stopping the dose finding. Each dose-level cohort will consist of newly enrolled patients. Estimation of the MTD during each dose finding cohort of the study will be based upon the estimation of the probability of a DLT in the MTD evaluation period in the set of evaluable patients for MTD. The corresponding methodology is described in Section 7.

The MTD estimate established during the dose finding cohort will be re-investigated after the corresponding expansion cohort by re-running the BLRM including all data from dose finding cohort and expansion cohort, in particular also considering the DLT information from all treatment cycles.

#### For expansion cohort E

The primary endpoint for expansion part is objective response (OR) defined as best overall response of complete response (CR) or partial response (PR), where best overall response is determined according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1 from date of first treatment administration (including run-in for cohort E) until the earliest of disease progression, death or last evaluable tumour assessment before start of subsequent anticancer therapy.

## For expansion cohorts D1 and D2:

The primary endpoint for expansion part is PFS rate at 18 month defined as the rate of absence of disease progression or death at 18<sup>th</sup> month, where progression is determined according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1.

## For expansion cohort F

The primary endpoint for expansion part is disease control (DC) defined as best overall response of complete response (CR) or partial response (PR) or confirmed stable disease (SD) (lasting for at least 24 weeks) or Non-CR/ Non-PD (lasting for at least 24 weeks) where best

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

overall response is defined according to RECIST version 1.1 from first treatment administration until the earliest of disease progression, death or last evaluable tumour assessment before start of subsequent anti-cancer therapy.

## 5.1.2 Secondary Endpoint(s)

### For dose finding cohorts A, B, C, and D (dose finding)

There are no secondary endpoints.

#### For expansion cohorts E, F, D1 and D2:

The secondary endpoints are:

- \* Cohorts D1, D2 and E only: Disease control (DC) defined as best overall response of complete response (CR) or partial response (PR) or confirmed stable disease (SD) (. lasting for at least 24 weeks) where best overall response is defined according to RECIST version 1.1 from first treatment administration until the earliest of disease progression, death or last evaluable tumour assessment before start of subsequent anticancer therapy.
- \* Time to objective response defined as the time from first treatment administration until first documented complete response (CR) or partial response (PR).
- \* Duration of objective response defined as the time from first documented complete response (CR) or partial response (PR) until the earliest of disease progression or death among patients with objective response.
- \* Duration of disease control defined as the time from first treatment administration until the earliest of disease progression or death, among patients with disease control.
- \* Progression-free survival (PFS) defined as the time from first treatment administration until tumour progression according to RECIST 1.1 or death from any cause, whichever occurs earlier.
- \* Cohorts D1, D2 and F only: Objective response (OR) defined as best overall response of complete response (CR) or partial response (PR), where best overall response is determined according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1 from date of first treatment administration until the earliest of disease progression, death or last evaluable tumour assessment before start of subsequent anticancer therapy.

09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

09049566-10 Trial Protocol 
Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies c09049566-10


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



#### 5.2 ASSESSMENT OF EFFICACY

Response Evaluation Criteria in Solid Tumours (RECIST) guideline (version 1.1) (<u>R09-0262</u>) will be applied as the primary measure for assessment of tumour response, date of disease progression, and as a basis for all protocol guidelines related to disease status (e.g. discontinuation of study therapy). See <u>Appendix 10.4</u> for details on lesion measurements and response assessment according to RECIST 1.1.

Tumour response will be assessed by Investigator review throughout the study and clinical decisions will be based on Investigator assessment.

Imaging will be performed as indicated in the Flow Chart and in Appendix 10.4.

Tumour assessment will be assessed per institutional practice. Only the overall response will be collected in the eCRF.

#### 5.3 ASSESSMENT OF SAFETY

### **5.3.1** Physical examination

A physical examination will be performed at the time points specified in the <u>Flow Chart</u>. A full physical exam must include cardiopulmonary examination, examination of the regional lymph nodes, and examination of the abdomen and an assessment of the mental and neurological status. Additional symptoms which have not been reported during a previous examination must be clarified. Wherever possible the same investigator should perform this examination.

When xentuzumab is discontinued, physical examination assessments can be done as per institutional practice.

#### 5.3.2 Vital Signs

Vital sign measurements (blood pressure [systolic blood pressure, diastolic blood pressure], pulse rate, respiratory rate, temperature and measurement of height (at screening) and body weight and the evaluation of the ECOG performance status will be performed at the times specified in the <u>Flow Chart</u> and Schedule of Procedures/Assessments (<u>Section 6.2</u>). Blood pressure and pulse will be measured after the patient has been recumbent or seated for 5 minutes.

When xentuzumab is discontinued, vital signs assessments can be done as per institutional practice.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 5.3.3 Safety laboratory parameters

Blood samples, including fasting serum samples (fasting state for at least 8 hours) and the fasting lipid profile, can be collected up to one day prior to the scheduled time points as specified in the <u>Flow Chart</u> and analysed in a laboratory facility at (or close to) the investigational site. Safety laboratory examinations include haematology, coagulation, biochemistry and urine examination. See <u>Table 5.3.3: 1</u> for details. In case of abnormal findings such as neutropenia or thrombocytopenia, further test may be done if clinically indicated at the discretion of the investigator. All analyses are to be performed by the local clinical laboratory. Unscheduled safety laboratory examinations will be documented in the eCRF along with the results.

Safety laboratory assessment may be performed according to local practice but must include at least all of the following parameters:

Table 5.3.3: 1 Clinical laboratory tests

| Category | Parameters |
|---|---|
| Haematology | Red blood cell count (RBC), haemoglobin, haematocrit, platelet count, white blood cell count (WBC) with differential (neutrophils <sup>1</sup> , lymphocytes, monocytes, eosinophils, basophils) |
| Coagulation | International Normalized Ratio (INR), activated Partia Thromboplastin Time (aPTT) |
| Chemistry | Blood urea or blood urea nitrogen (BUN), creatinine, cystatin-C (day 1 of every cycle), alkaline phosphatase (AP), aspartate aminotransferase (AST), alanine aminotransferase (ALT), γ-glutamyltransferase (GGT), bilirubin (total and direct), total protein, albumin, creatine phosphokinase (CPK); in case of pathological CPK further evaluation (e.g. by determination of isoenzymes, troponin assays, ECG exam) should be performed as clinically indicated |
| Pregnancy TEST | Serum (for women of childbearing potential only) |
| Electrolytes | Sodium, potassium, calcium, magnesium |
| Lipid profile (fasting) | Total cholesterol, triglycerides, LDL, HDL |
| Other (fasting) | Glucose, HbA1C and C-peptide |
| Urinalysis (only at screening and EOTV) | pH, protein, glucose, erythrocytes, leucocytes, ketones and nitrite will be analysed by dipstick (semi-quantitative measurements: -, +, ++, +++); in case of pathological finding further evaluation should be performed and results documented |

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 5.3.3: 1 Clinical laboratory tests (cont.)

| Category | Parameters |
|---|---|
| Post-menopausal status (at screening | FSH, estradiol |
| only for women <60 years old without prior bilateral oophorectomy) | |

Neutrophils reported by automated differential hematology instruments include both segmented and band forms. When a manual differential is needed to report the neutrophils, the segmented and band forms should be reported together

## When xentuzumab is discontinued, safety labs can be done as per institutional practice.

#### 5.3.4 Electrocardiogram

As per ICH E 14 large targeted proteins and monoclonal antibodies have a low likelihood of direct ion channel interactions and a thorough QT/QTc study is not necessary, unless the potential for proarrhythmic risk is suggested by mechanistic considerations or data from clinical or non-clinical studies, which is not the case for xentuzumab.

Therefore, only local reading of ECG will be conducted in this trial. 12-Lead resting electrocardiograms (ECG) are recorded locally and in triplicate. ECG will be performed at Screening, at Run in visit 2 Day -2 (in cohorts E and F), at EOTV and FUV. ECG will be repeated at Visit 1/Day 1, and Visit 3/Day 15 of Courses 1, 2, 3; and at Visit 1/Day 1 of Courses 6, 9, 12, etc. ECG should be performed prior to xentuzumab infusion.

#### When xentuzumab is discontinued, ECGs can be omitted.

#### 5.3.5 Other safety parameters

Not applicable.

#### **5.3.6** Assessment of adverse events

Safety assessments will consist of monitoring and recording all adverse events (AEs) and serious adverse events (SAEs) and includes periodic physical examinations, measurement of vital signs, assessment of performance status, monitoring of laboratory tests (i.e. haematology, chemistry, coagulation, urine, etc.)

#### 5.3.6.1 Definitions of AEs

## **Adverse** event

An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment.


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

#### **Adverse reaction**

An adverse reaction is defined as a response to a medicinal product which is noxious and unintended. Response in this context means that a causal relationship between a medicinal product and an adverse event is at least a reasonable possibility. Adverse reactions may arise from use of the product within or outside the terms of the marketing authorisation or from occupational exposure. Conditions of use outside the marketing authorization include off-label use, overdose, misuse, abuse and medication errors.

## Serious adverse event

A serious adverse event (SAE) is defined as any AE which:

- results in death,
- is life-threatening, this refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if more severe.
- requires inpatient hospitalisation or
- prolongation of existing hospitalisation,
- results in persistent or significant disability or incapacity, or
- is a congenital anomaly / birth defect, or
- is to be deemed serious for any other reason if it is an important medical event when based upon appropriate medical judgment which may jeopardise the patient and may require medical or surgical intervention to prevent one of the other outcomes listed in the above definitions.

The following hospitalizations are not considered to be serious adverse events (SAEs) because there is no "adverse event" (i.e., there is no untoward medical occurrence) associated with the hospitalization:

- Hospitalizations for respite care
- Hospitalization planned prior to informed consent (where the condition requiring the hospitalization has not changed post study drug administration)
- Hospitalization for administration of study drug or PK assessment

Medical and scientific judgement should be exercised in deciding whether other situations should be considered serious reactions, such as important medical events that might not be immediately life threatening or result in death or hospitalisation but might jeopardise the patient or might require intervention to prevent one of the other outcomes listed above. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalisation or development of dependency or abuse. Any suspected transmission via a medicinal product of an infectious agent is also considered a serious adverse reaction.

5-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

For Japan only: the following events will be handled as "deemed serious for any other reason". An AE which possibly leads to disability will be reported as an SAE.

#### AEs considered "Always Serious"

Every new occurrence of cancer of new histology must be reported as a serious event regardless of the duration between discontinuation of the drug and the occurrence of the cancer. In accordance with the European Medicines Agency initiative on Important Medical Events, Boehringer Ingelheim has set up a list of further AEs, which by their nature, can always be considered to be "serious" even though they may not have met the criteria of an SAE as given above.

The latest list of "Always Serious AEs" can be found in the EDC system.

These events should always be reported as SAEs as described above.

#### Adverse events of special interest (AESI)

The term AESI relates to any specific AE that has been identified at the project level as being of particular concern for prospective safety monitoring and safety assessment within this trial, e.g. the potential for AEs based on knowledge from other compounds in the same class. AESI need to be reported to the sponsor's Pharmacovigilance Department within the same timeframe that applies to SAE, please see above.

The following are considered as AESIs:

**Hepatic injury** is defined by the following alterations of hepatic laboratory parameters: For patients with normal liver function (ALT, AST, and bilirubin within normal limits) at baseline, an elevation of AST and/or ALT  $\geq 3$  fold ULN combined with an elevation of total bilirubin  $\geq 2$  fold ULN measured in the same blood draw sample, and/or marked peak aminotransferase (ALT, and/or AST) elevations  $\geq 10$  fold ULN.

For patients with abnormal liver function tests at baseline (AST and/or ALT > ULN), an elevation of transaminase  $\geq$  (baseline + 4x ULN) combined with an elevation of total bilirubin  $\geq$  2 fold ULN measured in the same blood draw sample, with the exclusion of the causes due to underlying diseases. Patients with abnormal liver function tests must have their abnormalities and the etiology documented **in detail as baseline conditions**. Every effort should be made to explain possible deteriorations of baseline conditions.

These lab findings constitute a hepatic injury alert and the patients showing these lab abnormalities need to be followed up according to the "DILI checklist" provided in the ISF. In case of clinical symptoms of hepatic injury (icterus, unexplained encephalopathy, unexplained coagulopathy, right upper quadrant abdominal pain, etc.) without lab results (ALT, AST, total bilirubin) available, the investigator should make sure these parameters are analysed, if necessary in an unscheduled blood test. Should the results meet the criteria of hepatic injury alert, the procedures described in the DILI checklist should be followed.

**DLT** occurs in the dose finding cohorts. Please refer to Section 5.3.7 for definition of DLTs.


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Cases of **pneumonitis** (including interstitial lung disease, non-infectious pneumonitis and other analogous terms) occurring at any cycle in both phases.

#### **Intensity of AEs**

The intensity of adverse events should be classified and recorded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 in the eCRF.

## Causal relationship of AEs

The definition of an adverse reaction implies at least a reasonable possibility of a causal relationship between a suspected medicinal product and an adverse event. An adverse reaction, in contrast to an adverse event, is characterised by the fact that a causal relationship between a medicinal product and an occurrence is suspected.

Medical judgment should be used to determine the relationship, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history.

Arguments that may suggest that there is a reasonable possibility of a causal relationship could be:

- The event is consistent with the known pharmacology of the drug.
- The event is known to be caused by or attributed to the drug class.
- A plausible time to onset of the event relative to the time of drug exposure.
- Evidence that the event is reproducible when the drug is re-introduced.
- No medically sound alternative aetiologies that could explain the event (e.g. preexisting or concomitant diseases, or co-medications).
- The event is typically drug-related and infrequent in the general population not exposed to drugs (e.g. Stevens-Johnson syndrome).
- An indication of dose-response (i.e. greater effect size if the dose is increased, smaller effect size if dose is diminished).

Arguments that may suggest that there is no reasonable possibility of a causal relationship could be:

- No plausible time to onset of the event relative to the time of drug exposure is evident (e.g. pre-treatment cases, diagnosis of cancer or chronic disease within days / weeks of drug administration; an allergic reaction weeks after discontinuation of the drug concerned).
- Continuation of the event despite the withdrawal of the medication, taking into account
  the pharmacological properties of the compound (e.g. after 5 half-lives).
   Of note, this criterion may not be applicable to events whose time course is prolonged
  despite removing the original trigger.
- Additional arguments amongst those stated before, like alternative explanation (e.g. situations where other drugs or underlying diseases appear to provide a more likely explanation for the observed event than the drug concerned).
- Disappearance of the event even though the study drug treatment continues or remains unchanged.


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 5.3.6.2 Adverse event collection and reporting

#### **AE Collection**

The Investigator shall maintain and keep detailed records of all AEs in their patient files. The following must be collected and documented on the appropriate eCRF(s) by the Investigator:

- From signing the informed consent onwards until the end of treatment (including the Residual Effect Period, REP):
  - All AEs (non-serious and serious) and all AESIs.
- After the end of treatment (including the REP) until the individual patient's end of trial:
  - All related SAEs and all related AESIs.
- After the individual patient's end of the trial:

The Investigator does not need to actively monitor the patient for AEs but should only report relevant SAEs and relevant AESIs of which the Investigator may become aware of. The rules for Adverse Event Reporting exemptions still apply.



Figure 5.3.6.2: 1 AE collection periods

The REP is defined as 42 days after the last trial medication application. All AEs which occurred through the treatment phase (which includes the run-in period) and throughout the REP will be considered as on treatment; please see Section 7.3.4. Events which occurred after the REP will be considered as post treatment events.

#### AE reporting to sponsor and timelines

The Investigator must report SAEs, AESIs, and non-serious AEs which are relevant for the reported SAE or AESI, on the BI SAE form via fax immediately (within 24 hours ) to the sponsor's unique entry point (country specific contact details will be provided in the ISF).

The same timeline applies if follow-up information becomes available. In specific occasions the Investigator could inform the sponsor upfront via telephone. This does not replace the requirement to complete and fax the BI SAE form.

For Japan only: all SAEs must be reported immediately to the head of the trial site.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

With receipt of any further information to these events, a follow-up SAE form has to be provided. For follow-up information the same rules and timeline apply as for initial information.

#### **Information required**

For each AE, the Investigator should provide the information requested on the appropriate CRF pages and the BI SAE form. The Investigator should determine the causal relationship to the trial medication and any possible interactions between the investigational drug(s) and a Non-Investigational Medicinal Product (NIMP) / Auxiliary Medicinal Product (AMP)

The following should also be recorded as an (S)AE in the CRF and SAE form (if applicable):

- Worsening of the underlying disease or of other pre-existing conditions (see <u>Section</u> <u>5.3.6.3</u> below)
- Changes in vital signs, ECG, physical examination and laboratory test results, if they are judged clinically relevant by the Investigator.

If such abnormalities already pre-exist prior trial inclusion they will be considered as baseline conditions.

All (S)AEs, including those persisting after individual patient's end of trial must be followed up until they have resolved, have been sufficiently characterised, or no further information can be obtained.

## **Pregnancy**

In rare cases pregnancy or pregnancy in a female partner of a male participant may occur in a clinical trial. Once a patient has been enrolled into this clinical trial and has taken trial medication, the Investigator must report immediately (within 24 hours) a potential drug exposure during pregnancy (DEDP) including drug exposure to female partners of male participants to the sponsor's unique entry point (country-specific contact details will be provided in the ISF). The Pregnancy Monitoring Form for Clinical Trials (Part A) should be used.

The outcome of the pregnancy associated with the drug exposure during pregnancy must be followed up and reported to the sponsor's unique entry point on the Pregnancy Monitoring Form for Clinical Trials (Part B).

The ISF will contain the Pregnancy Monitoring Form for Clinical Trials (Part A and B).

As pregnancy itself is not to be reported as an AE, in the absence of an accompanying SAE and/or AESI, only the Pregnancy Monitoring Form for Clinical Trials and not the SAE form is to be completed. If there is an SAE and/or AESI associated with the pregnancy an SAE form must be completed in addition.

#### 5.3.6.3 Exemption to (S)AE Reporting

Exempted outcome events are:

Disease progression Malignant neoplasm progression Neoplasm progression

## Boehringer Ingelheim BI Trial No.: 1280.18

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Disease Progression is a trial endpoint for analysis of efficacy and as such is exempted from reporting as an (S)AE. Progression of the subject's underlying malignancy will be recorded on the appropriate pages of the (e)CRF as part of efficacy data collection only and will not be reported on the SAE Form. It will therefore not be entered in the safety database (ARISg) and hence not get expeditiously reported. Death due to disease progression is also to be recorded on the appropriate (e)CRF page and not on the SAE Form.

However, when there is evidence suggesting a causal relationship between the study drug(s) and the progression of the underlying malignancy, the event must be reported as an SAE on the SAE Form and on the (e)CRF.

Examples of exempted events of PD may be:

- Progression of underlying malignancy (Progressive disease [PD]): if PD is clearly consistent with the suspected progression of the underlying malignancy as defined by the respective response criteria.
- Hospitalization/Procedures due solely to the progression of underlying malignancy (PD)
- Clinical symptoms and/or signs of progression (without confirmation by objective criteria e.g. imaging, clinical measurement): if the symptom can exclusively be determined to be due to the progression of the underlying malignancy and does meet the expected pattern of progression for the disease under study.

Exempted events are collected and tracked following a protocol-specified monitoring plan. Exempted events will be monitored at appropriate intervals by the Steering Committee.

## **5.3.7** Dose Limiting Toxicities (DLTs)

A <u>dose limiting toxicity</u> (DLT) in this study is defined as an adverse event or laboratory abnormality which 1) is considered related, probably related or possibly related to study drug and 2) meets any of the following criteria, unless that toxicity can be clearly attributed to cancer progression or to another clearly identified etiology:

- CTCAE Grade 3 hyperglycaemia lasting > 48 hours
- CTCAE Grade 4 hyperglycaemia
- CTCAE Grade  $\geq 3$  pneumonitis
- CTCAE Grade  $\geq$  3 febrile neutropenia
- CTCAE Grade 4 hematologic toxicity lasting longer than 5 days
- CTCAE Grade 4 thrombocytopenia of any duration and Grade 3 thrombocytopenia associated with bleeding
- AST or ALT > 5x ULN (for baseline AST/ALT ≤ ULN) or > (baseline value + 4x ULN) (for baseline AST/ALT > ULN)
- CTCAE Grade ≥ 3 diarrhoea, nausea, or vomiting lasting more than 2 days despite maximal supportive care
- CTCAE Grade  $\geq 3$  skin rash despite adequate supportive care measures
- CTCAE Grade  $\geq$  3 fatigue/asthenia lasting for more than seven days
- Grades 3 to 4 hyperlipidaemia (total cholesterol > 400 mg/dL or triglycerides > 500 mg/dL) not improving despite appropriate treatment for 2 weeks

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Any AE necessitating a 2-week treatment interruption (except for hematologic AEs)
- All other non-hematologic toxicities of CTCAE Grade  $\geq 3$  (except alopecia, infusion-related reaction and those mentioned above)
- Any other study drug related toxicity considered significant enough to be qualified as DLT in the opinion of the investigators, and confirmed by the safety review with the BI clinical monitor and BI project physician (TMM), will be reported as a DLT

For the purposes of dose finding, only DLT events that occur during the first treatment period of 28 days will be considered. Decisions regarding dose escalation/de-escalation steps will be made only after discussion between the sponsor and the investigators, and in consideration of all the available safety information. Available data of DLTs occurring after first treatment course and all unusual/unexpected AE at any time during treatment will be considered for the purpose of recommending the dose for cohorts B, C, D (dose finding), E, F, D1 and D2. All DLT events that meet AESI criteria need to be reported immediately to the sponsor's Pharmacovigilance Department within the same timeframe that applies to SAEs, please see Section 5.3.6.2, and documented in the eCRF.

## 5.4 DRUG CONCENTRATION MEASUREMENTS AND PHARMACOKINETICS

#### 5.4.1 Assessment of Pharmacokinetics

## As of 22 Oct 2021, samples for PK are no longer collected for ongoing patients.

PK samples will be collected from all patients in this trial at the time points specified in the Flow Chart and in Appendix 10.2 (minimal deviations in the time scheduled will not be considered as protocol violation). The actual sampling date and time for blood samples will be reported in the eCRF and will be used for determination of PK parameters. To allow a valid PK analysis, it is of utmost importance to document the exact clock time of trial medication administration and blood sample collection. Any occurrence of vomiting should be documented as well. The duration of the xentuzumab infusion will be reported with a start and end time in the eCRF. Every attempt should be made to adhere to an infusion time of approximately 1 h for xentuzumab with a constant infusion rate.

At days of PK sampling of abemaciclib (cohorts E, F, D1 and D2) patients should be instructed to take their morning dose of abemaciclib in the hospital (and not at home as usual). This is necessary in order to allow for a valid PK sampling schedule. For details of the PK sampling schedule, please refer to Appendix 10.2.

PK parameters will be evaluated according to <u>Section 5.1.3</u>. Non-compartmental PK analysis will be done in order to calculate PK parameters (<u>Section 5.1.3</u>) using Phoenix WinNonlin (or other validated software) according to BI SOP 001-MCS-36-472 (current version).

c09049566-10 Trial Protocol


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 5.4.2 Methods of sample collection

## As of 22 Oct 2021, samples for PK and ADA are no longer collected for ongoing patients.

Blood samples should be obtained from the arm opposite to the arm used for infusion. In case a central venous access is used for infusion, the blood sample can be collected from either forearm. The actual sampling date and time (24-hour clock time) for each sample has to be recorded accurately.

For quantification of xentuzumab plasma concentrations, blood samples will be taken at the time points listed in the <u>Flow Chart</u> under PK sampling. A detailed sampling schedule in the respective cohorts and courses is shown in <u>Appendix 10.2</u>. For details on blood volumes to be collected, sample handling and logistics refer to the ISF (Laboratory Manual).

For quantification of plasma concentrations of abemaciclib and relevant metabolites, blood samples will be taken at the time points listed in the <u>Flow Chart</u> under PK sampling. A detailed sampling schedule in the respective cohorts and courses is shown in <u>Appendix 10.2</u>. For details on blood volumes, sample handling and logistics refer to the ISF (Laboratory Manual).

For quantification of fulvestrant plasma concentrations, blood samples will be taken at the time points listed in the <u>Flow Chart</u> under PK sampling. A detailed sampling schedule in the respective cohorts and courses is shown in <u>Appendix 10.2</u>. For details on blood volumes, sample handling and logistics refer to the ISF (Laboratory Manual).

For ADA assessment, blood will be taken at the time points listed in the <u>Flow Chart</u> under ADA sampling. The exact timing of ADA sampling before, during and beyond the treatment phase is also shown in <u>Appendix 10.2</u>. For details on blood volumes, sample handling and logistics refer to the ISF (Laboratory Manual).

Plasma samples from the study may be used for further methodological investigations, e.g., stability testing. However, only data related to the analyte and/or bioanalytical assay will be generated by these additional investigations. Both PK and ADA study samples will be discarded after completion of the additional investigations but not later than 5 years after the final study report has been signed.




Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 5.4.4 Pharmacokinetic – Pharmacodynamic Relationship

No formal analysis of a pharmacokinetic/pharmacodynamic relationship is planned. Correlation between drug concentration and any type of response may be made if appropriate. Data may also be used to develop pharmacokinetic/pharmacodynamic models using nonlinear mixed effect modelling techniques, if feasible. For this purpose data may also be combined with those from other trials. Modelling activities will be planned and documented separately.

## 5.5 ASSESSMENT OF BIOMARKER(S)

# As of 22 Oct 2021, samples for biomarkers are no longer collected for ongoing patients.

In this clinical study explorative biomarkers will be measured and analysed. These analyses are hypothesis generating and will be used to expand our understanding of the study drug and the disease. Participation in the biomarker analyses is mandatory for patients from all cohorts.

#### Evaluation of molecular and biochemical biomarkers in tumour tissue:

Tumour tissue samples will be collected from all patients (except when there is no tumour tissue sample available) to explore the potential influence of molecular and biochemical alterations within the tumour on treatment response and outcome. No biopsies should be done for the only purpose of obtaining tumour tissue for this trial. Tumour tissue samples will be analysed for:

- Mutations and copy number alterations in genes related to the study drugs and involved in tumourigenesis, such as genes of the IGF, PI3K/mTOR, Ras/MAPK, Rb and related signalling pathways (e.g. IGF1R, PIK3CA, PTEN, KRAS, MYC, CCND1, CDK4, CDK6, RB1 and CDKN2A)
- RNA expression of IGF, PI3K/mTOR, Ras/MAPK and cell cycle-related signalling pathways (e.g. IGF1, IGF2, IGFBP-family genes, MYC, CCND1, CDK4, CDK6)
- Expression of Rb and p16 proteins via biochemical methods (e.g. IHC). According to additional knowledge gained from other studies with xentuzumab and/or abemaciclib broader analysis of the samples (including immunohistochemistry/in-situ hybridization/sequencing of e.g. IGF-1/2, PTEN, pAKT, pS6, Ki67) might be conducted to e.g. address predictive biomarkers, exceptional response or resistance mechanisms.

Individual analyses from tumour tissue will be prioritized based on availability of sufficient tissue material.

#### **Molecular evaluation in blood:**

Three kinds of blood samples will be collected for genomic analyses from blood and plasma.

One blood sample will be used to isolate genomic DNA, which will be used as a reference (normal tissue) to distinguish tumour acquired somatic mutations and will be analysed for the indicated panel of genes as in the tumour tissue and/or in the cfDNA (see above).

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Secondly, blood samples will be collected and used to isolate circulating nucleic acids such as e.g. cfDNA from plasma. Subsequent analyses of plasma cfDNA may be used for example to detect somatic mutations in cancer genes, e.g. IGF pathway-related and known cancer driver genes. Additionally, changes in nucleic acid concentration over course of treatment may be explored. Analysis of cfDNA provides a non-invasive technique that might help to find potential biomarkers to predict treatment response or resistance mechanisms to the study drug (R14-1645).

Thirdly, blood samples will be collected and used to evaluate exosomal RNA from plasma. Subsequent analyses of plasma exosomal RNA using standard molecular technology will include, but not be limited to, cell cycle and proliferation related genes, e.g. CCND1, Ki67, RB1, CDK4, CDK6 and CDKN2A.

#### Methods of sample collection

Formalin fixed paraffin embedded (FFPE) tumour tissue, preferably FFPE blocks, from the most recent time point before entering the study will be collected during screening or at a later timepoint (see Flow Chart, Table 5.5: 1 and Table 5.5: 2 and Appendix 10.3). The FFPE blocks will be used to prepare 25 slides at 5µm thickness. Alternatively, 25 freshly prepared slides at 5µm thickness from FFPE block can be provided but need to be prepared under RNase-free conditions. Isolated nucleic acids (e.g. DNA and RNA) from the tumour tissue will be analysed for genomic alterations such as somatic mutations and copy number alterations as well as RNA expression levels as described above.

In addition, patients will be asked for three kinds of blood samples:

One blood sample will be collected at C1V1 before treatment (see <u>Flow Chart</u> and <u>Table 5.5:</u> 1 and <u>Table 5.5:</u> 2). The isolated DNA will be analysed for genomic alterations in a panel of cancer -related genes as mentioned for the tissue and/or the cfDNA above serving as a reference to allow distinction of tumour-acquired somatic mutations from normal tissue.

For analysis of circulating nucleic acids, blood samples will be collected in plasma preparation tubes at each indicated time point before treatment (Run-in and/or C1V1), at C3V1 and at EOTV (see <u>Flow Chart</u> and <u>Table 5.5: 1</u> and <u>Table 5.5: 2</u>). The samples will be used to isolate and analyse circulating nucleic acids as described above.

For exosomal RNA analyses, blood samples will be collected in EDTA tubes at each indicated time point before treatment is administered to patient (where applicable): At Run-in and/or C1V1, at C1V3 (Day 15), at C2V1, at C3V1, at C4V1 onwards and at the EOTV, (see Flow Chart and Table 5.5: 1 and Table 5.5: 2). Separation of the plasma from the remaining blood should be performed. The samples will be used to isolate circulating exosomes and analyse exosomal components such as e.g. RNA.

Boehringer Ingelheim BI Trial No.: 1280.18

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 5.5: 1 Overview PGx sample collection timepoints for cohorts A-D (dose finding) and expansion cohorts D1, D2 and F.

| | Timepoints | | | | | | |
|---|---|---|---|---|---|---|---|
| Sample | Screening | C1V1 | C1V3 | C2V1 | C3V1 | C4V1<br>onwards <sup>1</sup> | EOT |
| Archival tumour tissue | X | | | | | | |
| PGx blood (gDNA) | | X | | | | | |
| PGx Plasma (cfDNA) | | X | | | X | | X |
| PGx Plasma (Exosomes) | | X | X | X | X | X | X |
| DNA<br>banking | | X | | | | | |

<sup>&</sup>lt;sup>1</sup> Refer to the central laboratory manual instructions.

Table 5.5: 2 Overview PGx sample collection timepoints for cohort E

| | Timepoints | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Sample | Screening | Run-<br>in V1 | C1V1 | C1V3 | C2V1 | C3V1 | C4V1<br>onwards <sup>1</sup> | ЕОТ |
| Archival tumour tissue | X | | | | | | | |
| PGx blood (gDNA) | | X | | | | | | |
| PGx Plasma (cfDNA) | | X | X | | | X | | X |
| PGx Plasma<br>(Exosomes) | | X | X | X | X | X | X | X |
| DNA<br>banking | | X | | | | | | |

<sup>&</sup>lt;sup>1</sup> Refer to the central laboratory manual instructions.

Remaining samples from pharmacogenomic analyses such as tumour tissue, blood or plasma samples (and isolated DNA and RNA) will be destroyed no later than 1 year after the end of the trial if no optional consent for sample biobanking is obtained from the patient (see <u>Section 5.5.1</u>).


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Detailed instructions for pharmacogenomic sampling, handling and shipment of samples will be provided in the lab manual.

The biomarker analyses will be performed by Boehringer Ingelheim or a central laboratory authorized by Boehringer Ingelheim.

#### **Protein biomarkers from blood:**

The following protein biomarkers are planned to be examined in this trial:

- Free and total IGF-1 in serum (and optionally free and total IGF-2, dissociable IGF-1 and IGF-2, and total IGFBP-3)
- Phosphorylated and total IGF-1R protein in platelet-rich plasma

Serial collection of blood samples for the assessment of these markers is mandatory. As medical knowledge in this field is constantly evolving, other tissue/blood biomarkers that come to be known as potentially relevant prognostic/predictive markers of treatment response may also be explored via available tissues/blood or acquisition of additional tumour tissues/blood. Biomarkers that come to be known or emerge as not relevant during the study may be discontinued.

All samples must be adequately labelled by the study site personnel. Details about blood sample collection, plasma/serum preparation, required tubes, labelling of tubes, storage and shipment (frequency and addresses) will be provided in the ISF (laboratory manual).

#### Biomarker assessments in blood samples

Levels of free and total IGF-1 (optionally IGF-2 and the amount of IGFBP-3) will be relatively quantified in serum using validated immunoassays. Free IGF-1 (and IGF-2) is defined as the fraction of total IGF-1 (and total IGF-2) that can be bound by xentuzumab under in vitro assay conditions. Dissociable IGF-1 (and IGF-2) is defined as the fraction of total IGF-1 (and total IGF-2) that can be bound by xentuzumab under modified, i.e. more highly diluted in vitro assay conditions. Total IGF-1 (and total IGF-2) is quantified in serum samples after splitting the IGF-IGF-binding protein complexes and the IGF-xentuzumab immune complexes. Optionally, total IGFBP-3 will be relatively quantified in serum using a validated immunoassay.

For quantification of free and total IGF-1 (and optionally free and total IGF-2 and IGFBP-3), blood will be taken from a forearm vein at those time points specified in the <u>Flow Chart</u> and <u>Appendix 10.2</u>.

Quantification of IGF-2 and IGFBP-3 will be performed if scientifically justified based on results of ongoing clinical studies with xentuzumab (e.g. 1280.4).

#### Biomarkers in platelet-rich plasma

In platelet rich plasma, the level of phosphorylated and total IGF-1R will be analysed via immunoassay as an exploratory target engagement biomarker. Based on insights from earlier clinical trials with xentuzumab or abemaciclib, the analysis of other proteins involved in IGF, insulin and/or cyclin-dependent kinase mediated signalling might be added.

0049566-10 Trial Protocol


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

For this purpose, blood samples will be taken from a forearm vein at screening and at those time points specified in the Flow Chart and in Appendix 10.2.

All analyses will be performed at Boehringer Ingelheim or a CRO with given authorization by BI.

Remaining samples from protein biomarker analyses such as tumour tissue and blood samples will be destroyed no later than 5 years after the end of the trial if no optional consent for sample biobanking is obtained from the patient (see Section 5.5.1).

## 5.5.1 Biobanking

If permission for biobanking is obtained from the patient via an optional informed consent, any leftover samples from the study might be stored at Boehringer Ingelheim or contract research organization for up to 30 years unless specified otherwise in the protocol.

These samples may be used to further address scientific questions as new information in regard to the disease or the study drug becomes available.

## 5.5.1.1 DNA Banking

One blood sample will be used for DNA Banking if participation and the separate informed consent is agreed upon by the patient as noted below. The DNA Banking sample, derived from the original blood sample, will be stored at the sponsor. The stored DNA may retrospectively be analysed, e.g. to identify whether there are other genetic factors that could contribute to a better therapeutic outcome or a higher risk of developing treatment-related adverse drug reactions.

Note: Participation in the DNA Banking sampling is voluntary and not a prerequisite for participation in the trial. The DNA Banking sample will be stored for up to 30 years after separate informed consent is given in accordance with local ethical and regulatory requirements.

A blood sample for DNA banking will be collected in a PAXgene Blood DNA tube preferably at C1V1 or at Run-in Visit 1 for cohorts with Run-in period (or at a later time) (see <u>Flow Chart</u> and <u>Table 5.5: 1</u> and <u>Table 5.5: 2</u>) for those patients who signed a separate PGx informed consent for DNA Banking.

#### 5.6 OTHER ASSESSMENTS

The following patient demographic, baseline characteristics and medical history will be collected on the eCRF:

- 1. General demography including sex, birth date and race as allowed by local law, information on smoking and alcohol history. Collection of race and/or ethnic information is necessary in this study because this is a multi-national trial and race and/or ethnicity are known to be associated with biology and outcome of breast cancer and NSCLC. Foreign regulatory agencies may request data or analysis based on race/ethnic information.
- 2. Medical history/current medical conditions (including history of menopause, prior and concomitant medications and concomitant diagnosis)

9566-10 Trial Protocol


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 3. History and current disease status including date of first histological diagnosis (month and year may be sufficient), type of tumour histology, tumour grade, other diagnosis information such as mutations or receptors overexpression, known tumour genetic alterations, TNM staging, number and locations of metastatic sites (bone, liver, lung, peritoneum, brain, other) at the study entry
- 4. Previous anticancer treatments: previous surgery, hormonotherapy, chemo-, targeted, or radiation therapy will be reported including setting (neoadjuvant vs. adjuvant vs. therapeutic), start and end dates (month and year may be sufficient), the therapy protocol with the number of courses (chemotherapy), total radiation dose and radiation field (radiotherapy), the best response obtained (complete response, partial response, stable disease/non-CR/non-PD, progressive disease, unknown) and reason for treatment discontinuation

## 5.6.1 Assessment of Immunogenicity

# As of 22 Oct 2021, samples for immunogenicity are no longer collected for ongoing patients.

For the determination of anti-drug antibodies (ADA) against xentuzumab, blood samples will be taken from a forearm vein in an EDTA anticoagulant blood drawing tube at time points specified in the <u>Flow Chart</u> and in <u>Appendix 10.2</u>. Details about blood sample collection, EDTA plasma preparation, storage and shipment will be provided in a laboratory manual.

A qualitative screening for anti-drug antibodies against xentuzumab in the plasma samples will be performed using a validated immunoassay with xentuzumab as capture reagent. The assay enables the sensitive detection of various types of anti-xentuzumab immunoglobulins. ADA samples will be analysed in a multi-tiered approach (Screening, confirmatory and Titration) where screening positive samples will be confirmed and the confirmed positive samples will be tested in titration.

To further characterize the immune response of the ADA, additional analysis may be conducted after the completion of this study. The results will be reported separately. For this purpose samples will be stored beyond end of study for a maximum period of 5 years or until termination of the development project, whichever occurs first.

A detailed description of the assay will be available prior to the start of sample analysis.

#### 5.7 APPROPRIATENESS OF MEASUREMENTS

The RECIST criteria version 1.1 (Appendix 10.4) to be used for evaluation of tumour response are well established and scientifically accepted. The Common Terminology Criteria, CTCAE version 4.03, 14 June 2010 are used in the assessment of adverse events in cancer patients. All measurements performed during this trial will be to monitor safety and tolerability of xentuzumab in combination with abemaciclib, with or without hormonal therapy, to determine the MTD and /or recommended phase II doses of these combinations.

c09049566-10

04 Mar 2022

**Trial Protocol** 


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The scheduled assessments are to monitor drug induced changes in respect to vital signs, standard laboratory values and ECG. Tumour evaluations are necessary for determination of tumour response to treatment and possible PD effects. Pharmacokinetic analysis and biomarker analysis are necessary for correlation with therapeutic outcome. Immunogenicity testing will ensure the detection of any anti-drug antibody reactions as a result of the infusion of xentuzumab.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 6. INVESTIGATIONAL PLAN

#### 6.1 VISIT SCHEDULE

All patients must provide written informed consent (ICF) before any study related screening procedures can be performed. Allowable time windows for visits are included in the <u>Flow Chart.</u>

Investigational drugs xentuzumab and abemaciclib will be dispensed at each visit according to the <u>Flow Chart.</u> This also applies to letrozole, anastrozole and fulvestrant in the corresponding cohorts (B, C, D (dose finding), F, D1 and D2)

Patients will receive a new medication kit number through the IRT system on each occasion for medications supplied by the sponsor.

All screening assessment including tumour assessments must be completed within 28 days of start of run-in/C1V1. However, upon clinical assessment, if a patient presents with clinical symptoms of progressive disease, the investigator may use clinical judgement to determine whether to have the patient undergo another scan prior to starting treatment. Tumour assessments required for study participation which are completed as part of Standard of Care before the patient sign the ICF can be used for the screening assessments if they are completed within the allowed timeframe.

All patients are to adhere to the visit schedule as specified in the <u>Flow Chart.</u> In the event of any study drug interruption or delay of treatment, the tumour assessment schedule should not be changed.

Blood samples for pharmacokinetics, biomarkers and immunogenicity will be collected from all patients in all cohorts as per <u>Appendix 10.2</u>. Actual clock time for study drug administration and for each blood draw needs to be documented in the eCRF.

On visit days when safety lab is scheduled, patients should show up in fasting condition, the blood draw can be done up to one day prior to the scheduled date.

In situations where a patient is unable to attend a clinic visit, the investigator must assess the risk-benefit for the individual patient and may decide to perform a visit remotely if this is in the best interests of the patient and if agreed with the sponsor.

#### 6.2 DETAILS OF TRIAL PROCEDURES AT SELECTED VISITS

#### 6.2.1 Screening and run-in period(s)

#### Screening Period

Refer to the <u>Flow Chart</u> for procedure details. Please review <u>Section 3.3.2</u> and <u>3.3.3</u> for eligibility criteria.

Patients who failed screening may repeat the screening after discussion between investigator and sponsor providing that reasons for screening failure were reversible and have resolved.

All screening assessments including tumour imaging scan and ECG must be completed within 28 days of start of run-in/C1V1.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The provision of tumour tissue is mandatory when available. Please refer to <u>Appendix 10.3</u> and Table 5.5: 1 and Table 5.5: 2 for details.

Demographics (sex, birth date and race as per each country regulation) and baseline conditions will be collected during the screening visit (See Section 5.6).

Cancer history will also be obtained.

#### Run-in Period (only applicable to cohort E)

Refer to the Flow Chart, Table 5.5: 2 and Appendix 10.2 for details.

Prior to starting therapy with xentuzumab, patients will receive continuous daily abemaciclib for a 9-days run-in period. Abemaciclib and patient's diary should be dispensed on Day -9 of run-in.

Both, on day -9 and on day -1 of the run-in period, patients must come fasted to the study site and must not take abemaciclib until they have been instructed to do so at the clinic visit.

On Day -9 of run-in, prior to the administration of abemaciclib, blood samples for biomarkers, pharmacokinetics, ADA, etc. will be collected as well as a safety lab blood draw. Please see <u>Appendix 10.2.2.1</u> and <u>Table 5.5: 2</u>.

On Day -1 of the run-in period, PK samples must be collected before and after the administration of abemaciclib. Please see Appendix 10.2.2.1.

#### 6.2.2 Treatment period(s)

Every treatment course is 28 days. All subsequent visit dates should be calculated based on Course 1 Visit 1 date. If a visit is missed there will be no re-scheduling; if a patient should attend the study site between the "missed" and the next scheduled visit, then the missed visit assessments should be performed except for xentuzumab infusion. The current date and the reason for the delay must be noted in the medical records.

One or more visits can be skipped in case of treatment interruption. However, in the event of any study drug interruption or delay of treatment, the tumour assessment schedule will not be changed.

In this trial, patients may be hospitalized for the day of xentuzumab treatment and PK sampling at the discretion of the investigator; patients may be discharged if tolerated the treatment well and no safety concerns are present as judged by the investigator. Hospitalizations for this purpose should not be recorded as SAEs.

#### 6.2.2.1 Cohort A, B, C, and D (dose finding)

Refer to the Flow Chart and Appendix 10.2.1 for details.

Course 1, Visit 1 (Day 1 of 1st treatment course)

All procedures must be completed on day 1 of Course 1 except for safety labs, which can be performed 1 day prior to the scheduled visit. Patients should come fasted to the study site for safety labs.

Sufficient abemaciclib should be made available for the patient.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

ECG will be collected prior to xentuzumab infusion.

Pharmacogenomics blood sample to evaluate exosomal RNA, blood sample to isolate genomic DNA, and a blood sample to analyse circulating nucleic acids will be collected before treatment. Also, blood samples for PK, biomarkers and immunogenicity will be collected during the visit. Please see <u>Appendix 10.2.1.1</u> and <u>Table 5.5: 1</u> for details on sampling time points during this visit.

Cohort B: Letrozole will be also dispensed at this visit.

Cohort C: Anastrozole will be also dispensed at this visit.

Cohort D: Fulvestrant will be also administered at this visit.

Course 1, Visit 2 (Day  $8\pm1$  of  $1^{st}$  treatment course)

Patients should come fasted to the study site for safety labs.

On Course 1 day 8, **prior** to the administration of xentuzumab infusion, trough PK as well as biomarker and immunogenicity blood samples must be collected. Please see <u>Appendix 10.2.1.1</u> for details on the sampling schedule for this visit.

Course 1, Visit 3 (15  $\pm 1$  days after start of xentuzumab)

Patients should come fasted to the study site for safety labs.

ECG will be collected prior to xentuzumab infusion.

Pharmacogenomics blood sample to evaluate exosomal RNA will be collected before treatment. This sample will be used to evaluate exosomal RNA. Please refer to <u>Table 5.5: 1</u>. Cohort D: Fulvestrant will be also administered at this visit.

Course 1, Visit 4 (22  $\pm 1$  days after start of xentuzumab) Patients should come fasted to the study site for safety labs.

Course 2 (Day 1, 8, 15,  $22 \pm 2$  days) and all subsequent visits

Refer to Flow Chart, Table 5.5: 1 and Appendix 10.2.1 for details.

Pharmacogenomics blood sample to evaluate exosomal RNA will be collected before treatment at Course  $\geq 2$  day 1.

PK, biomarkers, pharmacogenomics and ADA samples are also applicable to these visits. Please see <u>Table 5.5: 1</u> and <u>Appendix 10.2.1.2</u> for details on the samples to be obtained.

Safety labs on day 15±2 are only applicable to course 2.

6.2.2.2 Cohort E

Refer to the Flow Chart, Table 5.5: 2 and Appendix 10.2.2 for details.

Course 1, Visit 1 (Day 1 of 1st treatment course)

All procedures must be completed on day 1 of Course 1 except for safety labs, which can be performed 1 day prior to the scheduled visit. For safety labs and PK purposes patients should

## Boehringer Ingelheim BI Trial No.: 1280.18

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

come fasted to the study site and must not take abemaciclib until they have been instructed to do so at the clinic visit.

Sufficient abemaciclib should be made available for the patient at this visit.

ECG will be collected prior to xentuzumab infusion.

Pharmacogenomics blood sample to evaluate exosomal RNA will be collected before treatment (Flow Chart and Table 5.5: 2).

Blood samples for PK, biomarkers, pharmacogenomics and immunogenicity will also be collected during this visit. Please see <u>Table 5.5: 2</u> and <u>Appendix 10.2.2.1</u> for sampling schedule details.

Course 1, Visit 2 (Day  $8\pm1$  of  $1^{st}$  treatment course)

Patients should come fasted to the study site for safety labs.

On Course 1 day 8, **prior** to the administration of xentuzumab infusion, one trough PK as well as biomarker and immunogenicity blood samples must be collected. Please see <u>Appendix 10.2.2.1</u> for details on sampling schedule for this visit.

Course 1, Visit 3 (15  $\pm 1$  days after start of xentuzumab)

Patients should come fasted to the study site for safety labs.

ECG will be collected prior to xentuzumab infusion.

Pharmacogenomics plasma sample will be collected before treatment. This sample will be used to evaluate exosomal RNA (<u>Flow Chart</u> and <u>Table 5.5: 2</u>). Please see <u>Appendix 10.2.2.1</u> for details on sampling schedule.

Course 1, Visit 4 (22  $\pm 1$  days after start of xentuzumab)

Patients should come fasted to the study site for safety labs. Patient's diary will be dispensed to the patient at this visit.

Course 2 (Day 1, 8, 15,  $22 \pm 2$  days) and all subsequent courses/visits Refer to the Flow Chart, Table 5.5: 2 and Appendix 10.2.2.2 for details.

Pharmacogenomics blood sample to evaluate exosomal RNA will be collected before treatment at Course ≥2 day 1 (Flow Chart and Table 5.5: 2).

PK, biomarkers, pharmacogenomics and ADA samples will also be drawn at these visits. Please see <u>Table 5.5: 2</u> and <u>Appendix 10.2.2.2</u> for details on the sampling schedule.

At course 2 visit 1, and for PK purposes, patients should come fasted to the study site and must not take abemaciclib until they have been instructed to do so at the clinic visit. Safety labs on day 15±2 are only applicable to course 2

6.2.2.3 Cohorts D1, D2 and F

Refer to the revised and reduced Flow Chart, for details.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 6.2.3 Follow Up Period and Trial Completion

#### 6.2.3.1 End of treatment visit

End of Treatment Visit (0-7 days after permanent discontinuation of study drugs)

Refer to the <u>Flow Chart</u> for details. The patient must return all study drugs, and the site must document the reason for permanent discontinuation of study medication. If permanent discontinuation of study drug occurs during a scheduled visit, examinations as defined for EOTV should be performed instead of the examinations for the scheduled visit.

## 6.2.3.2 Follow-up period

All patients must have a follow-up visit 42 days (+7days) after the permanent discontinuation of study drugs.

This follow-up period is aimed for collection of additional AE and PD information. Refer to the Flow Chart for details.

The follow-up for progression period will end at the earliest if one of the following events is met:

- · Lost to follow-up
- · Disease progression
- · Start of a new anti-cancer therapy
- · Death
- · End of whole trial as specified in Section 8.6

Blood samples for soluble biomarkers, PK and ADA must be obtained at this visit. Please refer to <u>Appendix 10.2</u> for sampling schedule details.

#### 6.2.3.3 Trial Completion

Trial completion for an individual patient:

A patient is considered to have completed the trial in case any of the following applies:

- Completion of planned follow-up period (follow-up visit)
- Lost to follow-up
- Refusal to be followed-up
- Death

The end of the trial is defined in Section 8.6

c09049566-10 Trial Protocol


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 7. STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

#### 7.1 STATISTICAL DESIGN - MODEL

This trial will be performed as an open-label study. The primary objective of the dose finding cohorts of this trial is to determine the MTD and the RP2D of:

- \* Cohort A: xentuzumab in combination with abemaciclib (without endocrine background therapy)
- \* Cohort B: xentuzumab in combination with abemaciclib on a background therapy of letrozole
- \* Cohort C: xentuzumab in combination with abemaciclib on a background therapy of anastrozole
- \* Cohort D (dose finding): xentuzumab in combination with abemaciclib on a background therapy of fulvestrant

To determine the MTD, patients are entered sequentially into escalating or de-escalating dose-level cohorts. For each treatment combination, the dose finding will be guided by a Bayesian 5-parameter logistic regression model with overdose control (R15-4233, Chapter 6).

This logistic regression model is defined as follows. Let  $\pi_{1,d1}$  be the probability of having a DLT when giving dose  $d_1$  of xentuzumab as monotherapy, and  $\pi_{2,d2}$  the probability of having a DLT when giving dose  $d_2$  of the combination partner abemaciclib as monotherapy, respectively. A logistic regression is used to model the dose-toxicity relationship for each of these drugs individually:

```
Xentuzumab: logit(\pi_{1,d1}) = log(\alpha_1) + \beta_1 log(d_1/d_1^*)
Abemaciclib: logit(\pi_{2,d2}) = log(\alpha_2) + \beta_2 log(d_2/d_2^*)
```

Here, the doses  $d_1^* = 1000$  mg i.v. once weekly and  $d_2^* = 150$  mg every 12 hours represent the reference doses for xentuzumab and abemaciclib, respectively.

Assuming no toxicity interaction between the two compounds, the probability of a DLT when giving the combination dose  $d_1$ ,  $d_2$  is obtained as

```
\pi^0_{12,d1,d2} = \pi_{1,d1} + \pi_{2,d2} - \pi_{1,d1}\pi_{2,d2} with corresponding odds odds(\pi^0_{12,d1,d2})= \pi^0_{12,d1,d2}/(1 - \pi^0_{12,d1,d2}).
```

In order to account for a potential positive (higher toxicity than expected under independence) or negative (lower toxicity than expected under independence) interaction between xentuzumab and abemaciclib, a dose-dependent interaction term  $-\infty < \eta < \infty$  is introduced in the model by the following definition:

```
odds(\pi_{12,d1,d2}) = odds(\pi^0_{12,d1,d2}) exp(\eta d<sub>1</sub>/d<sub>1</sub>* d<sub>2</sub>/d<sub>2</sub>*) and \pi_{12,d1,d2} is used in the likelihood r_{d1,d2} \sim \text{Binomial}(n_{d1,d2},\pi_{12,d1,d2})
```

where  $r_{d1,d2}$  denotes the random variable describing the observed number of DLTs in  $n_{d1,d2}$  patients at the dose combination  $d_1, d_2$ .
Trial Protocol


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Since a Bayesian approach is applied, prior distributions f for each of the parameter vectors  $\theta_1 = (\log(\alpha_1), \log(\beta_1)), \theta_2 = (\log(\alpha_2), \log(\beta_2))$  and for the interaction term  $\eta$  need to be specified.

The prior distributions for  $\theta_k$  will be specified as a mixture of two bivariate normal distributions.

$$\begin{split} f(\theta_k) &= a_{1,k} \ f_1(\theta_k) + a_{2,k} \ f_2(\theta_k) \\ \text{with} \end{split}$$

 $a_{1,k}$ ,  $a_{2,k}$  the prior mixture weights  $(a_{1,k} + a_{2,k} = 1)$ , k = 1,2 and

 $f_i(\theta_k) = MVN(\mu_{ik}, \sum_{ik})$  a bivariate normal distribution with mean vector  $\mu_{ik}$  and covariance matrix  $\sum_{ik}$  where

$$\Sigma_{ik} = \begin{pmatrix} \sigma^2_{ik,11} & \sigma_{ik,11}\sigma_{ik,22}\rho_{ik} \\ \sigma_{ik,11}\sigma_{ik,22}\rho_{ik} & \sigma^2_{ik,22} \end{pmatrix}$$

Mixture prior distributions have the advantage that they allow for specification of different logistic dose-toxicity curves, therefore making the prior more robust.

A weakly informative normal prior distribution will be used for  $\eta$ .

The estimated probability of DLT  $\pi_{12,d1,d2}$  at each dose combination  $d_1$ ,  $d_2$  from the model will be summarized using the following intervals:

- \* Under dosing: [0.00, 0.16)
- \* Targeted toxicity: [0.16, 0.33)
- \* Over dosing: [0.33, 1.00]

The BLRM recommended dose combination for the next cohort is the combination with the highest posterior probability of the DLT rate falling in the target interval [0.16, 0.33) among the dose combinations fulfilling the EWOC principle. Per EWOC it should be unlikely (<25% posterior probability) that the DLT rate at the dose combination will exceed 0.33. However, the maximum allowable dose increment for the subsequent cohort will be no more than 100 % for each drug.

The MTD may be considered reached if one of the following criteria is fulfilled:

- 1. The posterior probability of the true DLT rate in the target interval [0.16 0.33) of the MTD is above 0.50, or
- 2. At least 6 patients have been treated at the MTD.

#### Prior derivation

To determine the prior distributions for  $\theta_1$  and  $\theta_2$ , a meta-analytic predictive (MAP) approach will be used. Toxicity information on xentuzumab and abemaciclib from earlier dose finding studies will be incorporated. Exact details on the evaluation of the model using hypothetical data scenarios and operating characteristics are provided in the statistical appendix; a brief description is given here.

The historical data for xentuzumab and abemaciclib can be found in <u>Table 7.1:1</u> and <u>Table 7.1:2</u>, respectively.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 7.1: 1 Historical data for xentuzumab

| Study | Dose | N of patients with DLTs<br>during MTD evaluation<br>period / N of patients |
|---|---|---|
| 1280.1 (weekly infusion) | 10 mg | 0/3 |
| | 20 mg | 0/3 |
| | 40 mg | 0/3 |
| | 60 mg | 0/3 |
| | 90 mg | 0/3 |
| | 135 mg | 0/3 |
| | 200 mg | 0/3 |
| | 300 mg | 0/3 |
| | 450 mg | 1/6 |
| | 600 mg | 0/3 |
| | 800 mg | 0/3 |
| | 1000 mg | 0/13 |
| | 1050 mg | 0/3 |
| | 1400 mg | 0/3 |
| | 1800 mg | 0/3 |
| 1280.15: Japan (weekly infusion) | 750 mg | 0/3 |
| | 1000 mg | 0/9 |
| | 1400 mg | 0/6 |

Table 7.1: 2 Historical data for abemaciclib

| Study | Dose | N of patients with DLTs<br>during MTD evaluation<br>period / N of patients |
|---|---|---|
| Study I3Y-MC-JPBA | 75 mg twice-daily | |
| | 100 mg twice-daily | 0/3 |
| | 150 mg twice-daily | 0/4 |
| | 200 mg twice-daily (=MTD) | 0/3 |
| | 275 mg twice-daily | 1/7 |
| | | 2/3 |

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 7.1: 2 Historical data for abemaciclib (cont.)

| Study | | N of patients with DLTs<br>during MTD evaluation<br>period / N of patients |
|---|---|---|
| Study I3Y-JE-JPBC | 100 mg twice-daily | 0/3 |
| | 150 mg twice-daily | 0/3 |
| | 200 mg twice-daily | 1/6 |

Study I3Y-MC-JPBA: Phase 1 Study of a CDK4/6 Dual Inhibitor in Patients with Advanced Cancer. Study I3Y-JE-JPBC: Phase 1 Study of LY2835219 in Japanese patients with Advanced Cancer.

The following steps were used to derive the prior distributions for all parameters:

- 1.  $\theta_1$ :
- 1. The meta-analytic-predictive prior was derived using the information in <u>Table 7.1:1</u>, allowing for substantial between-trial heterogeneity. This mixture component was assigned 90% mixture weight.
- 2. A second, weakly-informative component was added with 10% mixture weight.
- 2.  $\theta_2$ :
- 1. The meta-analytic-predictive prior was derived using the information in <u>Table 7.1:2</u>, allowing for moderate between-trial heterogeneity. This mixture component was assigned 90% mixture weight.
- 2. A second, weakly-informative component was added with 10% mixture weight.
- 3. η: based on the a priori assumption of no interaction between the two compounds, a normal distribution with mean 0 and standard deviation 0.707 was chosen. At the starting dose combination, the corresponding 95% prior interval covers an up to 4 fold increase (or decrease) in the odds of a DLT over no interaction.

The prior distribution is given in <u>Table 7.1: 3</u>. The corresponding prior probability of a DLT at different dose combinations and the corresponding probabilities of under-dosing, targeted dosing and overdosing are shown in <u>Table 7.1: 4</u>.

As seen in <u>Table 7.1: 4</u>, the dose combination 1000 mg xentuzumab and 150 mg abemaciclib has prior probabilities of overdosing below 25%. Hence, this dose combination fulfils the overdose criterion and is therefore suitable starting dose combination.

Table 7.1: 3 Prior distributions for the combination of xentuzumab and abemaciclib for Cohort A

| Parameter | Means, standard deviations, correlation | Mixture weight |
|---|---|---|
| Component 1: $log(\alpha_1)$ , $log(\beta_1)$ | (-3.697, -0.517), (1.031, 0.816), 0.034 | 0.9 |
| Component 2: $log(\alpha_1)$ , $log(\beta_1)$ | (-4, -0.5), (2, 1), 0 | 0.1 |

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 7.1: 3 Prior distributions for the combination of xentuzumab and abemaciclib for Cohort A (cont.)

| Parameter | Means, standard deviations, correlation | Mixture<br>weight |
|---|---|---|
| Component 1: $\log(\alpha_2)$ , $\log(\beta_2)$ | (-2.515, 0.898), (0.829, 0.808), -0.510 | 0.9 |
| Component 2: $\log(\alpha_2)$ , $\log(\beta_2)$ | (-3, 0.9), (2, 1), 0 | 0.1 |
| η | 0, 0.707, NA | NA |

Table 7.1: 4 Prior probabilities of DLTs for the combination of xentuzumab and abemaciclib for Cohort A

| ıab | lib | Probabili | ty of true DLT | rate in | | | Quanti | les | |
|---|---|---|---|---|---|---|---|---|---|
| Dose<br>xentuzumab | Dose<br>abemaciclib | [0,0.16) | [0.16,0.33) | [0.33,1] | Mean | StD | 2.5% | 50% | 97.5% |
| 750 | 100 | 0.873 | 0.106 | 0.021 | 0.083 | 0.087 | 0.006 | 0.056 | 0.316 |
| 750 | 150 | 0.706 | 0.226 | 0.067 | 0.137 | 0.117 | 0.017 | 0.102 | 0.454 |
| 1000 | 100 | 0.841 | 0.128 | 0.032 | 0.092 | 0.096 | 0.007 | 0.062 | 0.356 |
| 1000 | 150 | 0.664 | 0.238 | 0.098 | 0.150 | 0.134 | 0.015 | 0.109 | 0.517 |

The prior for cohort A may be updated once the trial has started in case new data that can be used will be available. The priors for cohorts B, C, and D(dose finding) will be additionally based on available data from this trial. The priors that are used for each BLRM analysis for the SC meetings will be documented in the SC minutes. The prior that is used for the final analysis will be documented in the TSAP.

### 7.2 NULL AND ALTERNATIVE HYPOTHESES

The analyses in this trial are descriptive and exploratory. No formal statistical test will be performed.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 7.3 PLANNED ANALYSES

No per protocol set will be used in the analysis. However, important protocol violations will be summarised. The TSAP will specify the important protocol violations in detail.

For the determination of the MTD, only MTD evaluable patients will be considered. For the analysis of primary and secondary endpoints of the expansion parts and further endpoints of dose finding and expansion parts, all patients in the treated set (i.e. patients treated with at least one dose of any trial medication, including hormonal therapy) will be included in the analysis. Any other analysis sets will be defined in the TSAP.

The analysis of the primary endpoint of the dose finding cohorts (cohorts A, B, C and D (dose finding) respectively) will be conducted when "last-patient-last-visit-primary-endpoint-dose-finding" has been reached (see <u>Section 8.6</u>).

Primary analysis of expansion cohorts (cohort E, F, D1 and D2) might be done before the end of the study. The further details will be described in TSAP.

The results of each dose finding cohorts (A, B, C, and D (dose finding)) and each expansion cohorts (E, F, D1 and D2) will be analysed separately.

### 7.3.1 Primary endpoint analyses

### For dose finding cohorts A, B, C, and D (dose finding):

In order to identify the MTD, the number of patients with DLTs during the MTD evaluation period at each dose level will be presented. Patients who discontinue during the first treatment course for reasons other than DLT will be excluded from the determination of MTD.

### For expansion cohort E:

Objective response will be analysed in terms of objective response rate, defined as the proportion of patients with best overall response of CR or PR (note that no confirmation is required for best overall response).

### For cohorts D1 and D2:

PFS rate at 18<sup>th</sup> month will be derived using Kaplan Meier method. Cohort D1 for visceral vs. cohort D2 for non-visceral will be displayed separately. The details will be described in the TSAP.

### For expansion cohort F

DC will be analysed in terms of DC rate, defined as the proportion of patients with best overall response of CR, PR, SD lasting for at least 24 weeks or non-CR/non-PD lasting for at least 24 weeks.

## 7.3.2 Secondary endpoint analyses

## For dose finding cohorts A, B, C, and D (dose finding):

There are no secondary endpoints.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### For expansion cohorts E, F, D1 and D2:

The secondary endpoints will be analysed descriptively.

Disease control for Cohorts D1, D2 and E will be analysed in the same way as the primary analysis for Cohort F.

Time to objective response can only be calculated for patients with an objective response: Time to objective response [days] = date of first documented CR or PR – date of first treatment administration  $\pm 1$ .

Duration of objective response can only be calculated for patients with an objective response:

- \* For patients with disease progression or death:

  Duration of objective response [days] = date of outcome date of first assessment indicating objective response +1
- \* For patients without disease progression or death:

  Duration of objective response (censored) [days] = date of outcome date of first assessment indicating objective response +1

The censoring rules for duration of objective response (i.e. outcome and date of outcome) will be described in the TSAP. Only radiological assessments after first assessment indicating objective response should be taken into account.

Duration of disease control will be derived as follows:

- \* For patients with disease progression or death:

  Duration of disease control [days] = date of outcome date of first treatment administration+1
- \* For patients without disease progression or death:

  Duration of disease control (censored) [days] = date of outcome date of first treatment administration +1

The censoring rules for duration of disease control (i.e. outcome and date of outcome) will be described in the TSAP.

Progression-free survival will be derived as follows:

- \* For patients with "event" as an outcome for PFS: PFS [days] = date of outcome – date of first treatment administration + 1
- \* For patients with "censored" as an outcome for PFS: PFS (censored) [days] = date of outcome – date of first treatment administration + 1

Censoring rules for PFS will be described in the TSAP.

Objective response for Cohorts D1, D2 and F will be analysed in the same way as the primary analysis for Cohort E.

c09049566-10 Trial Protocol 



### 7.3.4 Safety analyses

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) coding dictionary. Standard BI summary tables and listings will be produced. All adverse events with an onset between start of treatment and end of the residual effect period (REP), a period of 42 days after the last dose of trial medication, will be assigned to the treatment period for evaluation.

All treated patients will be included in the safety analysis. In general, safety analyses will be descriptive in nature and will be based on BI standards. No hypothesis testing is planned.

Statistical analysis and reporting of adverse events will concentrate on treatment-emergent adverse events. To this end, all adverse events occurring between start of treatment and end of the residual effect period will be considered 'treatment-emergent'. The residual effect period is defined as a period of 42 days after the last dose of trial medication. Adverse events that start before first drug intake and deteriorate under treatment will also be considered as 'treatment-emergent'.

Frequency, severity, and causal relationship of adverse events will be tabulated by system organ class and preferred term after coding according to the current version of the Medical Dictionary for Drug Regulatory Activities (MedDRA).

DLTs will be tabulated for each dose level in the dose escalation cohorts. The tabulation will be done in two ways:

- DLTs with onset in the first treatment course, and
- All DLTs regardless of treatment course at onset

The definition of DLT and determination of MTD are defined in <u>Section 5.3.7</u> and <u>Appendix 10.6</u> respectively.

Laboratory data will be analysed both quantitatively as well as qualitatively. The latter will be done via comparison of laboratory data to their reference ranges. Values outside the reference range as well as values defined as clinically relevant will be highlighted in the listings. Treatment groups will be compared descriptively with regard to distribution parameters as well

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

as with regard to frequency and percentage of patients with abnormal values or clinically relevant abnormal values.

The following analyses will be presented for the laboratory tests:

- Descriptive statistics at each planned assessment,
- Frequency of patients with transitions in CTCAE grade from baseline to worst and last values during treatment, and
- Frequency of patients with possible clinically significant abnormalities.

Additional more in-depth analyses of AEs and laboratory data will be performed as needed and detailed in the TSAP.

Vital signs, physical examinations, ECG, or other safety-relevant data observed at screening, baseline, during the course of the trial and at the end-of-trial evaluation will be assessed with regard to possible changes compared to findings before start of treatment.

### 7.3.5 Pharmacokinetic and pharmacodynamic analyses



Trial Protocol




### 7.4 INTERIM ANALYSES

No formal interim analysis is planned for efficacy.

In the dose finding cohorts A, B, C, and D, the SC and BI study team will continuously monitor and assess safety data to ensure patients' safety, as well as to determine the MTD and/or the RP2D of each dose finding cohorts. If considered necessary, as soon as the MTD and/or the RP2D of a particular dose finding cohort is determined, an evaluation of the safety (and potentially efficacy) aspects will be performed via a snapshot of the database. Results of this evaluation will be documented and stored.

Continuous monitoring of safety data for expansion cohorts E, F, D1 and D2 will be done by the SC and BI study team.

Earlier efficacy analyses than those currently planned may be performed to support future decision making and trial planning.

### 7.5 HANDLING OF MISSING DATA

In general, missing data will not be imputed and all reasonable efforts will be taken during the study to obtain such data.

Missing baseline laboratory values will be imputed by the respective values from the screening visit.

For partial or missing AE onset and/or end dates, BI internal rules will be applied for imputation.

No other imputations will be performed on missing data although every effort will be made to obtain complete information on all adverse events, with particular emphasis on potential DLTs.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### Pharmacokinetics:

Drug concentration-time profiles: Concentration data identified with NOS (no sample), NOR (no valid result), NOA (not analysed), BLQ (below the limit of quantification) and NOP (no peak detectable) will be ignored and not replaced by zero at any time point (including the lag phase). Descriptive statistics of concentrations at specific time points will be calculated only when at least 2/3 of the individuals have concentrations within the validated concentration range.

### Pharmacokinetic parameters:

In the non-compartmental analysis, concentration data identified with NOS, NOR and NOA will not be considered. BLQ and NOP values in the lag phase will be set to zero. The lag phase is defined as the period between time 0 and the first time point with a concentration above the quantification limit. All other BLQ and NOP values of the profile will be ignored. Descriptive statistics of parameters will be calculated only when at least 2/3 of the individual parameter estimates of a certain parameter are available. Pharmacokinetic parameters which cannot be determined will be identified by "not calculated" (NC).

### 7.6 RANDOMISATION

No randomisation will be performed. In the dose finding cohorts, patients will be assigned sequentially to the dose escalation groups. In the expansion cohorts, patients will be assigned to a cohort based upon previous MTD/RP2D. Medication numbers will be allocated by an IRT system.

### 7.7 DETERMINATION OF SAMPLE SIZE

No formal statistical power calculations to determine sample size were performed for this study. Approximately 148 patients (including patients at MTD) will be expected for this trial based on the number of dose levels/cohorts that are tested. Fewer or more patients might be needed based on the recommendation of the SC and BI Trial Team and the criteria specified (see Section 7.1).

### Dose finding cohorts A, B, C and D:

Approximately 12 patients in cohorts A, B, C and D (dose finding) will be needed to define a MTD. In total, approximately 48 patients will be needed for the dose finding cohorts. However, the actual number of patients will depend on the number of dose levels tested.

Based on the simulation study to evaluate operating characteristics of the BLRM (see <u>Appendix 10.6</u>), approximately 12 patients (in mean) are expected to be treated in the dose finding cohort A for the model to have reasonable operating characteristics relating to its MTD recommendation (see <u>Appendix 10.6</u>).

Considering the toxicity profile of individual compounds, we can assume the same number of patients will be needed in the dose finding cohorts B, C and D (dose finding).

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### **Expansion cohort E:**

In expansion cohort E, 20 patients will be treated at the MTD/RP2D.

Assuming a true objective response (OR) rate of 60%, a sample size of 20 patients leads to a probability of 87% of observing at least 10 ORs. If the true OR rate is higher, i.e. 80%, the probability of observing at least 10 ORs is higher than 99%. The probability to observe a false positive signal, i.e. to observe at least 8 ORs if the underlying true OR rate is 20%, is only 3%. Table 7.7: 1 summarizes the probabilities of observing certain OR rates based on different assumptions on underlying OR rates.

Table 7.7: 1 Objective response rates for Cohort E

| True<br>OR<br>rate | Patients | Probabil | Probability to observe at least | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | 7<br>events | 8<br>events | 9<br>events | 10<br>events | 11<br>events | 12<br>events | 13<br>events | 14<br>events | 15<br>events |
| 60% | 20 | 0.99 | 0.97 | 0.94 | 0.87 | 0.76 | 0.60 | 0.42 | 0.25 | 0.13 |
| 80% | 20 | >0.99 | >0.99 | >0.99 | >0.99 | >0.99 | 0.99 | 0.97 | 0.91 | 0.80 |
| 20% | 20 | 0.09 | 0.03 | < 0.01 | < 0.01 | < 0.01 | < 0.01 | < 0.01 | < 0.01 | < 0.01 |

An OR rate of 60% would be considered clinically relevant in NSCLC patients (cohort E).

These assumed OR rates and the expected ORs are according to the current knowledge and expectations regarding xentuzumab and its combination partners. The calculations were performed using R version 3.2.2.

### **Expansion cohorts D1 and D2:**

For each of cohort, D1 for visceral metastasis and D2 for non-visceral metastasis, 30 patients will be recruited respectively and treated at the RP2D<sub>4</sub>.

For cohort D1, assuming a true PFS rate of 60% at 18<sup>th</sup> month, 10 months recruitment period and 20% patient drop rate, a sample size of 30 patients leads to a probability of 62% of observing at least 57% PFS rate at 18<sup>th</sup> month. If the true PFS rate is higher, i.e. 63%, the probability of observing at least 57% PFS rate is higher than 73%. The probability to observe a false positive signal, i.e. to observe at least 57% PFS rate at 18<sup>th</sup> month if the underlying true PFS rate is 43%, is only 8%. Table 7.7: 2 summarizes the probabilities of observing certain PFS rates at 18<sup>th</sup> month based on different assumptions on underlying PFS rates.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 7.7: 2 PFS rates at 18<sup>th</sup> month for cohort D1

| True PFS rate at 18 | Patients | Probability to observe PFS rate at 18th month | | | | |
|---|---|---|---|---|---|---|
| month | | >0.47 | >0.52 | >0.57 | >0.6 | >0.63 |
| 43% | 30 | 0.33 | 0.18 | 0.08 | 0.04 | 0.02 |
| 60% | 30 | 0.90 | 0.79 | 0.62 | 0.51 | 0.39 |
| 63 % | 30 | 0.95 | 0.87 | 0.73 | 0.63 | 0.51 |

For Cohort D2, assuming a true PFS rate of 69% at 18<sup>th</sup> month, 10 months recruitment period and 20% patient drop rate, a sample size of 30 patients leads to a probability of 68% of observing at least 65% PFS rate at 18<sup>th</sup> month. If the true PFS rate is higher, i.e. 75%, the probability of observing at least 65% PFS rate is higher than 87%. The probability to observe a false positive signal, i.e. to observe at least 65% PFS rate at 18<sup>th</sup> month if the underlying true PFS rate is 52%, is only 10%. <u>Table 7.7: 3</u> summarizes the probabilities of observing certain PFS rates at 18<sup>th</sup> month based on different assumptions on underlying PFS rates.

Table 7.7: 3 PFS rates at 18<sup>th</sup> month for cohort D2

| True PFS rate at 18 month | Patients | Probability to observe PFS rate at 18th month | | | | |
|---|---|---|---|---|---|---|
| month | | >0.56 | >0.60 | >0.65 | >0.69 | >0.73 |
| 52% | 30 | 0.35 | 0.22 | 0.10 | 0.04 | 0.02 |
| 69% | 30 | 0.92 | 0.83 | 0.68 | 0.52 | 0.35 |
| 75% | 30 | 0.98 | 0.95 | 0.87 | 0.76 | 0.61 |

An PFS rate of 60% would be considered clinically relevant in each cohorts: visceral metastasis and non-visceral metastasis.

These assumed PFS rates and the expected PFS rates are based on the current knowledge and expectations regarding xentuzumab and its combination partners. The assumed true PFS rate for each cohort is considered clinically relevant. All calculations were performed using R version 3.2.2.

### Cohort F:

In expansion cohort F, 20 patients will be treated at the MTD/RP2D.

Assuming a true DC rate of 60%, a sample size of 20 patients leads to a probability of 87% of observing at least 10 events. If the true DC rate is higher, i.e. 80%, the probability of observing at least 10 events is higher than 99%. The probability to observe a false positive signal, i.e. to observe at least 8 events if the underlying true DC rate is 20%, is only 3%. Table 7.7: 4 summarizes the probabilities of observing certain DC rates based on different assumptions on underlying DC rates.

**Trial Protocol** 


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 7.7: 4 Disease Control rates for Cohort F

| True<br>DC<br>rate | Patients | Probabil | Probability to observe at least | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | 7<br>events | 8<br>events | 9<br>events | 10<br>events | 11<br>events | 12<br>events | 13<br>events | 14<br>events | 15<br>events |
| 60% | 20 | 0.99 | 0.97 | 0.94 | 0.87 | 0.76 | 0.60 | 0.42 | 0.25 | 0.13 |
| 80% | 20 | >0.99 | >0.99 | >0.99 | >0.99 | >0.99 | 0.99 | 0.97 | 0.91 | 0.80 |
| 20% | 20 | 0.09 | 0.03 | < 0.01 | < 0.01 | < 0.01 | < 0.01 | < 0.01 | < 0.01 | < 0.01 |

A DC rate of 60% would be considered clinically relevant in HR+, Her2- locally advanced and/or metastatic breast cancer patients after prior therapy with a different CDK4/6 inhibitor and aromatase inhibitor (cohort F).

These assumed and expected DC rates are according to the current knowledge and expectations regarding xentuzumab and its combination partners. The calculations were performed using R version 3.2.2.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 8. INFORMED CONSENT, TRIAL RECORDS, DATA PROTECTION, PUBLICATION POLICY

The trial will be carried out in accordance with the Medical Devices Directive (93/42/EEC) and the harmonised standards for Medical Devices (ISO 14155, current version).

The trial will be carried out in compliance with the protocol, the ethical principles laid down in the Declaration of Helsinki, in accordance with the ICH Harmonized Tripartite Guideline for Good Clinical Practice (GCP), relevant BI Standard Operating Procedures (SOPs), the EU regulation 536/2014 the Japanese GCP regulations (Ministry of Health and Welfare Ordinance No. 28, March 27, 1997) and other relevant regulations.

Standard medical care (prophylactic, diagnostic and therapeutic procedures) remains in the responsibility of the treating physician of the patient.

The Investigator will inform the sponsor immediately of any urgent safety measures taken to protect the trial subjects against any immediate hazard, and also of any serious breaches of the protocol or of ICH GCP.

The Boehringer Ingelheim transparency and publication policy can be found on the following web page: trials.boehringer-ingelheim.com. The rights of the Investigator and of the sponsor with regard to publication of the results of this trial are described in the Investigator contract. As a rule, no trial results should be published prior to finalization of the Clinical Trial Report.

For Japan only: the rights of the Investigator / trial site and of the sponsor with regard to publication of the results of this trial are described in the Investigator contract / trial site's contract. As a general rule, no trial results should be published prior to finalisation of the Clinical Trial Report.

The certificate of insurance cover is made available to the Investigator and the patients, and is stored in the ISF (Investigator Site File).

# 8.1 TRIAL APPROVAL, PATIENT INFORMATION, INFORMED CONSENT

This trial will be initiated only after all required legal documentation has been reviewed and approved by the respective Institutional Review Board (IRB) / Independent Ethics Committee (IEC) and competent authority (CA) according to national and international regulations. The same applies for the implementation of changes introduced by amendments.

Prior to patient participation in the trial, written informed consent must be obtained from each patient (or the patient's legally accepted representative) according to ICH / GCP and to the regulatory and legal requirements of the participating country. Each signature must be personally dated by each signatory and the informed consent and any additional patient-information form retained by the Investigator as part of the trial records. A signed copy of the informed consent and any additional patient information must be given to each patient or the patient's legally accepted representative."

Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

For Japan only: The Investigator must give a full explanation to trial patients based on the patient information form. A language understandable to the patient should be chosen, technical terms and expressions avoided, if possible. The patient must be given sufficient time to consider participation in the trial. The Investigator obtains written consent of the patient's own free will with the informed consent form after confirming that the patient understands the contents.

For Japan only: The Investigator must sign (or place a seal on) and date the informed consent form. If a trial collaborator has given a supplementary explanation, the trial collaborator also signs (or places a seal on) and dates the informed consent.

Re-consenting may become necessary when new relevant information becomes available and should be conducted according to the sponsor's instructions.

The consent and re-consenting process should be properly documented in the source documentation.

# 8.2 DATA QUALITY ASSURANCE

A quality assurance audit/inspection of this trial may be conducted by the sponsor, sponsor's designees, or by IRB / IEC or by regulatory authorities. The quality assurance auditor will have access to all medical records, the Investigator's trial-related files and correspondence, and the informed consent documentation of this clinical trial.

### 8.3 RECORDS

Case Report Forms (CRF) for individual patients will be provided by the sponsor. See <u>Section 4.1.5.2</u> for rules about emergency code breaks. For drug accountability, refer to <u>Section 4.1.8</u>.

#### **8.3.1** Source documents

If defined in the protocol, additional records may need to be requested from the Investigator, e.g. information from any referral physicians on patient history relevant for AE reporting or data required in connection with outcome event collection in outcome studies.

In accordance with regulatory requirements the Investigator should prepare and maintain adequate and accurate source documents and trial records that include all observations and other data pertinent to the investigation on each trial subject. Source data as well as reported data should follow good documentation practices and be attributable, legible, contemporaneous, original and accurate. Changes to the data should be traceable (audit trail).

Data reported on the CRF must be consistent with the source data or the discrepancies must be explained.

The current medical history of the subject may not be sufficient to confirm eligibility for the trial and the Investigator may need to request previous medical histories and evidence of any diagnostic tests. In this case the Investigator must make three documented attempts to retrieve previous medical records. If this fails a verbal history from the patient, documented in their medical records, would be acceptable.

Trial Protocol


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Before providing any copy of patients' source documents to the sponsor the investigator must ensure that all patient identifiers (e.g. patient's name, initials, address, phone number, social security number) have properly been removed or redacted to ensure patient confidentiality.

If the patient is not compliant with the protocol, any corrective action e.g. re-training must be documented in the patient file.

For the CRF, data must be derived from source documents, for example:

- \* Patient identification: gender, date or year of birth (in accordance with local laws and regulations)
- Patient participation in the trial (substance, trial number, patient number, date patient was informed)
- \* Dates of Patient's visits, including dispensing of trial medication
- Medical history (including trial indication and concomitant diseases, if applicable)
- \* Medication history
- \* Adverse events and outcome events (onset date (mandatory), and end date (if available))
- \* Serious adverse events (onset date (mandatory), and end date (if available))
- \* Concomitant therapy (start date, changes)
- \* Originals or copies of laboratory results and other imaging or testing results, with proper documented medical evaluation (in validated electronic format, if available)
- \* Completion of Patient's Participation in the trial" (end date; in case of premature discontinuation document the reason for it).
- \* Prior to allocation of a patient to a treatment into a clinical trial, there must be documented evidence in the source data (e.g. medical records) that the trial participant meets all inclusion criteria and does not meet any exclusion criteria. The absence of records (either medical records, verbal documented feedback of the patient or testing conducted specific for a protocol) to support inclusion/exclusion criteria does not make the patient eligible for the clinical trial.

### 8.3.2 Direct access to source data and documents

The sponsor will monitor the conduct of the trial by regular on-site monitoring visits and inhouse data quality review. The frequency of on-site monitoring will be determined by assessing all characteristics of the trial, including its nature, objective, methodology and the degree of any deviations of the intervention from normal clinical practice.

The Investigator /institution will allow on-site trial-related monitoring, audits, IRB / IEC review and regulatory inspections. Direct access must be provided to the CRF and all source documents/data, including progress notes, copies of laboratory and medical test results, which must be available at all times for review by the CRA, auditor and regulatory inspector (e.g. FDA). The CRA and auditor may review all CRFs and informed consents. The accuracy of the data will be verified by direct comparison with the source documents described in Section 8.3.1. The sponsor will also monitor compliance with the protocol and ICH GCP.

**Trial Protocol** 


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 8.3.3 Storage period of records

### Trial site(s):

The trial site(s) must retain the source and essential documents (including ISF) according to the national or local requirements (whatever is longer) valid at the time of the end of the trial. Sponsor:

The sponsor must retain the essential documents according to the sponsor's SOPs.

### 8.4 EXPEDITED REPORTING OF ADVERSE EVENTS

BI is responsible to fulfil their legal regulatory reporting obligation and in accordance with the requirements. Any exemptions from expedited reporting are described under <u>Section</u> 5.3.6.2 and <u>Section</u> 5.3.6.3.

### 8.5 STATEMENT OF CONFIDENTIALITY AND PATIENT PRIVACY

The rights of the trial patient to privacy and protection of the data / patient notes obtained during the trial have to be ensured in accordance with local laws and regulations. Procedures for data handling and data protection need to be described in the patient information and informed consent form. Individual patient data obtained as a result of this trial is considered confidential and disclosure to third parties is prohibited with the exceptions noted below. Patient privacy will be ensured by using patient identification code numbers. Data protection and data security measures are implemented for the collection, storage and processing of patient data in accordance with the principles 6 and 12 of the WHO GCP handbook.

Treatment data may be given to the patient's personal physician or to other appropriate medical personnel responsible for the patient's welfare. Data generated as a result of the trial need to be available for inspection on request by the participating physicians, the sponsor's representatives, by the IRB / IEC and the regulatory authorities.

# 8.5.1 Collection, storage and future use of biological samples and corresponding data

Measures are in place to comply with the applicable rules for the collection, storage and future use of biological samples from clinical trial participants and the corresponding data, in particular

- \* A Quality Management System has been implemented to ensure the adherence with the Principles of Good Clinical Practice as outlined in 'Note For Guidance On Good Clinical Practice' (CPMP/ICH/13 5/95)
- The BI-internal facilities storing and analysing biological samples and data from clinical trial participants as well as the laboratories' activities for clinical trials sponsored by Boehringer Ingelheim are regularly audited. The analytical groups and the banking facility are therefore assessed to be qualified for the storage and use of biological samples and data collected in clinical trials.
- Samples and data are used only if an appropriate informed consent is available.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 8.6 TRIAL MILESTONES

The **start of the trial** is defined as the date of the enrolment (screening) of the first patient in the whole trial.

The **end of the trial** is defined as the date when the last patient in the whole trial completes the trial as per definition of trial completion in <u>Section 6.2.3.3</u>.

The "last-patient-last-visit-primary-endpoint-dose-finding" is defined as the date when all patients in a respective dose finding cohort have completed at least the first treatment course. Thus, this milestone is defined for each dose finding cohorts (A, B, C and D (dose finding)).

The "last-patient-last-visit-primary-endpoint-expansion" (Cohorts E and F) is defined as the date when all patients in a respective expansion cohort have completed at least two tumour assessment time points or have permanently discontinued treatment or have completed the trial according to <u>Section 6.2.3</u>. Thus, this milestone is defined for each expansion cohorts (E and F).

The "last-patient-last-visit-primary-endpoint-expansion" (Cohorts D1 and D2) is defined as the date when all patients have completed 18 months PFS observation or have permanently discontinued treatment or have completed the trial according to <u>Section 6.2.3</u>. Thus, this milestone is defined for Cohorts D1 and D2.

The "Last Patient Drug Discontinuation" (LPDD) date is defined as the date on which the last patient at an individual trial site ends trial medication (as scheduled per protocol or prematurely). Individual Investigators will be notified of SUSARs occurring with the trial medication until 30 days after LPDD at their site. Early termination of the trial is defined as the premature termination of the trial due to any reason before the end of the trial as specified in this protocol.

**Temporary halt of the trial** is defined as any unplanned interruption of the trial by the sponsor with the intention to resume it.

**Suspension of the trial** is defined as an interruption of the trial based on a Health Authority request.

The IEC / competent authority in each participating EU member state will be notified about the trial milestones according to the respective laws.

A final report of the clinical trial data will be written only after all patients have completed the trial in all countries (EU or non-EU) to incorporate and consider all data in the report.

The sponsor will submit to the EU database a summary of the final trial results within one year from the end of a clinical trial as a whole, regardless of the country of the last patient (EU or non-EU).

For Japan only: when the trial is completed, the Investigator should inform the head of the trial site of the completion in writing, and the head of the trial site should promptly inform the IRB and sponsor of the completion in writing.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 8.7 PROTOCOL VIOLATIONS

For Japan only: the Investigator should document any deviation from the protocol regardless of their reasons. Only when the protocol was not followed in order to avoid an immediate hazard to trial subjects or for other medically compelling reason, the principal Investigator should prepare and submit the records explaining the reasons thereof to the sponsor, and retain a copy of the records.

# 8.8 COMPENSATION AVAILABLE TO THE PATIENT IN THE EVENT OF TRIAL RELATED INJURY

For Japan only: in the event of health injury associated with this trial, the sponsor is responsible for compensation based on the contract signed by the trial site.

c09049566-10 
 09049566-10
 Trial Protocol
 

 Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9. **REFERENCES**

| 9.1 | PURLISHED | REFERENCES |
|-----|-----------|------------|

| P15-00363 | King H, Aleksic T, Haluska P, Macaulay VM. Can we unlock the potential of IGF-1R inhibition in cancer therapy? Cancer Treat Rev 40 (9), 1096 – |
|---|---|
| P15-10237 | 1105 (2014) Boolell V, Alamgeer M, Watkins DN, Ganju V. The evolution of therapies in non-small cell lung cancer. Cancers 7 (3), 1815 – 1846 (2015) |
| P15-10395 | Iams WT, Lovly CM. Molecular pathways: clinical applications and future direction of insulin-like growth factor-1 receptor pathway blockade. Clin Cancer Res 21 (19), 4270 – 4277 (2015) |
| P16-09570 | Cortes J, Martinez N, Sablin MP, Perez-Fidalgo JA, Neven P, Hedayati E, et al |
| | Phase Ib/II trial of xentuzumab, an insulin-like growth factor ligand-<br>neutralizing antibody, combined with exemestane and everolimus in<br>hormone receptor-positive locally advanced or metastatic breast cancer:<br>primary phase Ib results. 52nd Ann Mtg of the American Society of Clinical |
| P1 6 00 555 | Oncology (ASCO), Chicago, 3 - 7 Jun 2016 (Poster) |
| P16-09577 | Rocco G, Morabito A, Leone A, Muto P, Fiore F, Budillon A. Management of non-small cell lung cancer in the era of personalized medicine. Int J Biochem Cell Biol 78, 173 - 179 (2016) |
| R07-4856 | European Medicines Agency (EMEA). Committee for Medicinal Products for Human Use (CHMP): guideline on clinical trials in small populations (London, 27 July 2006, doc. ref. CHMP/EWP/83561/2005). London: EMEA (2006) |
| R09-0262 | Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D et al., New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer 2009;45:228-247. |
| R10-4848 | Common Terminology Criteria for Adverse Events (CTCAE): version 4.0 (NIH publication no. 09-5410, published: May 28, 2009 (v4.03: June 14, 2010), revised June 2010, reprinted June 2010). |
| | http://evs.nci.nih.gov/ftp1/CTCAE/CTCAE_4.03_2010-06-14 QuickReference 8.5x11.pdf (2010) |
| R10-5355 | Samani AA, Yakar S, LeRoith D, Brodt P. The role of the IGF system in cancer growth and metastasis: Overview and recent insights. Endocr Rev 28 (1), 20 – 47 (2007) |
| R10-5694 | Souza AT de, Hankins GR, Washington MK, Orton TC, Jirtle RI. M6P/IGF2R gene is mutated in human hepatocellular carcinomas with loss of heterozygosity. Nature Genet 11, 447 – 449 (1995) |
| R12-2864 | Siegel R, Naishadham D, Jemal A. Cancer statistics, 2012. CA 62 (1), 10 – 29 (2012) |
| R12-4524 | Pollak M. The insulin and insulin-like growth factor receptor family in neoplasia: an update. Nat Rev Cancer 12, 159 – 169 (2012) |
| R12-5635 | Baselga J, et al. Everolimus in postmenopausal hormone-receptor-positive advanced breast cancer. N Engl J Med 366 (6), 520 - 529 (2012) |

c09049566-10 Trial Protocol 

| Proprietary confid | ential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|---|
| R13-1229 | Scher HI, et al, AFFIRM Investigators. Increased survival with |
| | enzalutamide in prostate cancer after chemotherapy. N Engl J Med 367 |
| | (13), 1187 - 1197 (2012) |
| R13-4802 | Jaki T, Clive S, Weir CJ. Principles of dose finding studies in cancer: a |
| K15 1002 | comparison of trial designs. Cancer Chemother Pharmacol 71, 1107 - 1114 |
| D12 4002 | (2013) |
| R13-4803 | Neuenschwander B, Branson M, Gsponer T. Critical aspects of the |
| | Bayesian approach to phase I cancer trials. Stat Med 27, 2420 - 2439 (2008) |
| R13-4804 | Rogatko A, Schoeneck D, Jonas W, Tighiouart M, Khuri FR, Porter A. |
| | Translation of innovative designs into phase I trials. J Clin Oncol 25 (31), |
| | 4982 - 4986 (2007) |
| R13-4805 | Tourneau C le, Gan HK, Razak ARA, Paoletti X. Efficiency of new dose |
| 1110 .000 | escalation designs in dose-finding phase I trials of molecularly targeted |
| | agents. Plos One 7 (12), e51039 (2012) |
| D14 1645 | • , , , , , |
| R14-1645 | Murtaza M, Dawson SJ, Tsui DWY, Gale D, Forshew T, Piskorz AM, |
| | Parkinson C, Chin SF, Kingsbury Z, Wong ASC, Marass F, Humphray S, |
| | Hadfield J, Bentley D, Chin TM, Brenton JD, Caldas C, Rosenfeld N |
| | Non-invasive analysis of acquired resistance to cancer therapy by |
| | sequencing of plasma DNA. |
| | Nature 497, 108 - 112 (2013) |
| R15-1307 | Beer TM, et al, PREVAIL Investigators. Enzalutamide in metastatic |
| | prostate cancer before chemotherapy. N Engl J Med 371 (5), 424 - 433 |
| | (2014) |
| R15-4233 | Zhao W, Yang H, editors. Statistical methods in drug combination studies. |
| 10 1200 | (CRC Biostatistics Series) Boca Raton: CRC Press (2015) |
| R16-0844 | Heilmann AM, Perera RM, Ecker V, Nicolay BN, Bardeesy N, Benes CH, |
| K10-00 <del>11</del> | Dyson NJ. CDK4/6 and IGF1 receptor inhibitors synergize to suppress the |
| | growth of p 16INK4A-deficient pancreatic cancers. Cancer Res 74 (14), 39- |
| | 47-3958 (2014). |
| R16-0845 | Miller ML, Molinelli EJ, Nair JS, Sheikh T, Samy R, Jing X, He Q, Korkut |
| | A, Crago AM, Singer S, Schwartz GK, Sander C. Drug synergy screen and |
| | network modelling in dedifferentiated liposarcoma identifies CDK4 and |
| | IGF1R as synergistic drug targets. Sci Signal 6 (294), ra85 (2013) |
| R16-2249 | Sherr CJ, Beach D, Shapiro GI. Targeting CDK4 and CDK6: from |
| 1110 == 1,7 | discovery to therapy. Cancer Discov 6, 353 - 367 (2016) |
| R16-2270 | Challenge and opportunity on the critical path to new medical products |
| 10-2270 | (page last updated: 01/25/2016, this report replaces the version posted on |
| | March 16, 2004). |
| | http://www.fda.gov/downloads/ScienceResearch/SpecialTopics/CriticalPath |
| | Initiative/CriticalPathOpportunitiesReports/ucm113411.pdf (access date: 18 |
| | May 2016); U.S. Department of Health and Human Services, Food and |
| | Drug Administration (2016) |
| R16-3704 | O'Leary B, Finn RS, Turner NC. Treating cancer with selective CDK4/6 |
| | inhibitors. Nat Rev Clin Oncol 13 (7), 417 - 430 (2016) |
| R16-3978 | Velasco-Velazquez MA, Li Z, Casimiro M, Loro E, Homsi N, Pestell RG. |
| | Examining the role of cyclin D1 in breast cancer. Future Oncol 7 (6), 753 - |
| | 765 (2011) |
| | 103 (2011) |

Boehringer Ingelheim BI Trial No.: 1280.18

c09049566-10 Trial Protocol 

| Proprietary confi | dential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|---|
| R16-3979 | VanArsdale T, Boshoff C, Arndt KT, Abraham RT. Molecular pathways: targeting the cyclin cancer research D-CDK4/6 axis for cancer treatment. |
| R16-3980 | Clin Cancer Res 21 (13), 2905 - 2910 (2015)<br>Kumar M, Ernani V, Owonikoko TK. Biomarkers and targeted systemic<br>therapies in advanced non-small cell lung cancer. Mol Aspects Med 45, 55 -<br>66 (2015) |
| R16-3981 | Hou X, Huang F, Macedo L, Harrington SC, Reeves KA, Greer A, et al Dual IGF-1R/InsR inhibitor BMS-754807 synergizes with hormonal agents in treatment of estrogen-dependent breast cancer. Cancer Res 71 (24), 7597 - 7607 (2011) |
| R16-3982 | Patnaik A, Rosen LS, Tolaney SM, Tolcher AW, Goldman JW, Gandhi L, et al Efficacy and safety of abemaciclib, an inhibitor of CDK4 and CDK6, for patients with breast cancer, non-small cell lung cancer, and other solid tumors. Cancer Discov 6 (7), 740 - 753 (2016) |
| R16-3983 | Cardoso F, Costa A, Norton L, Cameron D, Cufer T, Fallowfield L, et al. 1st international consensus guidelines for advanced breast cancer (ABC 1). Breast 21, 242 - 252 (2012) |
| R16-5327 | Dickler MN, Tolaney SM, Rugo HS, Cortés J, Diéras V, Patt D, Wildiers H, Frenzel M, Koustenis A, Baselga J. Monarch 1: results from a phase 2 study of abemaciclib, a CDK4 and CDK6 inhibitor, as monotherapy, in patients with HR+/HER2- breast cancer, after chemotherapy for metastatic disease. 52nd Ann Mtg of the American Society of Clinical Oncology (ASCO), Chicago, 3 - 7 Jun 2016 |
| R17-2796 | Sledge GW, Toi M, Neven P, Sohn J, Inoue K, Pivot X, et al. MONARCH 2: abemaciclib in combination with fulvestrant in women with HR+/HER2-advanced breast cancer who had progressed while receiving endocrine therapy. Journal of Clinical Oncology, Published online: 3 June 2017 |
| R18-2693 | FDA approves abemaciclib for HR-positive, HER2-negative breast cancer. https://www.fda.gov/Drugs/InformationOnDrugs/ApprovedDrugs/ucm5780 81.htm (access date: 23 August 2018); Silver Spring: U.S. Food and Drug Administration (2017) |
| 9.2 | UNPUBLISHED REFERENCES |
| c01690707-08 | Investigator's Brochure Xentuzumab (BI 836845) oncology, 1280.P1/P2/P3, 26-Jul-2018, Version 11 |
| c26540383 | Investigator's Brochure Abemaciclib LY2835219 07-Dec-2018 |
| c22665932-01 | 1280.4 Subgroup Analysis Report,<br>Version 1.0 dated 10 August 2018 |

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 10. APPENDICES

### 10.1 INDUCERS AND STRONG INHIBITORS OF CYP3A4

The information in this table is provided for guidance to investigators and does not preclude the use of these medications if clinically indicated.

### Strong Inducers of CYP3A

Carbamazepine

Dexamethasonea

Phenobarbital/phenobarbitone

Phenytoin

Rifapentine

Rifampin

Rifabutin

St John's wort

#### **Moderate Inducers of CYP3A**

Bosentan

Lenisurad

Modafinil

Primidone

Telotristat ethyl

### Strong Inhibitors of CYP3A

Aprepitant

Ciprofloxacin

Clarithromycin

Conivaptan

Diltiazem

Erythromycin

Fluconazole

Itraconazole

Ketoconazole

Nefazodone

Posaconazole

Troleandomycin

Verapamil

<sup>&</sup>lt;sup>a</sup> Important note: All patients may receive supportive therapy with dexamethasone, preferably ≤7 days, if clinically indicated.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 10.2 PHARMACOKINETICS PLAN

# 10.2.1 FLOW CHART for PK, immunogenicity, and biomarkers for cohorts A, B, C, and D (dose finding)

10.2.1.1 Flowchart for PK, immunogenicity, and biomarkers for Cohorts A, B, C, and D (dose finding) in treatment course 1

| Course | Visit | Day | Planned time<br>[h:min] | Event and comment | Xentuzumab PK | ADA | Total IGF-1/2, IGFBP-3 | Free /dissociable IGF-1/2 | pIGF-1R/IGF-1R in PRP |
|---|---|---|---|---|---|---|---|---|---|
| SCR | SCR | Within 28d<br>before C1V1 | -999:00* | Sampling at screening visit | | | | | X |
| 1 | 1 | 1 | -0:05 | Blood sampling prior to xentuzumab infusion | X | X | X | X | X |
| | | | 0:00 | Start of xentuzumab infusion | | | | | |
| | | | 1:00** | Immediately at the end of xentuzumab infusion | X | | | | |
| | 2 | 8 | 168:00 | Blood sampling ~5 minutes prior to xentuzumab infusion | X | X | | | X |

<sup>\*</sup>Planned time listed at visit SCR is considered to be a dummy planned time to set-up the database, the description in column "Day" defines the timing for these specific samples

<sup>\*\*</sup> If the infusion duration is different from 1h, please adapt the sampling time accordingly.

c09049566-10  Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

FLOW CHART for PK, immunogenicity, and biomarkers for cohorts A, B, C, 10.2.1.2 and D (dose finding) in courses 2-12, 15, and 18, EOTV and FU

| Course | Visit | Day | Planned time<br>[h:min] | Event and comment | Xentuzumab PK | ADA | Total IGF-1/2, IGFBP-3 | Free /dissociable IGF-1/2 | pIGF-1R/IGF-1R in PRP |
|---|---|---|---|---|---|---|---|---|---|
| 2-12,<br>15, 18 | 1 | 1 | -0:05 | Blood sampling prior to xentuzumab infusion | X | X | X | X | X |
| | | | 0:00 | Start of xentuzumab infusion | | | | | |
| | | | 1:00** | Immediately at the end of xentuzumab infusion | X | | | | |
| EOT<br>V | EOTV | Within 7d after last drug intake | 998:00* | End of treatment visit | X | X | X | X | X |
| FU | FU | 42 +7d after last<br>drug intake | 999:00* | Follow-up | X | X | X | X | X |

<sup>\*</sup>Planned times listed at visit EOTV and FU are considered to be dummy planned times to set-up the database, the description in column "Day" defines the timing for these specific samples

<sup>\*\*</sup> If the infusion duration is different from 1h, please adapt the sampling time accordingly.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 10.2.2 FLOW CHART for PK, immunogenicity, and biomarkers for cohort E

10.2.2.1 FLOW CHART for PK, immunogenicity, and biomarkers for cohort E in Run-in phase and treatment course 1

| Course | Visit | Day | Planned time<br>[h:min] | Event and comment | Xentuzumab PK | ADA | Abemaciclib and metabolites PK*** | Total IGF-1/2,<br>IGFBP-3 | Free /dissociable<br>IGF-1/2 | pIGF-1R/IGF-1R in<br>PRP |
|---|---|---|---|---|---|---|---|---|---|---|
| SCR | SCR | Within 28d<br>before Run<br>in V1 | -999:00* | Sampling at screening visit | | | | | | X |
| Run<br>in | 1 | -9 | -192:05 | 5 minutes prior to first abemaciclib treatment | X | X | X*** | X | X | X |
| | 3 | -1 | -0:05 | Blood sampling 5 minutes prior to abemaciclib administration | | | X*** | | | |
| | | | 0:00 | abemaciclib administration (morning dose) | | | | | | |
| | | | 1:00 | | | | X | | | |
| | | | 2:30 | | | | X | | | |
| | | | 4:00 | | | | X | | | |
| | | | 6:00 | | | | X | | | |
| | | | 8:00 | | | | X | | | |
| | | | 12:00<br>[± 2:00] | Blood sampling <b>before</b> intake of evening dose of abemaciclib | | | X | | | |
| 1 | 1 | 1 | -0:05 | Blood sampling prior to xentuzumab infusion and abemaciclib administration | X | X | X*** | X | X | X |
| | | | 0:00 | Start of xentuzumab infusion | | | | | | |
| | | | 0:01 | Abemaciclib administration | | | | | | |
| | | | 1:00** | Immediately at the end of xentuzumab infusion | X | | | | | |
| | 2 | 8 | 168:00 | Blood sampling prior to xentuzumab infusion | X | X | | | | X |

<sup>\*</sup>Planned time listed at visit SCR is considered to be a dummy planned time to set-up the database, the description in column "Day" defines the timing for these specific samples

<sup>\*\*</sup> If the infusion duration is different from 1h, please adapt the sampling time accordingly.

<sup>\*\*\*</sup> At days of abemaciclib PK sampling, patients have to take their morning dose of abemaciclib in the hospital in order to allow exact timing of PK sampling

c09049566-10


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 10.2.2.2 FLOW CHART for PK, immunogenicity, and biomarkers for cohort E in treatment course 2

| Course | Visit | Day | Planned time<br>[h:min] | Event and comment | Xentuzumab PK | ADA | Abemaciclib and metabolites PK*** | Total IGF-1/2, IGFBP-3 | Free dissociable IGF-1/2 | pIGF-1R/IGF-1R in PRP |
|---|---|---|---|---|---|---|---|---|---|---|
| 2 | 1 | 1 | -0:05 | Blood sampling prior to abemaciclib and xentuzumab administration | X | X | X*** | X | X | X |
| | | | 0:00 | Start of xentuzumab infusion | | | | | | |
| | | | 0:01 | Abemaciclib administration | | | | | | |
| | | | 1:00** | Immediately at the end of xentuzumab infusion | X | | X | | | |
| | | | 2:30 | | X | | X | | | |
| | | | 4:00 | | X | | X | | | |
| | | | 6:00 | | X | | X | | | |
| | | | 8:00 | | X | | X | | | |
| | | | 12:00<br>[± 2:00] | Blood sampling <b>before</b> intake of evening dose of abemaciclib | X | | X | | | |
| | 1 | 2 | 23:55 | Blood sampling prior to abemaciclib administration | X | | | | | |
| | | | 24:00 | Abemaciclib administration | | | | | | |
| | 1b | 4±1 | 72:00 | Blood sampling at this visit | X | | | | | |
| | 2 | 8±1 | 168:00 | Blood sampling ~ 5 min prior to abemaciclib administration and xentuzumab infusion | X | | | | | |

<sup>\*\*</sup> If the infusion duration is different from 1h, please adapt the sampling time accordingly.

<sup>\*\*\*</sup> At days of abemaciclib PK sampling, patients have to take their morning dose of abemaciclib in the hospital in order to allow exact timing of PK sampling

**Trial Protocol** 

c09049566-10  Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 10.2.2.3 FLOW CHART for PK, immunogenicity, and biomarkers for cohort E in treatment courses 3-12, 15, 18 and EOTV and FU visit

| Course | Visit | Day | Planned Time<br>[h:min] | Event and comment | Xentuzumab PK | ADA | Abemaciclib and metabolites PK | Total IGF-1/2, IGFBP-3 | Free /dissociable IGF-1/2 | pIGF-1R/IGF-1R in PRP |
|---|---|---|---|---|---|---|---|---|---|---|
| 3-12,<br>15, 18 | 1 | 1 | -0:05 | Blood sampling prior to abemaciclib administration and xentuzumab infusion | X | X | | X | X | X |
| | | | 0:00 | Start of xentuzumab infusion | | | | | | |
| | | | 0:01 | Abemaciclib administration | | | | | | |
| | | | 1:00** | Immediately at the end of xentuzumab infusion | X | | | | | |
| EOTV | EOTV | Within 7d<br>after last<br>drug<br>intake | 998:00* | End of treatment visit | X | X | | X | X | X |
| FU | FU | 42 +7d<br>after last<br>drug<br>intake | 999:00* | Follow-up | X | X | | X | X | X |

<sup>\*</sup>Planned times listed at visit EOTV and FU are considered to be dummy planned times to set-up the database, the description in column "Day" defines the timing for these specific samples

<sup>\*\*</sup> If the infusion duration is different from 1h, please adapt the sampling time accordingly.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 10.2.3 FLOW CHART for PK, immunogenicity, and biomarkers for cohort F

# As of 22 Oct 2021, samples for PK, immunogenicity and biomarkers are no longer collected for ongoing patients.

10.2.3.1 FLOW CHART for PK, immunogenicity, and biomarkers for cohort F in screening and treatment course 1

| Course | Visit | Day | Planned time<br>[h:min] | Event and comment | Xentuzumab PK | ADA | Abemaciclib and metabolites PK*** | Total IGF-1/2,<br>IGFBP-3 | Free /dissociable | pIGF-1R/IGF-1R |
|---|---|---|---|---|---|---|---|---|---|---|
| SCR | SCR | Within 28d<br>before Run | -999:00 | Sampling at screening visit | | | | | | X |
| | | in V1 | 0.05 | 71 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | | | | | | |
| 1 | 1 | 1 | -0:05 | Blood sampling prior to abemaciclib administration, xentuzumab infusion and fulvestrant injection | X | X | X*** | X | X | X |
| | | | 0:00 | Start of xentuzumab infusion | | | | | | |
| | | | 0:01 | Abemaciclib administration | | | | | | |
| | | | 0:00 | Fulvestrant injection up to 15min. after start of xentuzumab infusion | | | | | | |
| | | | 1:00** | Immediately at the end of xentuzumab infusion | X | | | | | |
| | 2 | 8 | 168:00 | Blood sampling prior to xentuzumab infusion | X | X | | | | X |

<sup>\*</sup>Planned time listed at visit SCR is considered to be a dummy planned time to set-up the database, the description in column "Day" defines the timing for these specific samples

<sup>\*\*</sup> If the infusion duration is different from 1h, please adapt the sampling time accordingly.

<sup>\*\*\*</sup> At days of abemaciclib PK sampling, patients have to take their morning dose of abemaciclib in the hospital in order to allow exact timing of PK sampling

c09049566-10

Trial Protocol


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 10.2.3.2 FLOW CHART for PK, Immunogenicity, biomarkers for cohort F in treatment courses 2-12, 15, 18, EOTV and FU

| Course | Visit | Day | Planned time<br>[h:min] | Event and comment | Xentuzumab PK | ADA | Abemaciclib and metabolites PK | Fulvestrant PK | Total IGF-1/2, IGFBP-3 | Free /dissociable IGF-1/2 | pIGF-1R/IGF-1R in PRP |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 2-12,<br>15, 18 | 1 | 1 | -0:05 | Blood sampling prior to abemaciclib administration, xentuzumab infusion and fulvestrant injection | X | X | X <sup>1</sup><br>*** | $X^1$ | X | X | X |
| | | | 0:00 | Start of xentuzumab infusion Abemaciclib administration | | | | | | | |
| | | | 0:00 | Fulvestrant injection up to 15min. after start of xentuzumab infusion | | | | | | | |
| | | | 1:00** | Immediately at the end of xentuzumab infusion | X | | | | | | |
| EOTV | EOTV | Within 7d<br>after last<br>drug<br>intake | 998:00* | End of treatment visit | X | X | | | X | X | X |
| FU | FU | 42 +7d<br>after last<br>drug<br>intake | 999:00* | Follow-up | X | X | | | X | X | X |

<sup>\*</sup>Planned times listed at visit EOTV and FU are considered to be dummy planned times to set-up the database, the description in column "Day" defines the timing for these specific samples

<sup>\*\*</sup> If the infusion duration is different from 1h, please adapt the sampling time accordingly.

<sup>\*\*\*</sup> At days of abemaciclib PK sampling, patients have to take their morning dose of abemaciclib in the hospital in order to allow exact timing of PK sampling

<sup>&</sup>lt;sup>1</sup> this sample needs to be collected in course 2 and 3 only

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 10.2.4 FLOW CHART for PK, immunogenicity, and biomarkers for cohorts D1 and D2

# As of 22 Oct 2021, samples for PK, immunogenicity and biomarkers are no longer collected for ongoing patients.

10.2.4.1 FLOW CHART for PK, immunogenicity, and biomarkers for cohorts D1 and D2 in treatment course 1

| | | | atiliciti co | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Course | Visit | Day | Planned time<br>[h:min] | Event and comment | Xentuzumab PK | ADA | Abemaciclib and<br>metabolites PK | Total IGF-1/2,<br>IGFBP-3 | Free /dissociable | pIGF-1R/IGF-1R |
| SCR | SCR | Within 28d<br>before<br>C1V1 | -999:00* | Sampling at screening visit | | | | | | X |
| 1 | 1 | 1 | -0:05 | Blood sampling prior to abemaciclib administration, xentuzumab infusion and fulvestrant injection | X | X | | X | X | X |
| | | | 0:00 | Start of xentuzumab infusion | | | | | | |
| | | | 0:01 | Abemaciclib administration | | | | | | |
| | | | 0:00 | Fulvestrant injection up to 15min. after start of xentuzumab infusion | | | | | | |
| | | | 1:00** | Immediately at the end of xentuzumab infusion | X | | | | | |
| | 2 | 8 | 168:00 | Blood sampling prior to xentuzumab infusion | X | X | | | | X |
| | 3 | 15 | 336:00 | Blood sampling prior to xentuzumab infusion | X | | | | | |
| | 4 | 22 | 504:00 | Blood sampling prior to xentuzumab infusion | X | | | | | |

<sup>\*</sup>Planned time listed at visit SCR is considered to be a dummy planned time to set-up the database, the description in column "Day" defines the timing for these specific samples

<sup>\*\*</sup> If the infusion duration is different from 1h, please adapt the sampling time accordingly.


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 10.2.4.2 FLOW CHART for PK, immunogenicity, and biomarkers for cohorts D1 and D2 in treatment course 2

| Course | Visit | Day | Planned time<br>[h:min] | Event and comment | Xentuzumab PK | ADA | Abemaciclib and<br>metabolites PK*** | Fulvestrant PK | Total IGF-1/2, IGFBP-3 | Free / dissociable IGF-1/2 | pIGF-1R/IGF-1R in PRP |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 2 | 1 | 1 | -0:05 | Blood sampling prior to<br>abemaciclib administration,<br>xentuzumab infusion and<br>fulvestrant injection | X | X | X*** | X | X | X | X |
| | | | 0:00 | Start of xentuzumab infusion | | | | | | | |
| | | | 0:01 | Abemaciclib administration | | | | | | | |
| | | | 0:00 | Fulvestrant injection up to 15min. after start of xentuzumab infusion | | | | | | | |
| | | | 1:00** | Immediately at the end of xentuzumab infusion | X | | $X^1$ | $X^1$ | | | |
| | | | 2:30 | | $X^1$ | | $X^1$ | | | | |
| | | | 4:00 | | $X^1$ | | $X^1$ | | | | |
| | | | 6:00 | | $X^1$ | | $X^1$ | | | | |
| | | | 8:00 | | $X^1$ | | $X^1$ | | | | |
| | | | 12:00<br>[± 2:00] | Blood sampling ~5 minutes <b>before</b> intake of evening dose of abemaciclib | X <sup>1</sup> | | $X^1$ | X <sup>1</sup> | | | |
| | 1 | 2 | 23:55 | | $X^1$ | | | $X^1$ | | | |
| | | | 24:00 | Abemaciclib administration | | | | | | | |
| | 1b | 4 | 72:00 | Blood sampling prior to abemaciclib administration | $X^1$ | | | $X^1$ | | | |
| | 2 | 8 | 168:00 | Blood sampling prior to xentuzumab infusion | $X^1$ | | | $X^1$ | | | |
| | 3 | 15 | 336:00 | Blood sampling prior to xentuzumab infusion | | | | X <sup>1</sup> | | | |
| | 4 | 22 | 504:00 | Blood sampling prior to xentuzumab infusion | | | | X <sup>1</sup> | | | |

<sup>\*\*</sup> If the infusion duration is different from 1h, please adapt the planned time accordingly.

<sup>\*\*\*</sup> At days of abemaciclib PK sampling, patients have to take their morning dose of abemaciclib in the hospital in order to allow exact timing of PK sampling

<sup>&</sup>lt;sup>1</sup> these PK samples will be collected for at least 15 subjects in cohort D1 and at least 15 subjects in cohort D2.

c09049566-10 Trial Protocol


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 10.2.4.3 FLOW CHART for PK, Immunogenicity, biomarkers for cohorts D1 and D2 in treatment courses 3, 4, 6, 12, 24, EOTV and FU

| Course | Visit | Day | Planned time<br>[h:min] | Event and comment | Xentuzumab PK | ADA | Abemaciclib and metabolites PK | Fulvestrant PK | Total IGF-1/2, IGFBP-3 | Free /dissociable IGF-1/2 | pIGF-1R/IGF-1R in PRP |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 3, 4, 6,<br>12, 24 | 1 | 1 | -0:05 | Blood sampling prior to abemaciclib administration, xentuzumab infusion and fulvestrant injection | X | X | $X^1$ | $X^1$ | $X^2$ | $X^2$ | X |
| | | | 0:00 | Start of xentuzumab infusion | | | | | | | |
| EOTV | EOTV | Within 7d<br>after last<br>drug<br>intake | 998:00* | End of treatment visit | X | X | | | X | X | X |
| FU | FU | 42 +7d<br>after last<br>drug<br>intake | 999:00* | Follow-up | X | X | | | X | X | X |

<sup>\*</sup>Planned times listed at visit EOTV and FU are considered to be dummy planned times to set-up the database, the description in column "Day" defines the timing for these specific samples

<sup>&</sup>lt;sup>1</sup> this sample needs to be collected in course 3 and course 4 only

<sup>&</sup>lt;sup>2</sup> this sample needs to be collected in course 3, course 4, and course 6 only

09049566-10 Trial Protocol 
Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies c09049566-10

#### TUMOUR TISSUE SAMPLE REQUIREMENTS 10.3

| Marker | Tissue | Amount of tissue | Time point of | Analysis type |
|---|---|---|---|---|
| category | type | | sample taking | |
| PGx | FFPE | Preferably FFPE | screening | RNA expression |
| | (RNase- | tumour tissue block | | |
| | free) | for preparation of | | |
| | | 8x 5μm sections | | |
| PGx/Protein | FFPE | Preferably FFPE | screening | DNA isolation + |
| Biomarkers | | tumour tissue block | | mutational/CNA |
| | | for preparation of | | analysis and |
| | | 17x 5μm sections | | biochemical protein |
| | | | | analysis (e.g. IHC) |

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 10.4 TUMOUR RESPONSE ASSESSMENT ACCORDING TO RECIST 1.1

# Response criteria for target lesions

| 1. Complete Response (CR): | Disappearance of all target lesions. Any pathological |
|---|---|
| | lymph nodes (whether target or non-target) must have a |
| | reduction in short axis to <10mm) |
| 2. Partial Response (PR): | At least a 30% decrease in the sum of diameters of |
| | target lesions taking as reference the baseline sum |
| | diameters |
| 3. Progression (PD): | At least a 20% increase in the sum of diameters of |
| | target lesions, taking as references the smallest sum on |
| | study (this includes the baseline sum if that is the |
| | smallest on study). In addition to the relative increase |
| | of 20%, the sum must also demonstrate an absolute |
| | increase of at least 5mm (note: the appearance of one or |
| | more new lesions is also considered progression). |
| 4. Stable Disease (SD): | Neither sufficient shrinkage to qualify for PR nor |
| | sufficient increase to qualify for PD, taking as |
| | references the smallest sum diameters while on study |

# Response criteria for non-target lesions

| 1. Complete Response (CR): | Disappearance of all non-target lesions and normalization of tumour marker level. All lymph nodes must be non-pathological in size (<10mm short axis) |
|---|---|
| 2. Non-CR/ Non-PD: | Persistence of one or more non-target lesion(s) or/and maintenance of tumour marker level above the normal limits |
| 3. Progression (PD): | Unequivocal progression of existing non-target lesions (Note: the appearance of one or more new lesions is also considered progression) |

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### Time point response for patients with measurable disease at baseline

| Target lesions | Non-Target lesions | New lesions | Overall |
|-------------------|-----------------------------|-------------|----------|
| | | | response |
| CR | CR | No | CR |
| CR | Non-CR/Non-PD | No | PR |
| CR | Not evaluated | No | PR |
| PR | Non-PD or not all evaluated | No | PR |
| SD | Non-PD or not all evaluated | No | SD |
| Not all evaluated | Non-PD | No | NE |
| PD | Any | Yes or No | PD |
| Any | PD | Yes or No | PD |
| Any | Any | Yes | PD |

Time point response for patients with non-measurable disease at baseline

| Non-target lesions | New lesions | Overall response |
|--------------------|-------------|------------------|
| CR | No | CR |
| Non-CR/ Non-PD | No | Non-CR/ Non-PD |
| Not all evaluated | No | NE |
| Unequivocal PD | Yes or No | PD |
| Any | Yes | PD |

### RECIST 1.1 is as published in Eur. J. Cancer <u>R09-0262</u>

Best overall response is evaluated from first treatment administration until the earliest of disease progression, death or last evaluable tumour assessment before start of subsequent anticancer therapy. When stable disease is believed to be best response, it must also meet a minimum time from first treatment administration of 48 days (i.e. according <u>Flow Chart</u>, the first post–baseline imaging should be performed within 63 days after start of xentuzumab). Note that clinical disease assessment will not be considered for determination of best overall response. No confirmation is required for best overall response
c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 10.5 CLINICAL EVALUATION OF LIVER INJURY

# 10.5.1 Introduction

Alterations of liver parameters, as described in <u>Section 5.3.6.1</u> (Protocol-Specified Adverse events of special interest), are to be further evaluated using the following procedures:

# 10.5.2 Procedures

Any elevation of ALT/AST and bilirubin qualifying as laboratory alert should be confirmed using the initial sample if possible.

If the alert is confirmed on initial sample, or it is not possible to repeat testing using initial sample, the following must be completed:

- 1) Evaluate patient within 48 hours and
- 2) Perform the following laboratory tests:
  - 1. Repeat of AST, ALT, bilirubin (with fractionation to total and direct)
  - 2. Haptoglobin
  - 3. Complete blood count and cell morphology
  - 4. Reticulocyte count
  - 5. Creatine Kinase (CK)
  - 6. Lactate dehydrogenase (LDH)
  - 7. Alkaline Phosphatase

The results of these laboratory tests must be reported to BI as soon as possible.

If the initial alert values (i.e. AST,ALT, and bilirubin) are confirmed on the second sample described as above, then an abdominal ultrasound or clinically appropriate alternate imaging (to rule out biliary tract, pancreatic or intrahepatic pathology, e.g. bile duct stones or neoplasm) must be completed within 48 hours.

The findings from the hepatic imaging (including comparison to prior imaging if available) must be made available as soon as possible as part of the adverse event reporting process. In the event the etiology of the abnormal liver tests results is not identified based on the imaging (e.g. biliary tract, pancreatic or intrahepatic pathology), then the "DILI checklist" must be completed. Details of the "DILI checklist" are provided in the ISF. The following assessments need to be performed in order to complete the "DILI checklist" and results will be reported via the eCRF:

obtain a detailed history of current symptoms and concurrent diagnoses and medical history according to the "DILI checklist" provided in the ISF;

obtain history of concomitant drug use (including non-prescription medications, herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets according to the "DILI checklist" provided in the ISF;

obtain a history of exposure to environmental chemical agents (consider home and work place exposure) according to the "DILI checklist" provided in the ISF;

complete the following laboratory tests as detailed in the DILI checklist provided in the ISF: Clinical chemistry c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Alkaline phosphatase, cholinesterase (serum)\*, albumin, PT or INR, CK, CK-MB, coeruloplasmin\*, α-1 antitrypsin\*, transferrin\*, amylase, lipase, fasting glucose, cholesterol, triglycerides

# Serology

Hepatitis A (Anti-IgM, Anti-IgG), Hepatitis B (HbsAg, Anti-HBs, DNA), Hepatitis C (Anti-HCV, RNA if Anti-HCV positive), Hepatitis D (Anti-IgM, Anti-IgG), Hepatitis E (Anti-HEV, Anti-HEV IgM, RNA if Anti-HEV IgM positive), Anti-Smooth Muscle antibody (titer), Anti-nuclear antibody (titer), Anti-LKM (liver-kidney microsomes) antibody, Anti-mitochondrial antibody, Epstein Barr Virus (VCA IgG, VCA IgM), cytomegalovirus (IgG, IgM), herpes simplex virus (IgG, IgM)\*, varicella (IgG, IgM)\*, parvovirus (IgG, IgM)\*

Hormones, tumour marker Thyroid-stimulating hormone (TSH)\*

Haematology Thrombocytes, eosinophils

\*If clinically indicated (e.g. immunocompromised patients)

# Long term follow-up

Initiate close observation of subjects by repeat testing of ALT, AST, and bilirubin (with fractionation to total and direct) at least weekly until the laboratory ALT and or AST abnormalities stabilize or return to normal, then according to the protocol. Depending on further laboratory changes, additional parameters identified e.g. by reflex testing will be followed up based on medical judgement and Good Clinical Practices (GCP). and report these via the eCRF.

# 10.6 STATISTICAL APPENDIX

A Bayesian logistic regression model with overdose control will be used to guide dose escalation/ de-escalation in cohorts A, B, C and D(dose finding). The BLRM is introduced in Section 7.1, which also specifies the prior for the model in cohort A. The priors for other dose finding cohorts (B, C and D(dose finding)) will be documented in the TSAP. After patients in each dose group have completed at least one course of treatment, the prior distributions will be updated through Gibbs sampling procedures with the accumulated DLT data from the MTD evaluation period. Posterior probabilities for the rate of DLT will be summarised from BLRM. Selection of the next dose combinations will be based on these probabilities as well as on other safety and laboratory data.

The purpose of this statistical appendix is to present performance metrics (operating characteristics) that illustrate the precision of the design in estimating the MTD under various dose-toxicity relationships through computer simulation. These results are summarized in <u>Table 10.6: 3</u>. In addition, recommendations of the next dose combination by the BLRM with overdose control principle are also provided under various hypothetical outcome scenarios in

Trial Protocol


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

early dose groups to show how it facilitates on-study dose-escalation decisions (see <u>Table 10.6:</u> <u>1</u>).

# Hypothetical data scenarios

Hypothetical data scenarios are shown in <u>Table 10.6: 1</u>. These scenarios reflect potential on-study data constellations and related escalation as allowed by the model. For each scenario, the probability of target dose and overdose for the current dose combination, as well as the next potential dose combination and related probabilities of under-dosing, target dose, and overdosing are shown.

For example, scenario 1 shows the example, that at the starting dose combination 150 mg abemaciclib and 1000 mg xentuzumab none of 3 patients experiences a DLT. Then, the BLRM allows treating patients at the same dose which is the maximum combination dose allows by the protocol.

Scenario 4 shows the example, that at the starting dose combination 150 mg abemaciclib and 1000 mg xentuzumab none of 6 patients experiences a DLT. Therefore, the MTD in this case would be the combination of 150 mg / 1000 mg.

Scenario 6 shows the example that at the starting dose combination 150 mg abemaciclib and 1000 mg xentuzumab 2 out of 3 patients experiences a DLT, then none of 3 patients treated at 100 mg / 1000 mg experiences a DLT. The overdose control of the BLRM suggests escalating to 150 mg / 750 mg.

All these scenarios illustrate the adaptive behaviour of the model even in extreme situations.

Table 10.6: 1 Hypothetical data scenarios for cohort A

| Scenario | Dose combination (mg/mg) | # patient<br>/ # DLT | | nt dose | Next recommended dose combination* | | Next dos<br>ombination | |
|---|---|---|---|---|---|---|---|---|
| | | | P(TD) | P(OD) | | P(UD) | P(TD) | P(OD) |
| 1 | 150/1000 | 3 / 0 | 0.179 | 0.027 | 150/1000 | 0.794 | 0.179 | 0.027 |
| 2 | 150/1000 | 3 / 1 | 0.376 | 0.141 | 150/1000 | 0.483 | 0.376 | 0.141 |
| 3 | 150/1000 | 3 / 2 | 0.397 | 0.430 | 100/1000 | 0.473 | 0.365 | 0.162 |
| 4 | 150/1000<br>150/1000 | 3 / 0<br>3 / 0 | 0.116 | 0.009 | 150/1000 | 0.876 | 0.116 | 0.009 |
| 5 | 150/1000<br>150/1000 | 3 / 1<br>3 / 0 | 0.312 | 0.048 | 150/1000 | 0.640 | 0.312 | 0.048 |
| 6 | 150/1000<br>100/1000 | 3 / 2<br>3 / 0 | 0.309 | 0.053 | 150/750 | 0.324 | 0.491 | 0.185 |

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 10.6: 1 (cont.) Hypothetical data scenarios for cohort A

| Scenario | Dose combination (mg/mg) | # patient<br>/ # DLT | | nt dose | Next recommended dose combination* | | Next dos | |
|---|---|---|---|---|---|---|---|---|
| 7 | 150/1000<br>100/1000<br>100/1000 | 3 / 2<br>3 / 0<br>3 / 1 | 0.428 | 0.081 | 100/1000 | 0.491 | 0.428 | 0.081 |

<sup>\*</sup> Recommended dose combination is the dose combination with the highest target probability. Note that other combinations have similar target toxicity probabilities.

# **Operating characteristics**

Operating characteristics are a way to assess the long-run behaviour of a model by illustrating the precision of the design in estimating the MTD. Under an assumed true dose-toxicity curve, metrics such as the probability of recommending a dose combination with true DLT rate in the target interval can be approximated via simulation.

<u>Table 10.6: 2</u> describes 4 assumed true dose-toxicity scenarios which were used to assess the operating characteristics of this model. These scenarios reflect a wide range of possible cases as follows:

- \* Scenario 1: aligned with prior means
- \* Scenario 2: high-toxicity scenario
- \* Scenario 3: low-toxicity scenario
- \* Scenario 4: low-high-toxicity scenario

Table 10.6: 2 Assumed true dose-toxicity scenarios for cohort A

| Dose | | | Scen | nario | |
|---|---|---|---|---|---|
| combination (mg/mg) | | 1: Prior | 2: High Tox | 3: Low Tox | 4: Low-High |
| 100/750 | | 0.083 | 0.16 | 0.03 | 0.08 |
| 150/750 | D(DI T) | 0.137 | 0.24 | 0.08 | 0.16 |
| 100/1000 | P(DLT) | 0.092 | 0.17 | 0.06 | 0.10 |
| 150/1000 | | 0.150 | 0.31 | 0.10 | 0.20 |

For each of these scenarios, 1000 trials were simulated. Each cohort consisted of 3 patients and dose escalation complied with the following rule:

• Escalate to the dose combination which maximises the probability of the targeted toxicity region and satisfies the overdose criterion

Trial Protocol


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The MTD was considered reached if at least 6 patients have been evaluated at a dose combination which is the model's recommendation for the next dose-level cohort and for which the posterior probability of targeted toxicity was at least 50%. Or if in total 6 patients have been evaluated at a dose combination which is the model's recommendation for the next dose-level cohort.

It was then assessed how often a dose combination was declared as MTD with true DLT rate in the under-, targeted or over-dose range.

Furthermore, the average, minimum and maximum number of patients per trial and the average number of DLTs per trial are reported. Results are shown in <u>Table 10.6: 3</u> below.

| Table 10.6: 3 | Simulated operating | characteristics | for cohort A |
|---------------|---------------------|-----------------|--------------|
|---------------|---------------------|-----------------|--------------|

| Scenario | % of trials declaring a MTD with true DLT rate in | | | DLT rate in | # Patients | # DLTs |
|---|---|---|---|---|---|---|
| | underdose | target dose | overdose | Stopped | Mean<br>(Min-Max) | Mean<br>(Min-Max) |
| 1: Prior | 43.7 | 54.3 | 0 | 2.0 | 10.86<br>(3, 21) | 2.19 (0, 8) |
| 2: High<br>Tox | 0 | 68.3 | 23.3 | 8.4 | 10.68<br>(3, 21) | 3.10<br>(1, 9) |
| 3: Low<br>Tox | 23.9 | 73.3 | 0 | 2.8 | 11.94<br>(3, 21) | 1.75<br>(0, 7) |
| 4: Low-<br>High | 3.9 | 55.1 | 38.9 | 2.1 | 12.10<br>(3, 21) | 2.91<br>(1, 9) |

In scenario 1, which reflects the case that the true dose-toxicity is aligned with prior means, almost all of the simulated trials (54%) that have found a MTD declared the MTD with true toxicity rate in the target interval. Few simulated trials (2.0%) have been stopped before declaring a MTD. None of trials declared a MTD with true DLT rate in the overdose interval.

In scenario 2 (high-toxicity scenario) 68% of the simulated trials that have found a MTD declared the MTD with true toxicity rate in the target interval and 23% declared a MTD with true DLT rate in the overdose interval. Few simulated trials (8%) have been stopped before declaring a MTD.

Scenario 3 (low-toxicity scenario) illustrates a behaviour similar to scenario 1.

Scenario 4, a mixture of the high toxicity and the low toxicity scenario, shows characteristics of both of these.

The mean patient numbers range from 10.68 patients (Scenario 2) to 12.10 patients (Scenario 4) and the maximum number of patients was 21. Therefore, the patient numbers are as expected.

Trial Protocol


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

By reviewing the metrics presented, it can be seen that the model is not sensitive to different scenarios of truth. In general, this model is conservative due to the overdose control criteria. In all scenarios, the probabilities of recommending a dose combination with true  $P(DLT) \ge 33\%$  as MTD are much smaller than probabilities of recommending a dose combination with true P(DLT) between 16% and 33% as MTD.

On-study recommendations based on the model are consistent with the clinical decision making process, and should be considered in conjunction with other available clinical information by the SC in deciding the dose levels to be tested in order to determine the MTD estimates.

R version 3.2.2 was used for data scenarios and simulations.

c09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 11. DESCRIPTION OF GLOBAL AMENDMENT(S)

# 11.1 GLOBAL AMENDMENT 1

| Number of global amendment | 1 |
|---|---|
| Date of CTP revision | 30 January 2017 |
| EudraCT number | 2016-003142-85 |
| BI Trial number | 1280.18 |
| BI Investigational Product(s) | Xentuzumab (BI 836845) |
| Title of protocol | An open label, phase Ib, dose-escalation study |
| This of protocor | evaluating the safety and tolerability of |
| | xentuzumab and abemaciclib in patients with |
| | locally advanced or metastatic solid tumours and |
| | in combination with endocrine therapy in patients |
| | with locally advanced or metastatic hormone |
| | receptor-positive, HER2-, breast cancer, followed |
| | by expansion cohorts |
| To be implemented only after | Yes |
| approval of the IRB / IEC / | |
| <b>Competent Authorities</b> | |
| To be implemented | No |
| immediately in order to | |
| eliminate hazard – | |
| IRB / IEC / Competent | |
| Authority to be notified of | |
| change with request for | |
| approval | |
| Can be implemented without | No |
| IRB / IEC / Competent | |
| Authority approval as changes | |
| involve logistical or | |
| administrative aspects only | 1 |
| | Oli i IT i ID a di Gia |
| Section to be changed | Clinical Trial Protocol Synopsis – Main Criteria |
| D : ( C ) | for inclusion – Cohort A (Solid Tumours) |
| Description of change | Clarification of the inclusion criteria referring to |
| D. C. L. C. L. | previous treatment for trial disease |
| Rationale for change | Revision of the wording as per FDA request |
| Soution to be above at | Clinical Trial Protectal Communic Main C. ' |
| Section to be changed | Clinical Trial Protocol Synopsis – Main Criteria |
| Description of shares | for inclusion – Cohort E |
| Description of change | Additional request to have NSCLC disease confirmed by histology or cytology |
| Dationals for shares | i ei i ei |
| Rationale for change | Revision of the criteria as per FDA request |
| Section to be shared | Clinical Trial Duotagal Samanaia Main Cuitaria |
| Section to be changed | Clinical Trial Protocol Synopsis – Main Criteria |
| | for inclusion – Exclusion criteria |

09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies c09049566-10

| Description of change | Revision of the starting time of trial treatment 3 half-lives after previous immunotherapy instead |
|---|---|
| | of 2. |
| Rationale for change | As per FDA request and in order to minimize |
| 0 | overlapping toxicities |
| Section to be changed | Flow Chart Cohort E and F – Blood sample for |
| | Biomarkers |
| Description of change | Correction of sampling timepoint at Run-In V3 |
| Rationale for change | Revision of the whole protocol and in order to |
| | keep consistency between sections. No Biomarker |
| | sampling needed at Run-In V3 for Cohorts E and F. |
| | 1. |
| Section to be changed | Flow Chart Cohort F – Footnote #11 |
| Description of change | Change details form Cohort G to Cohort F |
| Rationale for change | Correction of a typographic error, as no Cohort G |
| | planned in the final protocol |
| Section to be changed | Section 3.3.2. Inclusion Criteria – Cohort A – |
| | Criteria #7 |
| Description of change | Clarification of the inclusion criteria referring to |
| | previous treatment for trial disease |
| Rationale for change | Revision of the wording as per FDA request |
| Section to be changed | Section 3.3.2. Inclusion Criteria – Cohort B, C, D, |
| Section to be changed | F (Breast Cancer) – Criteria #8 |
| Description of change | Definition of the HER2 negativity as per |
| Description of change | ASCO/CAP guidelines |
| Rationale for change | Inclusion of this references as per FDA request |
| Section to be changed | Section 3.3.2. Inclusion Criteria – Cohort B, C, D, |
| | F (Breast Cancer) – Criteria #10 |
| Description of change | Change from Cohort G to Cohort F |
| Rationale for change | Correction of a typographic error, as no Cohort G |
| | planned in the final protocol |
| Cookien to be altered | Section 2.2.2 Inclusion Cuitaria Colont E |
| Section to be changed | Section 3.3.2. Inclusion Criteria – Cohort E |
| Description of change | (NSCLC) – Criteria #6 Additional request to have NSCLC disease |
| Description of change | confirmed by histology or cytology |
| Rationale for change | Revision of the criteria as per FDA request |
| randinale for change | 1 Revision of the effects as per 1 DA fequest |
| Section to be changed | Section 3.3.3. Exclusion Criteria #7 |

**c**09049566-10 Trial Protocol 

| D | D |
|---|---|
| Description of change | Revision of the starting time of trial treatment 3 |
| | half-lives after previous immunotherapy instead |
| | of 2. |
| Rationale for change | As per FDA request and in order to minimize |
| | overlapping toxicities |
| Section to be changed | Section 4.1.2.2 Part 2 – Dose finding cohorts B, |
| | C, D |
| <b>Description of change</b> | Clarification of the text referring to starting dose |
| - | of the study drugs |
| Rationale for change | Wording error corrected, in order to add clarity to |
| J | the text |
| | · · |
| Section to be changed | Section 4.1.4.2 Temporary treatment interruption |
| 9 | and dose reduction |
| Description of change | Clarification of the dose interruption |
| 1 8 | recommendations, with special clarification for |
| | potential overlapping toxicities. |
| Rationale for change | As per FDA request and in order to minimize |
| <b>-</b> | overlapping toxicities |
| Section to be changed | Section 4.4.1 Increased serum creatinine |
| Description of change | Inclusion of the need to perform serum cystatin-C |
| • | testing to identify true renal function beyond |
| | monitoring creatinine |
| Rationale for change | As per FDA request and in order to give more |
| 8 | detailed guidelines in case of renal dysfunction |
| Section to be changed | Section 5.3.7. Dose Limiting Toxicities (DLTs) |
| Description of change | Revision of the DLT definition and protocol |
| r | defined DLTs |
| Rationale for change | As per FDA request and in order to give more |
| g | details to this section. |
| | stimus to mis stitusii. |

 
 09049566-10
 Trial Protocol
 

 Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies
 c09049566-10

## 11.2 **GLOBAL AMENDMENT 2**

| Number of global amendment | 2 |
|---|---|
| Date of CTP revision | 22 September 2017 |
| EudraCT number | 2016-003142-85 |
| BI Trial number | 1280.18 |
| BI Investigational Product(s) | Xentuzumab (BI 836845) |
| Title of protocol | An open label, phase Ib, dose-escalation study |
| P | evaluating the safety and tolerability of |
| | xentuzumab and abemaciclib in patients with |
| | locally advanced or metastatic solid tumours and in |
| | combination with endocrine therapy in patients |
| | with locally advanced or metastatic hormone |
| | receptor-positive, HER2-, breast cancer, followed |
| | by expansion cohorts |
| To be implemented only after | Yes |
| approval of the IRB / IEC / | |
| Competent Authorities | |
| To be implemented | No |
| immediately in order to | |
| eliminate hazard – | |
| IRB / IEC / Competent | |
| Authority to be notified of | |
| change with request for | |
| approval Can be implemented without | No |
| Can be implemented without IRB / IEC / Competent | NO |
| Authority approval as changes | |
| involve logistical or | |
| administrative aspects only | |
| The state of the s | |
| Section to be changed | Clinical Trial Protocol Synopsis – Main Criteria for |
| | inclusion – Cohort E |
| Description of change | Clarification on number of prior lines that |
| | participants must have received |
| Rationale for change | To make text consistent with inclusion criteria in |
| | section 3.3.2. |
| Section to be changed | Clinical Trial Protocol Synopsis – Main Criteria for |
| | exclusion |
| Description of change | Clarification on prior therapies and unresolved |
| | toxicities |
| Rationale for change | To make text consistent with exclusion criteria in |
| | section 3.3.3. |
| Section to be changed | Flow Chart Cohort E – Footnote #6 |
| Description of change | Change detail for Run-in visit 2 |

| Dationals for shares | Compation against to the Flory Chart |
|---|---|
| Rationale for change | Correction according to the Flow Chart |
| Castian ta ha aba | Eleve Chart Calcart E |
| Section to be changed | Flow Chart Cohort F |
| Description of change | Added footnote reference for Fulvestrant |
| Rationale for change | Correction of typographic error |
| Section to be changed | Section 3.3.3. Exclusion Criteria #3 |
| Description of change | Change the word enrolment for treatment |
| Rationale for change | To avoid confusing terminology |
| Section to be changed | Section 3.3.3. Exclusion Criteria #7 |
| Description of change | Exclusion of prior corticosteroids is deleted |
| Rationale for change | To keep consistency with section 4.2.2. |
| The state of the s | |
| Section to be changed | Section 3.3.3. Exclusion Criteria #10 |
| Description of change | Clarification of the exclusion criteria referring to |
| Description of change | unresolved toxicities from prior treatment |
| Rationale for change | To add clarity to the criteria |
| Rationale for Change | 10 add clarity to the criteria |
| Cootion to be abouted | Section 3.3.3. Exclusion Criteria #18 |
| Section to be changed | |
| Description of change | Threshold added for diabetes |
| Rationale for change | To keep consistency with the synopsis |
| Section to be changed | 4.1.4.1 Initial study drug assignment and |
| | administration |
| Description of change | Change of term referring to dose finding cohorts |
| Rationale for change | Correct wording error |
| Section to be changed | 4.1.4.2 Temporary treatment interruption and dose |
| | reduction |
| Description of change | Clarification on re-escalation possibilities |
| Rationale for change | To improve wording clarity |
| Section to be changed | 4.1.4.2 Temporary treatment interruption and dose |
| | reduction |
| Description of change | Clarification on dose reduction requirements |
| Rationale for change | To keep consistency within the section |
| , | |
| Section to be changed | 4.1.4.2 Temporary treatment interruption and dose |
| Description of change | Footnote added referring to toxicity management |
| Rationale for change | To clarify instructions for toxicity management |
| Nationale for Change | 10 Clarity instructions for toxicity management |
| Section to be shanged | 1.4.2 Management and grading of infusion |
| Section to be changed | 4.4.2 Management and grading of infusion |
| December 4: first | reactions Clarification on CRE nagaranasting |
| Description of change | Clarification on CRF page reporting |
| Rationale for change | To be consistent with CRF design |

**c**09049566-10 Trial Protocol 

| Section to be changed | 5.3.4 Electrocardiogram |
|---|---|
| Description of change | Correction of cohorts with run-in visits |
| Rationale for change | To correct the typo error |
| | , |
| Section to be changed | 5.3.6.1 Definitions of AEs |
| Description of change | The requirement specific for Japan about the reason |
| • | of the decision about causality is deleted |
| Rationale for change | The requirement is no longer applicable in Japan, |
| Section to be changed | 5.3.7 Dose Limiting Toxicities |
| <b>Description of change</b> | The list of DLTs definitions is revised |
| Rationale for change | To make the text consistent with the study drugs |
| | toxicity profile |
| Section to be changed | 5.4.1 Assessment of Pharmacokinetics |
| Description of change | Clarification is added about sample timepoints |
| Rationale for change | To add some flexibility in the sample time schedule |
| Section to be changed | 5.5 Assessment of biomarker(s) |
| Description of change | Biomarker name corrected and dissociable IGF |
| | added |
| Rationale for change | To correct a typo error and introduce the |
| | dissociable IGF definition |
| Section to be changed | 5.6.1 Assessment of Immunogenicity |
| Description of change | Appendix reference corrected |
| Rationale for change | To correct a typo error |
| Section to be changed | 8.1 Trial approval, patient information, informed |
| D | consent. |
| Description of change | A clause is added to identify the text that is only |
| Dationals for shangs | applicable to Japan To clarify that the toyt is not applicable to all |
| Rationale for change | To clarify that the text is not applicable to all participant countries |
| | participant countries |
| Section to be changed | 10.1 Inducers and Strong Inhibitors of CYP3A4 |
| Description of change | Topical medication considerations |
| Rationale for change | For clarification purposes |
| rationale for change | 1 of clarification purposes |
| Section to be changed | 10.2 Pharmacokinetics plan |
| Description of change | Dissociable IGF is mentioned in the flowcharts for |
| Description of change | the different cohorts |
| Rationale for change | To be consistent with section 5.5 |
| ixationale for change | 10 be consistent with section 3.3 |

 
 09049566-10
 Trial Protocol
 

 Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies
 c09049566-10

## 11.3 **GLOBAL AMENDMENT 3**

| Number of global amendment | 3 |
|---|---|
| Date of CTP revision | 11 Dec 2018 |
| EudraCT number | 2016-003142-85 |
| BI Trial number | 1280.18 |
| BI Investigational Product(s) | Xentuzumab (BI 836845) |
| Title of protocol | An open label, phase Ib, dose-escalation study |
| Time or process | evaluating the safety and tolerability of |
| | xentuzumab and abemaciclib in patients with |
| | locally advanced or metastatic solid tumours and |
| | in combination with endocrine therapy in patients |
| | with locally advanced or metastatic hormone |
| | receptor-positive, HER2-, breast cancer, followed |
| | by expansion cohorts |
| To be implemented only after | Yes |
| approval of the IRB / IEC / | |
| Competent Authorities | |
| To be implemented immediately | No |
| in order to eliminate hazard –<br>IRB / IEC / Competent Authority | |
| to be notified of change with | |
| request for approval | |
| Can be implemented without IRB | No |
| / IEC / Competent Authority | |
| approval as changes involve | |
| logistical or administrative | |
| aspects only | |
| Section to be changed | Clinical Trial Protocol Synopsis |
| Description of change | Different sections updated |
| Rationale for change | To match with the updates in the different |
| | protocol sections. |
| | CILL THE LICE OF THE CILL OF |
| Section to be changed | Clinical Trial Protocol Synopsis-Flow Chart for |
| D : (: 6.1 | Cohorts A, B, C and D (dose finding) |
| Description of change | Footnote #16 corrected |
| Rationale for change | To clarify an bone scan requirement and correct |
| | on day windows for week 60 and week 72 |
| Section to be shared | Clinical Trial Drotocal Symposis Elevy Chart for |
| Section to be changed | Clinical Trial Protocol Synopsis-Flow Chart for |
| Description of shange | Cohort D (dose finding) Footnote #6 modified |
| Description of change | |
| Rationale for change | To reduce the screening window for local FSH and estradiol |
| | and estiation |
| Section to be changed | Clinical Trial Protocal Symansis Flavy Chart |
| Section to be changed | Clinical Trial Protocol Synopsis-Flow Chart<br>Cohort E and F |
| | COHOIT E ANG F |

| Description of change | Footnote #18 corrected |
|---|---|
| Rationale for change | To clarify an bone scan requirement and correct on day windows for week 60 and week 72 |
| Section to be changed | Clinical Trial Protocol Synopsis-Flow Chart |
| | Cohort F |
| <b>Description of change</b> | Footnote #7 modified |
| Rationale for change | To reduce the screening window for local FSH and estradiol |
| Section to be changed | Clinical Trial Protocol Synopsis-Flow Chart<br>Expansion cohorts D1 and D2 |
| Description of change | New Flow Chart added |
| Rationale for change | To describe the schedule of activities for BC expansion cohorts D1 and D2 |
| Section to be changed | 1.2 Drug Profile |
| Description of change | Text added in the IMPs profile information |
| Rationale for change | To update with available information |
| Section to be changed | 2.1 Rationale for performing the trial |
| Description of change | Text added |
| Rationale for change | Updated information and added rationale for expansion cohorts D1 and D2 |
| Section to be changed | 2.2 Trial Objectives |
| Description of change | Text added |
| Rationale for change | Primary objective for expansion cohorts D1 and D2 is described |
| Section to be changed | 3.1 Overall Trial Design and Plan |
| Description of change | Part 3 design update |
| Rationale for change | To include and describe expansion cohorts D1 and D2 |
| Section to be changed | 3.2 Discussion of Trial Design |
| Description of change | Section updated |
| Rationale for change | For expansion cohorts D1 and D2 description |
| Section to be changed | 3.3 Selection of Trial Population |
| Description of change | Change the total number of subjects and sites |
| Rationale for change | To update the figures needed as per the new cohorts addition |
| Section to be changed | 3.3.2 Inclusion criteria-Cohort A and E: #5 |

**c**09049566-10 Trial Protocol 

| Description of change | Required contraception methods timelines updated |
|---|---|
| Rationale for change | According to the updated abemaciclib risk profile |
| Section to be changed | 3.3.2 Inclusion criteria-B, C, D(dose finding) and F Cohorts: #5 |
| Description of change | Postmenopausal status requirements wording revision |
| Rationale for change | To improve specificity and clarity in the criteria |
| Section to be changed | 3.3.2 Inclusion criteria- cohorts D1 and D2 |
| Description of change | Cohorts D1 and D2 inclusion criteria added |
| Rationale for change | To describe inclusion criteria for expansion cohorts D1 and D2 |
| Section to be changed | 3.3.3 Exclusion criteria(cohorts A, B, C, D(dose finding), E and F: #7 |
| Description of change | Text modified |
| Rationale for change | To relax washout required periods |
| Section to be changed | 3.3.3 Exclusion criteria (cohorts A, B, C, D(dose finding), E and F: #12 |
| Description of change | Clarifications on central nervous system disease |
| Rationale for change | To further clarify |
| Section to be changed | 3.3.3 Exclusion criteria (cohorts A, B, C, D(dose finding), E and F: #24 |
| Description of change | Clarification added on active infections |
| Rationale for change | To be more specific on active infection definition |
| Section to be changed | 3.3.3 Exclusion criteria:#27 |
| Description of change | New criteria |
| Rationale for change | To exclude prior everolimus treatment for cohort F |
| Section to be changed | 3.3.3 Exclusion criteria- cohorts D1 and D2 |
| Description of change | Cohorts D1 and D2 exclusion criteria added |
| Rationale for change | To describe exclusion criteria for expansion cohorts D1 and D2 |
| Section to be changed | 3.3.5 Replacement of patients |
| Description of change | Text added for dose interruption both for xentuzumab and abemaciclib. Also replacement for cohorts E and F is added. |
| Rationale for change | For clarification purposes for dose interruption and provide new instruction for cohort E and F |

09049566-10 Trial Protocol 
Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies c09049566-10

| Section to be changed | 4.1.2 Selection of doses in the trial |
|---|---|
| Description of change | Updated information for Part 3 |
| Rationale for change | To include the information for cohorts D1 and D2 |
| 2 | |
| Section to be changed | 4.1.4.2 Temporary treatment interruption and |
| | dose reduction |
| <b>Description of change</b> | Text revised for overlapping toxicities and DLT |
| | management |
| Rationale for change | Clarification on the management of overlapping |
| | toxicities and DLTs |
| | 4 1 4 2 2 T-11. |
| Section to be changed | 4.1.4.2:2 Table |
| Description of change | Header changed To clarify that the table is about abemaciclib |
| Rationale for change | possibly related toxicity. |
| | possibly related toxicity. |
| Section to be changed | 4.2.2.1 Restrictions regarding concomitant |
| section to be enanged | treatment |
| <b>Description of change</b> | Paragraph deleted as per restrictions for |
| I | abemaciclib. |
| Rationale for change | Revise the text about CYP3A4 restrictions |
| Section to be changed | 4.2.2.3 Restrictions regarding men and women of |
| | childbearing potential |
| <b>Description of change</b> | Required contraception methods timelines |
| | updated |
| Rationale for change | According to the updated abemaciclib risk profile |
| | 1 1227 B 4 1 4 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 |
| Section to be changed | 4.2.2.7 Restrictions regarding ovarian suppression New section added |
| Description of change | Requirement added to ensure the postmenopausal |
| Rationale for change | status is maintained |
| | Status is maintained |
| Section to be changed | 4.4.2 Management and grading of infusion |
| Section to be enumera | reactions |
| Description of change | IRR Management instructions revised |
| Rationale for change | To be in alignment with other xentuzumab trials |
| 9 | |
| Section to be changed | 4.4.3 Management on neutropenia |
| Description of change | New section added |
| Rationale for change | To reinforce and ensure the monitoring of |
| | neutropenia as expected adverse event. |
| Section to be changed | 4.4.4 Management of hepatotoxicity |
| <b>Description of change</b> | New section added |

09049566-10 Trial Protocol 
Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies c09049566-10

| Rationale for change | To provide guidance on the management of |
|-----------------------|-----------------------------------------------------|
| | hepatotoxicity as expected adverse event. |
| Section to be changed | 5.1.1 Primary endpoint(s) |
| Description of change | Section updated for expansion cohorts D1 and D2 |
| Rationale for change | To describe primary endpoint for expansion |
| ge | cohorts D1 and D 2 |
| | Volicito D I wild D 2 |
| Section to be changed | 5.1.2 Secondary endpoint(s) |
| Description of change | Section updated for expansion cohorts D1 and D2 |
| Rationale for change | Secondary endpoint added for expansion cohorts |
| Kationale for change | D1 and D2 |
| | D1 and D2 |
| Carting to be about 1 | |
| Section to be changed | |
| Description of change | |
| D. (1. 1. 0. 1. | |
| Rationale for change | |
| Section to be changed | 5.2 Assessment of efficacy |
| Description of change | Text added for bone scans requirements |
| Rationale for change | To clarify on the follow up requirements for bone |
| | metastasis assessments |
| Section to be changed | 5.3.6.2 Adverse event collection and reporting |
| Description of change | Instructions added for female partner in the |
| | pregnancy section |
| Rationale for change | To extend the requirements of DEDP reporting to |
| G | the female partner of a male participant |
| Section to be changed | 5.3.7 Dose limiting toxicities (DLTs) |
| Description of change | Revision of DLT definitions |
| Rationale for change | To excluded some hematologic toxicities and IRR |
| Section to be changed | 5.4.2 Methods of sample collection |
| Description of change | Clarification on plasma samples use |
| Rationale for change | No needed to wait until completion of the study to |
| radionale for change | use them. |
| | doc mem. |
| Section to be changed | 5.5 Assessment of biomarker(s) |
| 9 | |
| Description of change | Addition of sample retention plan |
| Rationale for change | To clarify on remaining sample retention |
| | timelines |
| Section to be changed | 6.2. Details of trial procedures at selected visits |

09049566-10 Trial Protocol 
Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies c09049566-10

| Description of change | Description added for cohorts D1 and D2 |
|---|---|
| | procedures (6.2.2.3) |
| Rationale for change | To describe the procedures required for expansion cohorts D1 and D2 |
| Section to be changed | 7.3 Planned analysis |
| Description of change | Description added for the possibility of primary |
| • | analysis for the expansion cohorts |
| Rationale for change | To clarify on the primary analyses planned |
| Section to be changed | 7.3.1 Primary endpoints analysis |
| Description of change | Addition of planned analysis for expansion cohorts D1 and D2 |
| Rationale for change | To update for cohorts D1 and D2 addition |
| 100 01 | |
| Section to be changed | 7.3.2 Secondary endpoint analyses |
| Description of change | Addition of secondary endpoint analyses for |
| | cohorts D1 and D2 |
| Rationale for change | To update for cohorts D1 and D2 addition |
| | • |
| Section to be changed | 7.3.5 Pharmacokinetic and pharmacodynamics |
| S | analyses |
| Description of change | Addition of a clarification on the NCA |
| Rationale for change | To clarify that only applies to the expansion |
| | cohorts |
| Section to be changed | 7.4 Interim analyses |
| <b>Description of change</b> | Added an statement about earlier efficacy analyses |
| Rationale for change | To clarify that other efficacy analyses may be |
| G | performed |
| Section to be changed | 7.7 Determination of sample size |
| Description of change | Descriptions added for cohorts D1 and D2 |
| Rationale for change | To update for cohorts D1 and D2 addition |
| Section to be changed | 8.6 Trial milestones |
| Description of change | Addition of description of LPLVPE-expansion for |
| | cohorts D1 and D2 |
| Rationale for change | To specify different milestone for different |
| | expansion cohorts |
| Section to be changed | 10.2.3.2 Flow chart for PK, immunogenicity, and |
| | biomarkers for Cohort F in treatment course 2 |
| Description of change | Updates on the events |

c09049566-10

99049566-10 Trial Protocol 
Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Rationale for change | Clarifications on the requirements about the sampling related to the abemaciclib intake |
|---|---|
| Section to be changed | 10.2.4 Flow chart for PK, immunogenicity, and |
| <u> </u> | biomarkers for cohorts D1 and D2 |
| Description of change | New flow charts |
| Rationale for change | To describe the required sampling for cohorts D1 |
| | and D2 |

 
 09049566-10
 Trial Protocol
 

 Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies
 c09049566-10

## 11.4 **GLOBAL AMENDMENT 4**

| Number of global amendment | 4 |
|---|---|
| Date of CTP revision | 09 Apr 2019 |
| EudraCT number | 2016-003142-85 |
| BI Trial number | 1280.18 |
| BI Investigational Product(s) | Xentuzumab (BI 836845) |
| Title of protocol | An open label, phase Ib, dose-escalation study |
| Title of protocor | evaluating the safety and tolerability of |
| | xentuzumab and abemaciclib in patients with |
| | locally advanced or metastatic solid tumours and |
| | in combination with endocrine therapy in patients |
| | with locally advanced or metastatic hormone |
| | receptor-positive, HER2-, breast cancer, followed |
| | by expansion cohorts |
| To be implemented only after | Yes |
| approval of the IRB / IEC / | |
| Competent Authorities | |
| To be implemented immediately | No |
| in order to eliminate hazard – | |
| IRB / IEC / Competent Authority | |
| to be notified of change with | |
| request for approval Can be implemented without IRB | No |
| / IEC / Competent Authority | INO |
| approval as changes involve | |
| logistical or administrative | |
| aspects only | |
| Section to be changed | Clinical Trial Protocol Synopsis |
| Description of change | Main criteria for inclusion for diagnosis of breast |
| | cancer corrected |
| Rationale for change | To be consistent with section 3.3.2 |
| Section to be changed | Clinical Trial Protocol Synopsis |
| Description of change | Correction of flowchart for cohorts C and D for |
| | baseline tumour assessment timepoint |
| Rationale for change | For consistency |
| Section to be changed | Clinical Trial Protocol Synopsis |
| Description of change | Footnote #16 in Flowchart for Cohorts D1 and |
| | D2 corrected |
| Rationale for change | To be consistent with 10.2.4.3 flowchart |
| Section to be changed | 1.2 Drug profile |
| Description of change | Safety profile for xentuzumab updated |
| Rationale for change | Updated data as per cut off of 2019 |

| Section to be changed | 2.1 Rationales for performing the trial |
|---|---|
| Description of change | Correction made when describing expansion |
| z everiperon or enunge | cohorts |
| Rationale for change | Letrozole and anastrozole are not used |
| 9 | |
| Section to be changed | 2.3 Benefit-Risk Assessment |
| Description of change | Data for xentuzumab updated |
| Rationale for change | To keep the information up to date |
| | • |
| Section to be changed | 3.3.2 Inclusion criteria |
| <b>Description of change</b> | In #9 for cohorts D1 and D2 corrected |
| Rationale for change | To be consistent with abemaciclib risk profile |
| | • |
| Section to be changed | 3.3.3 Exclusion criteria |
| Description of change | Ex #17 for Cohorts D1 and D2 corrected |
| Rationale for change | Letrozole and anastrozole do not apply for those |
| | cohorts |
| Section to be changed | 4.1.4.2 temporary treatment interruption and dose |
| | reduction |
| Description of change | Guidelines for abemaciclib toxicity management |
| | update |
| Rationale for change | To be aligned with the most recent abemaciclib |
| | safety information |
| Section to be changed | 4.2.2 Restrictions |
| Description of change | Updated instructions and guidelines as per |
| | inducers and inhibitors of CYP3A |
| Rationale for change | To be aligned with the most recent abemaciclib |
| | safety information |
| Coation to be allowed | AAA Managamant af II tatai -ita- |
| Section to be changed | 4.4.4 Management of Hepatotoxicity |
| Description of change | Updated information and guidelines To be aligned with the most recent change is like |
| Rationale for change | To be aligned with the most recent abemaciclib |
| | safety information |
| Section to be changed | 4.4.5 Venous Thromboembolism |
| Section to be changed Description of change | New section added |
| Rationale for change | To provide information ad instructions to manage |
| Nationale for change | the adverse event |
| | the adverse event |
| Section to be changed | 10.1 Inducers and strong inhibitors of CYP3A4 |
| Description of change | The lists of the strong inhibitors and substrates are |
| Description of change | updated |
| | updated |

Boehringer Ingelheim BI Trial No.: 1280.18

| Rationale for change | To be aligned with the most recent abemaciclib |
|---|---|
| | safety information |
| Section to be changed | 10.2.4.1 Flowchart for PK, AD and biomarkers |
| S | for cohorts D1 and D2 in course 1 |
| <b>Description of change</b> | Footnote deleted |
| Rationale for change | For consistency |
| Section to be changed | 10.2.4.2 Flowchart for PK, AD and biomarkers |
| J | for cohorts D1 and D2 in course 2 |
| <b>Description of change</b> | Fulvestrant PK sample correction |
| Rationale for change | For consistency |
| | · |
| Section to be changed | 10.2.4.3 Flowchart for PK, AD and biomarkers |
| 5 | for cohorts D1 and D2 in courses 3, 4, 6, 12 and |
| | 24 |
| Description of change | Header and footnotes corrected |
| Rationale for change | For consistency |

 
 09049566-10
 Trial Protocol
 

 Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies
 c09049566-10

## **GLOBAL AMENDMENT 5** 11.5

| Number of global amendment | 5 |
|---|---|
| Date of CTP revision | 03 Jul 2019 |
| EudraCT number | 2016-003142-85 |
| BI Trial number | 1280.18 |
| BI Investigational Product(s) | Xentuzumab (BI 836845) |
| Title of protocol | An open label, phase Ib, dose-escalation study evaluating the safety and tolerability of xentuzumab and abemaciclib in patients with locally advanced or metastatic solid tumours and in combination with endocrine therapy in patients with locally advanced or metastatic hormone receptor-positive, HER2-, breast cancer, followed by expansion cohorts |
| To be implemented only after approval of the IRB / IEC / Competent Authorities | Yes |
| To be implemented immediately in order to eliminate hazard – IRB / IEC / Competent Authority to be notified of change with request for approval | No |
| Can be implemented without IRB / IEC / Competent Authority approval as changes involve logistical or administrative aspects only | No |
| Section to be changed | 3.3.3 Exclusion criteria |
| Description of change | Exclusion criteria #13 was updated to exclude subjects with ILD and other respiratory disorders |
| Rationale for change | To be in accordance with updated abemaciclib safety information |
| Section to be changed | 4.4.6 Guidance for ILD/Pneumonitis |
| Description of change | New section added |
| Rationale for change | To be in accordance with updated abemaciclib safety information |

 
 09049566-10
 Trial Protocol
 

 Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies
 c09049566-10

## **GLOBAL AMENDMENT 6** 11.6

| Date of amendment | 23 Dec 2019 |
|---|---|
| EudraCT number | 2016-003142-85 |
| BI Trial number | 1280.18 |
| BI Investigational Product(s) | Xentuzumab (BI 836845) |
| Title of protocol | An open label, phase Ib, dose-escalation study |
| Title of proceed | evaluating the safety and tolerability of |
| | xentuzumab and abemaciclib in patients with |
| | locally advanced or metastatic solid tumours and |
| | in combination with endocrine therapy in patients |
| | with locally advanced or metastatic hormone |
| | receptor-positive, HER2-, breast cancer, followed |
| | by expansion cohorts |
| Global Amendment due to urgent safet | |
| Global Amendment | |
| Section to be changed | Clinical Trial Protocol Synopsis |
| Description of change | Asia region included for trial sites |
| Rationale for change | To extend to other Asian sites participation |
| Section to be changed | Clinical Trial Protocol Synopsis |
| Description of change | Tablets mentioned in the eligibility criteria |
| Rationale for change | To be consistent with section 3.3.2 |
| Section to be changed | Clinical Trial Protocol Synopsis |
| Description of change | Alpelisib added as prior treatment in the |
| | exclusion criteria for cohorts D1 and D2 |
| Rationale for change | For a better definition of trial population in |
| | reaction to a newly approved treatment |
| Section to be changed | 3.3.2 Inclusion criteria |
| Description of change | Tablets added to inclusion criteria #4 for all |
| | cohorts |
| Rationale for change | To be consistent with the possibility of tablets |
| | intake |
| Coation to be abouted | 2.2.2 In alwais a suitania |
| Section to be changed | 3.3.2 Inclusion criteria Inclusion criteria #9 for cohorts D1 and D2 |
| Description of change | |
| | updated as per the contraception period required for xentuzumab |
| Dationals for shange | Re-assessment of contraception requirements for |
| Rationale for change | xentuzumab for WOCBP, including PK |
| | variability and normalization of PD effects. |
| | variability and normalization of FD effects. |
| Section to be changed | 3.3.3 Exclusion criteria |
| Section to be changed | J.J.J EXCLUSION CHICHA |

09049566-10 Trial Protocol 
Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies c09049566-10

| Description of change | Alpelisib added as prior treatment excluded for |
|---|---|
| D. C. L. C. L. | cohorts D1 and D2 |
| Rationale for change | For a better definition of trial population in |
| | reaction to a newly approved treatment |
| Section to be changed | 4.1.1 Identity of the Investigational Medicinal |
| section to be changed | Products |
| Description of change | Information added about abemaciclib tablets |
| Description of enunge | formulation |
| Rationale for change | Abemaciclib tablets can be administered to the |
| | study subjects |
| Section to be changed | 4.1.4 Drug assignment and administration of |
| | doses for each patient |
| Description of change | The possibility to reduce the abemaciclib dose to |
| D 41 1 6 1 | 50 mg BID was added |
| Rationale for change | To facilitate abemaciclib AE management |
| Section to be changed | 4.1.4 Drug assignment and administration of |
| section to be enauged | doses for each patient |
| <b>Description of change</b> | Guidelines for abemaciclib dose adjustment to |
| Description of enunge | manage ILD/pneumonitis were added |
| Rationale for change | To be consistent with the abemaciclib IB |
| 9 | information |
| Section to be changed | 4.1.7 Storage conditions |
| Description of change | Abemaciclib tablets added |
| Rationale for change | To provide instruction on tablets storage |
| | requirements |
| | 14221 Participation |
| Section to be changed | 4.2.2.1 Restrictions regarding concomitant |
| Description of shapes | Instructions and dated |
| Description of change | Instructions updated To include the options to reduced abemaciclib |
| Rationale for change | dose to 50 mg twice daily. |
| | dose to 50 mg twice daily. |
| Section to be changed | 4.2.2.3 Restrictions regarding men and women of |
| | childbearing potential |
| <b>Description of change</b> | Update on the contraception period required for |
| r | xentuzumab |
| Rationale for change | Re-assessment of contraception requirements for |
| 5 | xentuzumab for WOCBP, including PK |
| | variability and normalization of PD effects. |
| Section to be changed | 4.4.6 Guidance for Interstitial lung |
| | disease/Pneumonitis |

**Boehringer Ingelheim** BI Trial No.: 1280.18

c09049566-10

04 Mar 2022

99049566-10 Trial Protocol 
Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Description of change | Text updated |
|-----------------------|---------------------------------------|
| Rationale for change | To be consistent with table 4.1.4.2:2 |

 
 09049566-10
 Trial Protocol
 

 Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies
 c09049566-10

## 11.7 **GLOBAL AMENDMENT 7**

| Date of amendment | 02 Jul 2020 |
|---|---|
| EudraCT number | 2016-003142-85 |
| BI Trial number | 1280.18 |
| BI Investigational Product(s) | Xentuzumab (BI 836845) |
| Title of protocol | An open label, phase Ib, dose-escalation study |
| Title of protocol | evaluating the safety and tolerability of |
| | xentuzumab and abemaciclib in patients with |
| | locally advanced or metastatic solid tumours and |
| | in combination with endocrine therapy in patients |
| | with locally advanced or metastatic hormone |
| | receptor-positive, HER2-, breast cancer, followed |
| | by expansion cohorts |
| Global Amendment due to urgent safet | |
| Global Amendment | |
| | 1 <del>[</del> ] |
| Section to be changed | Clinical Trial Protocol Synopsis |
| Description of change | Text amended in different sections of the synopsis |
| Rationale for change | To update the synopsis according to the changes |
| | made in different sections of the protocol |
| ' | * |
| Section to be changed | Flow Chart-Cohort F |
| Description of change | Run-in visits and corresponding procedures were |
| | removed |
| Rationale for change | The run-in data from cohort F is no longer |
| | required for analysis |
| | Pl Cl + C 1 + F |
| Section to be changed | Flow Chart-Cohort F |
| Description of change | A number PK samples in cycle 2 were removed |
| Rationale for change | Those PK samples in cohort F no longer required |
| | for analysis were removed to simplify the study procedures |
| | procedures |
| Section to be changed | Flow Chart-Cohort F |
| Description of change | Tumour assessment requirements in follow up |
| Description of change | period were highlighted |
| Rationale for change | To clarify the instructions to follow up for |
| | progression of disease |
| | 11 0 |
| Section to be changed | Flow Chart Cohorts D1 and D2 |
| Description of change | Tumour assessment requirements in follow up |
| | period were highlighted |
| Rationale for change | To clarify the instructions to follow up for |
| | progression of disease |

99049566-10 Trial Protocol 
Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies c09049566-10

| Section to be changed | 2.2 Trial Objectives |
|---|---|
| Description of change | Trial objectives reworded for cohort F |
| Rationale for change | To accurately describe primary and secondary |
| | objectives for cohort F |
| Section to be changed | 2.3 Benefit-Risk Assessment |
| <b>Description of change</b> | Language was added about Covid-19 infection |
| Rationale for change | To provide information and guidance on Covid- |
| | 19 considerations for the trial |
| Section to be changed | 3.1 Overall Trial Design Plan |
| Description of change | Section updated for cohort F information |
| Rationale for change | To accurately describe the design of cohort F |
| Section to be changed | 3.2 Discussion of Trial Design, including the |
| <b>D</b> | choice of control Group(s) |
| Description of change | Section updated for cohort F |
| Rationale for change | To amend the PK plan for cohort F |
| Section to be abanged | 3.3.2 Inclusion criteria |
| Section to be changed Description of change | Modified for cohort F |
| Description of change Rationale for change | To provide a detailed definition of the inclusion |
| Rationale for change | criteria for cohort F |
| | Criteria for conort i |
| Section to be changed | 3.3.3 Exclusion criteria |
| Description of change | Modified for cohort F |
| Rationale for change | To provide a detailed definition of the exclusion |
| Turionale for enange | criteria for cohort F |
| Section to be changed | 3.3.5 Replacement of patients |
| Description of change | Amended for cohort F |
| Rationale for change | To be consistent with the endpoints updates for |
| | cohort F |
| Section to be changed | 4.2.2.1 Restrictions regarding concomitant |
| | treatment |
| <b>Description of change</b> | Abemaciclib related information was updated |
| Rationale for change | Modified according to the most current |
| | information in the abemaciclib SmPC |
| | 1 1.0 m |
| Section to be changed | 4.3 Treatment compliance |
| <b>Description of change</b> | Patient diary requirement for cohort F was |
| | removed |
| Rationale for change | To be consistent with the run-in visits removed |
| | 10 0 0 |
| Section to be changed | 4.4.1 Increased Serum Creatinine |

**c**09049566-10 Trial Protocol 

| Description of change | Language was updated |
|---|---|
| Rationale for change | According to the latest abemaciclib information |
| | available |
| Section to be changed | 5.1 Trial Endpoints |
| Description of change | Specific endpoints for cohort F were revised |
| Rationale for change | To accurately describe the primary and secondary |
| G | endpoints for cohort F |
| Section to be changed | 5.5 Assessment of Biomarker(s) |
| Description of change | Headers and footnotes of tables 5.5: 1 and 5.5:2 |
| | were corrected |
| Rationale for change | Correction needed to resolve an inconsistency |
| | with the biomarker sampling plan |
| Section to be changed | 6.1 Visit Schedule |
| Description of change | Language added about the possibility to visit the |
| | patient remotely |
| Rationale for change | That is to mitigate the difficulties to visit the |
| | patient at the site under extraordinary |
| | circumstances such as relevant infection |
| | outbreaks or similar. |
| | COD CT ID 1 CC I CT IV |
| Section to be changed | 6.2 Details of Trial Procedures at Selected Visits |
| Description of change | The procedures description were corrected |
| Rationale for change | To be consistent with the flow charts |
| Section to be changed | 6.2.3.2 Follow up period |
| Description of change | Details added for follow up period for progression |
| Description of change | of disease |
| Rationale for change | To improve the description of the procedures |
| rationale for enange | required during the follow up period |
| Section to be changed | 7.3. Planned Analyses |
| Description of change | Information added for cohort F |
| Rationale for change | To describe the analyses planned for cohort F |
| ) | endpoints |
| Section to be changed | 7.7 Determination of sample size |
| <b>Description of change</b> | Specific description for cohort F was added |
| Rationale for change | Accurately describe the assumptions for cohort F |
| Section to be changed | 10.1 Inducers and strong inhibitors of CYP3A4 |
| Description of change | The list of drugs was revised |
| Rationale for change | According to the most updated abemaciclib |
| | information |

BI Trial No.: 1280.18 c09049566-10

09049566-10 Trial Protocol 

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Section to be changed | 10.2.3 Flow chart for PK, immunogenicity, and |
|-----------------------|------------------------------------------------|
| | biomarkers for cohort F |
| Description of change | The PK profile for cohort F was reduced |
| Rationale for change | To simplify the PK profile removing samples no |
| | longer required |

 
 09049566-10
 Trial Protocol
 

 Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies
 c09049566-10

## 11.8 **GLOBAL AMENDMENT 8**

| Date of amendment | 04 Mar 2022 |
|---|---|
| EudraCT number | 2016-003142-85 |
| BI Trial number | 1280.18 |
| BI Investigational Product(s) | Xentuzumab (BI 836845) |
| Title of protocol | An open label, phase Ib, dose-escalation study |
| Title of protocol | evaluating the safety and tolerability of |
| | xentuzumab and abemaciclib in patients with |
| | locally advanced or metastatic solid tumours and |
| | in combination with endocrine therapy in patients |
| | with locally advanced or metastatic hormone |
| | receptor-positive, HER2-, breast cancer, followed |
| | by expansion cohorts |
| Global Amendment due to urgent safet | |
| Global Amendment | <u> </u> |
| Section to be changed | Flow Chart-Cohort F |
| Description of change | Schedule of activities revised. Some procedures |
| - Francisco Sa sumage | removed |
| Rationale for change | To reflect reduced procedures and assessments to |
| g- | support ongoing patients because of 1280-0022 |
| | primary endpoint analysis results |
| Section to be changed | Flow Chart-Cohorts D1 and D2 |
| Description of change | Schedule of activities revised. Some procedures |
| | removed |
| Rationale for change | To reflect reduced procedures and assessments to |
| | support ongoing patients because of 1280-0022 |
| | primary endpoint analysis results |
| Section to be changed | 2.3 Benefit-Risk assessment |
| Description of change | New text added |
| Rationale for change | Based on the 1280-0022 study results of primary |
| | endpoint analysis |
| | 100417 |
| Section to be changed | 3.3.4.1 Removal of individual patients |
| Description of change | New text added |
| Rationale for change | To refer to the trial termination possibilities |
| | · |
| No atriona do la o algoração d | |
| Section to be changed | 3.3.4.2 Discontinuation of the trial by the sponsor |
| <b>Description of change</b> | New text added |
| Description of change | New text added |

99049566-10 Trial Protocol 
Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies c09049566-10

| Description of change | Xentuzumab treatment discontinuation |
|---|---|
| | recommendation added |
| Rationale for change | Based on benefit-risk change after 1280-022 |
| | primary endpoint analysis results |
| Section to be changed | 5.2 Assessment of efficacy |
| Description of change | Requirements for response assessments reduced |
| Rationale for change | Based on benefit-risk change after 1280-022 |
| Rationale for change | primary endpoint analysis results |
| | primary enuponit anarysis results |
| Section to be changed | 5.3 Assessment of safety |
| Description of change | Requirements for safety assessments reduced |
| Rationale for change | Based on benefit-risk change after 1280-022 |
| iturionare for enunge | primary endpoint analysis results |
| | printery enumerous resource |
| Section to be changed | 5.4.1 Assessment of Pharmacokinetics |
| Description of change | PK samples are no longer collected |
| Rationale for change | Based on benefit-risk change after 1280-022 |
| 8 | primary endpoint analysis results |
| Section to be changed | 5.4.2 Methods of sample collection |
| Description of change | Blood for PK and ADA is no longer collected |
| Rationale for change | Based on benefit-risk change after 1280-022 |
| | primary endpoint analysis results |
| Section to be changed | 5.5 Assessment of biomarker(s) |
| Description of change | biomarkers samples are no longer collected |
| Rationale for change | Based on benefit-risk change after 1280-022 |
| | primary endpoint analysis results |
| Section to be shanged | 5.6.1 A googgament of Immuna oppositive |
| Section to be changed | 5.6.1 Assessment of Immunogenicity |
| <b>Description of change</b> | blood samples for immunogenicity assessments are no longer collected |
| Rationale for change | Based on benefit-risk change after 1280-022 |
| Rationale for change | primary endpoint analysis results |
| | primary enupoint anarysis results |
| Section to be changed | 6.2.2.3 Cohorts D1, D2 and F |
| Description of change | Reference to reduced flow chart |
| Rationale for change | To be consistent with the revised flowcharts for |
| Rationale for change | cohorts D1, D2 and F |
| | conorto D1, D2 unu 1 |
| Section to be changed | 6.2.3.1 End of treatment visit |
| Description of change | Sample collection details removed |
| Rationale for change | To be consistent with flowchart revision |
| Tantonuic ivi change | 10 00 consistent with nowellast tevision |
| Section to be changed | 7.3 Planned analysis |
| Section to be changed | 7.5 I faithful affail yold |

BI Trial No.: 1280.18

| Description of change | Final analysis timepoint description removed |
|---|---|
| Rationale for change | To conduct final analyses before last patient out |
| Section to be changed | 10.2.3 FLOW CHART for PK, immunogenicity, |
| _ | and biomarkers for cohort F |
| <b>Description of change</b> | Blood samples no longer collected |
| Rationale for change | To be consistent with the revised flowchart for |
| G | cohort F |
| Section to be changed | 10.2.4 FLOW CHART for PK, immunogenicity, |
| g | and biomarkers for cohorts D1 and D2 |
| Description of change | Blood samples no longer collected |
| Rationale for change | To be consistent with the revised flowchart for |
| 5 | cohorts D1 and D2 |